

# Clinical Development

# API015A (Cohort I)

#### CAPI015A2201J / NCT02565511

A randomized, double-blind, placebo-controlled cohort to evaluate the efficacy of CAD106 in participants at risk for the onset of clinical symptoms of Alzheimer's disease

Statistical Analysis Plan (SAP)

Author: Trial Statistician,

Document type: SAP Documentation

Document status: Addendum 4

Release date: 29-Jan-2021

Number of pages: 97

Property of Novartis
For business use only
May not be used, divulged, published or otherwise disclosed
without the consent of Novartis

# Document History – Changes compared to previous final version of SAP.

| Date | Time point | Reason for update | Outcome for update | Section<br>and title<br>impacted<br>(Current) |
|---|---|---|---|---|
| 23-JUN-<br>2020 | Prior to<br>DB Lock | Newly created based<br>on existing SAP for<br>the study and the SAP<br>for the corresponding<br>sister study<br>CNP520A2202J and<br>API015A2201J<br>Cohort II for<br>API015A2201J<br>Cohort I CAD106 | Separating Cohort I<br>CAD106 SAP from<br>study API015A2201J<br>SAP | |
| 16-July-<br>2020 | Post-DBL | Creation of addendum 1 | 1. The subgroup of responders/non-responders based on titer data are removed as well as all related reports. 2. A new flag of "on trt" is introduced. The creation of this flag is to indicate whether a visit is on trt or not. This "on trt" flag will be applied all post-baseline cognitive and biomarker endpoint summary tables (replacing the ones of by responder status). 3. Add AUC be one of the titer summary statistics in Section 2.7.2. The calculation of AUC is based on "on trt" visits only with imputation rules. 4. Cmax definition is updated to be: maximum Titer concentration of any post-baseline "on | |

| Date | Time point | Reason for update | Outcome for update | Section<br>and title<br>impacted<br>(Current) |
|---|---|---|---|---|
| | | | treatment" visit in Section 2.7.2 5. Correlation between centiloid and titer is updated to be correlation | ( 7 |
| | | | between centiloid and AUC of "on trt" titer in Section 2.7.2. | |
| | | | 6. Correcting the unit of CSF Abeta 40 at programming level for reporting in Section 4. | |
| 03-Nov-<br>2020 | Post-DBL | Further investigate<br>Amyloid PET outputs | <ol> <li>Add annualized chg<br/>and annualized %<br/>change for both<br/>SUVr by ligand and<br/>centiloids</li> </ol> | |
| | | | <ol> <li>Add Last Assessment visit</li> <li>Add boxplot for post-</li> </ol> | |
| | | | baseline change 4. Add scatter plot for amyloid change vs baseline to assess correlation | |
| | | Further investigate cognitive outputs | <ul><li>5. Add forest plot for<br/>APCC and RBANS</li><li>6. Add scatter plot for<br/>APCC and RBANS</li></ul> | |
| | | | with smoothing curves 7. Add Last Assessment visit | |
| | | Further investigate<br>VolMRI | 8. Add annualized chg to summary tables 9. Add Last Assessment visit | |
| | | Evaluate correlation brain volume vs amyloid | 10. Add scatter plot | |


| Date | Time point | Reason for update | Outcome for update | Section<br>and title<br>impacted<br>(Current) |
|---|---|---|---|---|
| | | Assess AE within 7 days of injection | 11. Add AE tables | |
| | | Evaluate relationship<br>between exposure vs.<br>Amyloid level | 12. Report exposure by Amyloid level | |
| 12-Nov-<br>2020 | Post-DBL | Vital sign should be reported by visit and time point as applicable. | <ul><li>13. Vital sign figure is removed. Vital sign table is modified to be by visit and time point.</li><li>14. Table 5-6 is updated to add body temperature category</li></ul> | |
| 18-Nov-<br>2020 | Post-DBL | Add plasma Abeta-40 to CSR | 15. Tables are added for plasma Abeta-40 | |
| 14-Dec-<br>2020 | Post-DBL | Remove subgroup of CAD on treatment group as it's very much overlapping with CAD group | 16. Impact all cognitive and biomarker reports | |
| | | To better understand<br>the timing of "last<br>assessment" | 17. Add summary tables of "last assessment" for RBANS and VolMRI | |
| | | To summarize NFL data without outlier(s) | 18. Add criteria to exclude outlier(s) | |
| | | Update cut-off date of LPLV to be April 15 2020 | 19. The cut-off is applied to TTE reports | |
| 27-Jan-<br>2021 | Addendum<br>4 | Baseline centiloid<br>values can be<br>negative, and<br>therefore % chg<br>statistics is no longer<br>valid | 20. Remove summary statistics about % chg and annualized % chg for centiloid | |

# **Table of contents**

| | Table | of conte | nts | 5 |
|---|---|---|---|---|
| | List o | of tables | | <mark>7</mark> |
| | List o | of abbrevi | ations | 8 |
| 1 | Intro | duction | | 11 |
| | 1.1 | Study d | lesign | 12 |
| | | 1.1.1 | Study Design Summary | 12 |
| | | 1.1.2 | Planned Number of Participants | 12 |
| | | | | 13 |
| | | 1.1.4 | Primary Analysis Time Point | 13 |
| | | 1.1.5 | Interim Analyses | 13 |
| | 1.2 | Study o | objectives and endpoints | 14 |
| 2 | Statis | tical met | hods | 14 |
| | 2.1 | Data ar | nalysis general information | 14 |
| | | 2.1.1 | General definitions | 15 |
| | 2.2 | Analys | is sets | 17 |
| | | 2.2.1 | Subgroup of interest | 17 |
| | 2.3 | Patient | disposition, demographics and other baseline characteristics | 18 |
| | | 2.3.1 | Patient disposition | 18 |
| | | 2.3.2 | Background and demographic characteristics | 18 |
| | 2.4 | | ents (study treatment, rescue medication, concomitant therapies, ance) | 20 |
| | | 2.4.1 | Study treatment / compliance | |
| | | 2.4.2 | Prior, concomitant and post therapies | |
| | 2.5 | Analys | is of the primary objective | 20 |
| | | 2.5.1 | Primary endpoint | 20 |
| | | 2.5.2 | Statistical hypothesis, model, and method of analysis | 22 |
| | | 2.5.3 | Handling of missing values/censoring/discontinuations | 24 |
| | | 2.5.4 | Supportive analyses | 25 |
| | 2.6 | Analys | is of the key secondary objective | 25 |
| | | 2.6.1 | Key secondary endpoint | |
| | | 2.6.2 | Statistical hypothesis, model, and method of analysis | 25 |
| | | 2.6.3 | Handling of missing values/censoring/discontinuations | 25 |
| | 2.7 | Analys | is of secondary and other efficacy objective(s) | 25 |
| | | 2.7.1 | Secondary and other efficacy endpoints | 25 |
| | | 2.7.2 | Statistical hypothesis, model, and method of analysis | 30 |
| | | 2.7.3 | Handling of missing values/censoring/discontinuations | |

| 2.8 | Safety a | analyses | 35 |
|-------|------------|----------------------------------------|----|
| | 2.8.1 | Adverse events (AEs) | 35 |
| | 2.8.2 | Deaths | 37 |
| | 2.8.3 | Laboratory data | 37 |
| | 2.8.4 | Other safety data | 38 |
| | | | 42 |
| | | | 42 |
| 2.11 | Patient- | -reported outcomes | 42 |
| 2.12 | Biomar | kers | 42 |
| | | | 42 |
| 2.14 | Interim | analysis | 42 |
| | | | 42 |
| Chan | ge to prot | ocol specified analyses | 43 |
| Appe | ndix | | 44 |
| 5.1 | Imputat | tion rules | 44 |
| | 5.1.1 | Study drug | 44 |
| | 5.1.2 | AE date imputation | 44 |
| | 5.1.3 | Concomitant medication date imputation | 44 |
| 5.2 | AEs co | ding/grading | 45 |
| 5.3 | Laborat | tory parameters derivations | 45 |
| 5.4 | Statistic | cal models | 46 |
| | 5.4.1 | Primary analysis | 46 |
| 5.5 | Rule of | exclusion criteria of analysis sets | 46 |
| 5.6 | Notable | e and abnormality criteria | 47 |
| 5.7 | Analysi | is windows rules | 49 |
| 5.8 | RBANS | S Index tables | 58 |
| Refer | ences | | 97 |

| List of tables | | |
|---|---|---|
| Table 2-1 | Amyloid Level Stratification Criteria | 29 |
| Table 2-2 | Calculation of summary parameters for immunogenicity | 34 |
| Table 2-3 | The ARWMC Rating Scale for MRI | 39 |
| Table 5-1 | Latent construct variables and their corresponding subtests | 44 |
| Table 5-2 | Liver Event and Laboratory Trigger Definitions | 45 |
| Table 5-3 | Specific renal alert criteria and actions | 46 |
| Table 5-4 | Deviation codes description | 47 |
| Table 5-5 | Participant Classification | 47 |
| Table 5-6 | Clinically notable criteria for vital signs | 47 |
| Table 5-7 | Clinically notable criteria for selected hematology tests | 47 |
| Table 5-8 | Clinically notable criteria for selected blood chemistry tests | 48 |
| Table 5-9 | ECG Abnormality Ranges | 48 |
| Table 5-10 | Raven's, MMSE and CDR, ECog | 49 |
| Table 5-11 | RBANS, | 50 |
| Table 5-12 | Physical / Neurological exams, ECG, laboratory tests | 52 |
| Table 5-13 | Safety MRI, volumetric MRI, functional MRI | 53 |
| Table 5-14 | Vital signs | 54 |
| Table 5-15 | Injections of CAD106 | 55 |
| Table 5-16 | Antibody response | 56 |
| Table 5-17 | Immediate Memory Index Score Equivalents of Subtest Raw Score | 58 |
| Table 5-18 | Visuospatial/Constructional Index Score Equivalents of Subtest<br>Raw Scores | 63 |
| Table 5-19 | Language Index Score Equivalents of Subtest Raw Scores | 66 |
| Table 5-20 | Attention Index Score Equivalents of Subtest Raw Scores | 73 |
| Table 5-21 | Delayed Memory Index Score Equivalents of Subtest Raw Scores . | 87 |
| Table 5-22 | Total Scale Index Score Equivalents of Sum of Index Scores | 94 |

### List of abbreviations

| List of abbre | viduolio |
|---------------|-------------------------------------------------|
| Αβ | Amyloid-beta |
| AD | Alzheimer's Disease |
| AE | Adverse event |
| AESI | Adverse Event of Special Interest |
| ALT | Alanine Aminotransferase |
| AOPE4 | Apolipoprotein E ε4 allele |
| APCC | API Preclinical Composite Cognitive Battery |
| API | Alzheimer's Prevention Initiative |
| APOE | Apolipoprotein E |
| APP | Amyloid Precursor Protein |
| ARIA | Amyloid Related Imaging Abnormalities |
| ARIA-E | Amyloid Related Imaging Abnormality-edema |
| ARIA-H | Amyloid Related Imaging Abnormality-hemorrhages |
| AST | Aspartate Aminotransferase |
| ATC | Anatomic Therapeutic Chemical classification |
| AUC | Area Under the Curve |
| Αβ | Amyloid-beta |
| BACE | Beta-site-APP Cleaving Enzyme |
| bid | bis in diem/twice a day |
| BSI | boundary shift integral |
| CDR | Clinical Dementia Rating |
| CDR-SOB | Clinical Dementia Rating Sum of Boxes |
| CFR | US Code of Federal Regulations |
| ChEls | Cholinesterase-Inhibitors |
| CMRglu | Cerebral Metabolic Rate for glucose |
| CNS | Central Nervous System |
| CRF | Case Report/Record Form (paper or electronic) |
| CRO | Contract Research Organization |
| CRS | Case Retrieval Sheet |
| CSF | Cerebrospinal fluid |
| CSR | Clinical Study report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CTC | Common Toxicity Criteria |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DDI | Drug-Drug-Interaction |
| DMC | Data Monitoring Committee |
| DNA | Deoxyribonucleic Acid |

| DSPP | Development Safety Profiling Plan |
|---|---|
| DTI | Diffusion Tensor Imaging |
| ECG | Electrocardiogram |
| ECog | Everyday Cognition scale |
| eCRF | Electronic Clinical Report Form |
| EDC | Electronic Data Capture |
| ELISA | Enzyme Linked Immunosorbent Assay |
| ELISPOT | Enzyme-Linked ImmunoSpot |
| EoS | End of Study |
| FAS | Full Analysis Set |
| FIH | First-in-human |
| FLAIR | Fluid-Attenuated Inversion Recovery |
| GCP | Good Clinical Practice |
| HA | Health Authorities |
| Hb | Hemoglobin |
| HMs | Homozygotes |
| i.m | Intramuscular |
| i.v. | Intravenous |
| IA | Interim Analysis |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use |
| IEC | Independent Ethics Committee |
| IES | Impact of Events Scale |
| IgG | Immunoglobulin G |
| IGT-AD | Impact of Genetic Testing for Alzheimer's Disease |
| IPW | Inverse Probability Weighting |
| IRB | Institutional Review Board |
| IRT | Interactive Response Technology |
| IVR | Interactive Voice Response |
| IWR | Interactive Web Response |
| LDH | Lactate Dehydrogenase |

| LFT | Liver Function Test |
|---------|-----------------------------------------------------|
| LLOQ | Lower Limit of Quantification |
| LOAD | Late Onset Alzheimer's Disease |
| MAR | Missing at Random |
| MCI | Mild Cognitive Impairment |
| MedDRA | Medical Dictionary for Drug Regulatory Affairs |
| MFAS | Modified Full Analysis Set |
| MMRM | Mixed Model Repeated Measure |
| MMSE | Mini-Mental State Examination |
| MRI | Magnetic Resonance Imaging |
| MTD | Maximum Tolerated Dose |
| NCI | National Cancer Institute |
| non-HMs | non-Homozygotes, i.e. Heterozygotes or non-carriers |
| NYHA | New York Heart Association |
| o.d. | Once Daily |
| OC/RDC | Oracle Clinical/Remote Data Capture |
| OS | Overall Survival |
| p.o. | Oral (per os) |
| PAC | Progression Adjudication Committee |
| PBMC | Peripheral Blood Mononuclear Cells |
| PET | Positron Emission Tomography |
| PFS | Progression-Free Survival |
| PPS | Per-Protocol Set |
| PPW | Premature Participant Withdrawal |
| PRO | Patient Reported Outcomes |
| PS | Propensity Score |
| PT | Preferred Term |
| PT-INR | Prothrombin Time-International Normalized Ratio |
| q.d. | Quoque die (once each day) |
| qd | Qua'que di'e / once a day |
| QTcF | Fridericia QT correction formula |

| RAP | Report and Analysis Process |
|---|---|
| RBANS | Repeatable Battery for the Assessment of Neuropsychological Status |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| REVEAL | Risk Evaluation & Education for Alzheimer's Disease |
| RNA | Ribonucleic Acid |
| ROI | Region of Interest |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SMQ | Standardized MedDRA Query |
| SOC | System Organ Class |
| SR/NR | Serological Responders/ Serological Non-Responders |
| SSRI | Selective Serotonin Re-uptake Inhibitor |
| STAI-AD | State Trait Anxiety Inventory for AD |
| SUV | Standardized Uptake Value |
| SUVR | Standardized Uptake Value Ratio |
| SD | Standard Deviation |
| TBL | Total Bilirubin |
| TE | Target Engagement |
| TFLs | Tables, Figures, Listings |
| TTE | Time-To-Event |
| ULN | Upper Limit Of Normality |
| VAS | Visual Analogue Scale |
| WHO-DD | World Health Organization Drug Dictionary |
| γ-GT | Gamma-Glutamyl Transferase |

## 1 Introduction

The intention of this document is to describe main efficacy and safety analyses of Cohort I of Generation Study CAPI015A2201J investigating CAD106 versus placebo (short Cohort I CAD106). The Cohort I CAD106 has been terminated prematurely as per Investigator Notification dated 23-Sep-2019. After study initiation, a halt of recruitment was introduced to

Cohort I when 65 participants were randomized in 2017 (see protocol amendment #4). Due to the early termination, only an abbreviated Clinical Study Report (a-CSR) will be created for Cohort I. This SAP will not cover the analysis of genetic disclosure (GD) follow-up. GD follow-up data will be reported in the CAPI015A2201J Cohort II a-CSR. The content of this SAP is based on the final amendment version 6.0 of protocol CAPI015A2201J.

#### 1.1 Study design

#### 1.1.1 Study Design Summary

This study protocol has multiple epochs with two informed consents required:

- 1. Pre-screening Epoch and Genetic Disclosure Follow-up (Informed consent #1)
- 2. Screening, Treatment and Follow-up Epochs (Informed consent #2).

This SAP will mainly focus on reporting data from Treatment and Follow-up Epochs. Prescreening and Screening Epoch will only be shown on disposition tables.



#### 1.1.2 Planned Number of Participants

In the original plan, Cohort I participants are planned to be treated for at least 60 months up to a maximum of 96 months to access of efficacy for the investigational treatment CAD106. The Treatment Epoch followed a randomized, double-blind, placebo-controlled parallel group

design in which participants receive the investigational treatment or matching placebo. Overall, sample sizes of 430 participants in the active treatment arm CAD106, and 260 in the matching placebo arm were planned. In 2017 a halt was introduced to Cohort I when 65 participants are randomized. Therefore, the CAD106 (Cohort I) data contains only 65 ongoing participants and the analysis will be mainly based on the 65 participants.



#### 1.1.4 Primary Analysis Time Point

There are two primary endpoint variables: time to first diagnosis of MCI due to AD or dementia due to AD (TTE), and the APCC test score. TTE will be analyzed only after the target number of events has been observed. The APCC score is analyzed after all participants have completed 60 months follow-up.

#### 1.1.5 Interim Analyses

The main purposes of the planned analyses during the course of the trial are safety monitoring by the DMC and assessment of futility with the potential consequence of discontinuing a futile active treatment arm and the corresponding placebo.

Interim Analyses are planned at various stages throughout the trial.

- 1. Safety monitoring
  - Regular semi-annual evaluation of safety parameters, worsening in cognition as a safety measure together with data allowing risk/benefit assessment to be defined with the DMC
  - Safety monitoring of T-cell activation data of n = 50 participants in Cohort I
- 2. Unblinded futility IA of Immunogenicity of CAD106
- 3. CNS activity based on biomarkers when a pre-defined number of participants reach 24 months.
  - Cerebrospinal fluid (CSF): tau pathology (tau and p-tau)
  - PET imaging data: amyloid,


- Blood/CSF NFLs
- 4. Primary endpoints: Analyses of Primary efficacy parameters (TTE and APCC) when a sufficient number of events are observed to assess futility or stopping due to overwhelming efficacy.

#### 1.2 Study objectives and endpoints

The original planned primary objective and all other key secondary, secondary and other efficacy objectives aimed to evaluate effects of CAD106 versus Placebo by comparing changes from baseline to Month 60 (reference to v06 of protocol CAPI015A2201J section 2). Due to the early termination of CAD106, no data have been collected at Month 60. Some participants have provided data on active treatment with CAD106 beyond one year of follow-up. Hence, the originally planned inferential and model based statistical analyses cannot be performed and are no longer applicable.

#### 2 Statistical methods

Due to the premature termination of the study, the originally planned inferential statistical analyses comparing efficacy readouts at Month 60 across treatment groups will not be conducted, but data collected on primary, secondary and other efficacy variables will be reported descriptively.

All the efficacy and biomarker endpoints except for events and TTE itself will be summarized using descriptive statistics by treatment groups as follows

- Raw values by visit including the TEC and the end of study visit (EoS) follow-up visit
- Change from baseline by visit including TEC and EoS

Subgroup of Amyloid level will be applied to all reports based on efficacy and biomarker endpoints except for time to events

Amyloid level (A+/A-). Definition of Amyloid level is in Section 2.7.

#### 2.1 Data analysis general information

The statistical analysis will be performed by Novartis internal statisticians and programmers.

Unless otherwise stated, summary tables/listings/figures will be presented by treatment group in the respective analysis set. Tables showing only baseline data will also include a total column.

Categorical data will be summarized as frequencies and percentages. Percentages will be calculated as below:

- For population level summaries (like AEs, Medical history...etc.), percentages will be calculated using number of participants in each treatment group as the denominator.
- For by visit summaries (including baseline demographic), percentages will be calculated using the number of participants in the analysis set with an assessment at the specified visit as the denominator.
- For specific event based summaries, the denominator will only include the subset of the analysis population of participants at risk at a specific point in time (Kaplan-Meier approach).

Continuous data will be summarized by presenting the number of non-missing observations, mean, standard deviation (SD), median, minimum and maximum, both for raw (absolute) values and for changes from baseline. Summary tables will be presented wherever applicable by visit if not otherwise specified.

Specified parameters of interest will be listed by treatment group, records will be ordered by country/center/participant and time of assessment.

General information on treatment group labels, decimal places and other output related information will be specified in the specification document for tables, figures and listing (TFLs) shells accompanying this analysis plan.

Statistical analysis will be performed using SAS® statistical software (SAS Institute, Cary, NC, USA.) version 9.4 or higher.

#### 2.1.1 General definitions

#### Study Drug

Study drug refers to the administration of either CAD106 450 µg (quarterly i.m.) with Alum or matching placebo with Alum in Cohort I (referred to as CAD106 or CADPBO respectively).

#### **Date of First Study Drug Administration of (Day 1)**

Day 1 is defined as the first day of randomized study drug administration. All other days will be labelled relative to Day 1. For event dates on or after Day 1, study day for an event date is calculated as (event date – first dose date + 1) which could be Day 2, Day 3 etc. For event dates before Day 1, study day for an event date is calculated as (event date – first dose date), which could be Day -1, Day -2, etc., referring to one day, two days, etc., before Day 1, respectively. Thus, Day -1 is the day preceding Day 1. Day 0 is not defined.

#### **Date of Last Study Drug Administration**

The date of last study drug administration is the day of the last dose of study drug.

#### **Baseline**

A baseline value refers to the last (most recent) evaluable measurement prior to the first administration of study drug. Typically, baseline values will be the values obtained on the day of randomization. If the Baseline visit is missing or the assessment was not done at Baseline, the last assessment of an earlier visit (scheduled or unscheduled) which is closest to the Baseline visit will be used as Baseline value. In case an assessment is repeated at a later visit during the screening epoch, the latest one will be used as Baseline value.

Note: Assessments at the day of randomization are assumed to have been taken as per protocol, i.e. if the assessment should be performed before dosing, the assessment will be treated as predose as per protocol. Practically, i.e. that the time part of the date/time entry (when collected) will be ignored. Exception: In case there is a protocol deviation or a comment that specifically indicates that the assessment has been taken post-dose, the assessment will not be handled as pre-dose.

#### Post-baseline

For safety and efficacy evaluations, all assessments after Day 1 are defined as post-baseline assessments.

#### Re-screened participants

Participants who screen-failed due to a temporary condition (e.g. physical, concomitant medications, etc.) or due to administrative reasons may be re-screened after resolution. The participant will receive a new subject identifier at re-screening. The latest screening assessment will be considered for reporting at screening visit. Assessments (like genotype, volumetric MRI, etc.) that are not repeated, will be carried over. This is based on mapping the old subject identifier to the new subject identifier.

In general, all data collected under the old subject identifier is kept after mapping to the new subject identifier. This comprises for instance AEs, vital signs, ECG, and laboratory data. In case of missing values under the new subject identifier, the latest available value from the old subject identifier will be used. In study Cohort I, the earliest consent date is kept, if the subject is re-screened.

#### **Prior and Concomitant Medication**

Prior medication will be defined as any medication taken prior to the first dose of the study drug, irrespective of whether the medication continued into the treatment period.

Any medication administered at least once between Day 1 and end of the study is defined as concomitant medication.

#### **Visit Windows**

In general, by-visit analyses will include data from scheduled as well as un-scheduled visits using visit windows for scheduled visits except for TEC/PPW and EoS. In general, the lower and upper bound of a visit window will be defined as the midpoint between scheduled visits. The visit window rules for efficacy and safety parameters are defined in Appendix 5.7.

For efficacy parameters: In case of competing assessments within a visit window, the assessment value closest to the scheduled visit day will be used. In case of equal distances, the earliest assessment value will be used. Visit window will not be applicable for TEC/PPW and EoS.

For safety parameters: In case of competing assessments within a visit window, the worst assessment value within the visit window will be used.

Listings will include all assessments, sorted by date of assessment, flagging unscheduled visits. The listings will include analysis windows and corresponding flags to indicate the assessment's inclusion in the analysis.

# Treatment Epoch Completion (TEC) and End of Study (EoS) and other points in time of interest

TEC is the end of treatment phase visit (i.e., visit 399) that will be completed for all participants after discontinuation of treatment. The same visit will also be completed in case of PPW. PPW is the premature study withdrawal.

EoS (visit 401) is a Follow-up visit scheduled after TEC/PPW, per urgent safety measure (USM) on 23-Sep-2019. 3 months are expected between TEC and EoS. Participants who were attending study visits (i.e., continuing in the study) but already off-treatment at time of USM were to come for EoS straight (no TEC required).

"Last assessment" is defined as the last post-baseline assessment across all visits including TEC and EoS. "Last assessment" may be different for different variables. This concept is applied for cognitive and biomarker endpoints to summarize changes at maximum exposure regardless of on/off treatment. This is due to the fact that CAD106 has long half-lives so that it's valid to assume all post-baseline assessments are on treatment. Note that, "last assessment" is a mixture of scheduled visits and TEC and/or EoS. In order to better understand the timing of "last assessment", summary tables and frequency tables will be provided for variables of RBANS and volMRI.

### 2.2 Analysis sets

The following analysis sets will be used.

The **Randomized analysis set (RAS)** will consist of all participants who received a randomization number, regardless of receiving study medication.

The Safety analysis set (SAF) will consist of all participants who have received study medication.

Note: The above SAF definition is different from the protocol defined SAF definition which restricts to include only those participants in SAF if they have had at least one safety assessment after first dose administration.

All efficacy analyses and safety analyses will be conducted on the SAF.

In addition, the following sets of participants will be used to understand the composition of analysis sets and disposition of participants.

**Screened set** will consist of all participants (HMs only) who have signed ICF#2 and proceeded into Screening epoch.

#### 2.2.1 Subgroup of interest

Subgroup of Amyloid level will be applied to all the efficacy (except for TTE) and biomarker endpoints on top of the by treatment groups:

• Amyloid level (A+/A-). Definition of Amyloid level is in <u>Section 2.7</u>.

# 2.3 Patient disposition, demographics and other baseline characteristics

Summary tables for demographic variables and other baseline characteristics as well as relevant medical history will include a total column in addition to the treatment arms.

#### 2.3.1 Patient disposition

The number and percentage of participants in each analysis set described above will be presented including all participants that started screening. Primary reason for screen failure will be summarized for all participants.

Participant disposition will be summarized for the RAS showing the flow of participants through the treatment epoch and completing the End of Study disposition page. The disposition summary will show the number and proportion of participants who discontinued treatment epoch and End of Study status along with the reason for discontinuation. The number and proportion of participants with missing End of Study assessment will also be reported. The primary reasons for premature discontinuation of study treatment will also be summarized. Listings will be provided showing the primary reason for premature discontinuation of study and of study treatment.

All the important protocol deviations reported during the study will be summarized in the following five categories:

- Selection criteria not met
- Subject not withdrawn as per protocol
- Treatment deviation
- Prohibited concomitant medication
- Other deviations (important deviations that do not fall in the above four categories)

Important PDs are defined as subset of PDs that may significantly impact a subject's rights, safety, and well being or the completeness, accuracy, and/or reliability of the study data. The PD codes to identify the above categories are listed in Table 5-4 in the Appendix.

#### 2.3.2 Background and demographic characteristics

The following demographic and baseline variables will be summarized on the SAF. No listings will be provided.

#### **Demographic variables:**

**Continuous variables:** 

- Age (years)
- Height (cm)
- Weight (kg)
- BMI (kg/m<sup>2</sup>) will be calculate as (body weight in kilograms) / (height in meters)<sup>2</sup>
- Volumetric MRI-Whole Brain (cm<sup>3</sup>)

- Volumetric MRI-Hippocampus (cm<sup>3</sup>)
- Centiloid

#### Categorical variables:

- Age group (<=64, 65-69, >=70)
- Sex (Male, Female)
- Years of education (<=12 years, 13-16 years, >= 17 years)
- BMI (< 25 vs >= 25)
- Race (Caucasian, Black, Asian, Native American, Pacific Islander, Other, Unknown)
- Ethnicity (Hispanic or Latino, Other East Asian, Southeast Asian, South Asian, West Asian, Russian, Japanese, Chinese, Mixed Ethnicity, Other, Unknown, Not reported)
- Amyloid level (Positive/ Negative)
   Amyloid level will be derived using PET and CSF criteria described in <u>Table 2-1</u>.

#### Cognitive scales at baseline

#### Continuous variables:

- MMSE
- RBANS Total score
- Immediate Memory Index
- Delayed Memory Index
- Visuospatial/constructional Index
- Language Index
- Attention Index
- CDR-SOB

#### Categorical variables:

• CDR Global (Score = 0, Score = 0.5, Score > 0.5)

Comparability of randomized groups (active versus placebo) at baseline will be assessed via Fisher's exact tests for  $2\times2$  tables or the corresponding Freeman-Halton test for general  $1\times k$  tables (1,k>=2) for selected categorical variables. If Fisher's exact tests are not estimable (e.g. sample size is too large to calculate the statistic) or not adequate, then Chi-squared tests will be performed. Baseline comparability for selected continuous variables will be assessed using t-tests assuming unequal variances in the two groups (active versus placebo). The tests performed together with the test statistic and the p-value will be reported for each baseline variable that has been investigated for comparability. The selected variables for comparisons will be indicated in the TFL shells.

#### **Medical history**

Any condition entered as medical history or current medical conditions at baseline will be coded using the MedDRA dictionary effective at the time of the database lock and summarized by system organ class (SOC) and preferred term (PT) on the SAF. No listing will be provided.

# 2.4 Treatments (study treatment, rescue medication, concomitant therapies, compliance)

#### 2.4.1 Study treatment / compliance

#### **Duration of Exposure**

The duration of exposure to study drug is defined as the time (in days) from the first study drug administration to last study drug administration + 180 days.

The duration of exposure will be calculated as

(last dose date + 180 days) – first dose date + 1

Duration of exposure to CAD106 will be summarized as continuous variable (in days) and categorical variable, using categories >=1 day (any exposure), >= 6 months, >=1 year, >= 1.5 years, >=2 years, >=2.5 years and >=3 years.

The participant-years will be calculated as

(sum of the durations of exposure for all participants in the group)/365.25) and will be summarized.

For each treatment group, summary statistics will be presented by subgroups A+ and A- as defined in Table 2-1.

#### 2.4.2 Prior, concomitant and post therapies

The number and percentage of participants receiving concomitant medications will be summarized on the SAF by ATC class and preferred term (according to the latest World Health Organization drug dictionary (WHO-DD) at the time of database lock, including Anatomical Therapeutic Chemical (ATC) classification code).

The number and percentage of participants receiving significant non-drug therapies will be summarized on the SAF by primary system organ class, preferred term (according to the latest MedDRA dictionary version available at the time of database lock).

### 2.5 Analysis of the primary objective

#### 2.5.1 Primary endpoint

There are two primary endpoint variables:

- Time-to-event (TTE), with an event defined as a confirmed diagnosis of MCI due to AD or dementia due to AD (whichever occurs first), and
- Change in the API preclinical cognitive composite (APCC), from baseline to Week 260 (M 60)

Due to the early termination of the study, only a small number of events following the TTE definition have been observed, and reporting change in APCC 60-month from baseline is no longer applicable. Hence, for the abbreviated CSRs, events and APCC will be summarized based on data availability.

#### Time to event (MCI due to AD or dementia due to AD)

Time-to-event (TTE), with event defined as the first confirmed diagnosis of MCI due to AD or dementia due to AD (whichever occurs first). An event is identified as a Progression Adjudication Committee (PAC)-confirmed diagnosis triggered either by an investigator diagnosis or an increase in the CDR global score. The confirmation by the PAC consists of two confirmed adjudications based on data from two consecutive visits.

In case of an identified event, TTE will be calculated as the time from randomization to the first confirmed diagnosis. For each event (confirmed diagnosis), the date of the initial investigator diagnosis will be used to establish the date of the event (neither the date of adjudication, nor the date of the confirmation). In case no confirmed event has been observed for an individual, the observation will be censored, and the censoring date will be defined as the last date where the diagnosis classification has been assessed. Time to censoring date will be calculated from day of randomization.

The team agreed on the LPLV date April 15, 2020 as the cut-off date/point for the final analysis. The final TTE analysis will include data until this cut-off point. Any data collected after this cut-off point will not be used for the primary analysis of TTE. That means specifically that only confirmed events collected up to the data cut-off point will be counted. Confirmation information collected after the cut-off point to confirm an earlier (meaning before the cut-off point) adjudicated diagnosis of MCI or AD due to dementia will not be taken into consideration. As a consequence, the observation will be censored at the last date prior to cut-off point that the TTE endpoint was evaluated, and the unconfirmed diagnosis will not be counted as an event in the primary analysis.

Due to the early termination of the studies, only a small number of events following the above definition have been observed. Hence, for the abbreviated CSR, the number (%) of participants meeting the following additional situations (change in diagnosis classification) will also be reported:

- 1. Participants with a change in diagnostic classification from cognitively unimpaired by the principal investigator at any time
  - MCI due to AD.
  - MCI not due to AD,
  - Dementia due to AD,
  - Dementia not due to AD.
- 2. Participants with an increase in CDR global score from baseline at any time (any increase, increase less than 1, increase of 1 or more).
- 3. Participants where data was sent for adjudication to PAC (regardless of confirmation at the following visit) split by the result of the adjudication:
  - Cognitively unimpaired,
  - MCI due to AD,
  - MCI not due to AD,
  - Dementia due to AD,
  - Dementia not due to AD,

• Other (Unable to adjudicate, data not collected, not known).

Note that cut-off date/point (16 APR 2020) used for protocol defined event (MCI due to AD or dementia due to AD) will not be applicable for the above defined additional situations. Data up to the database lock date will be used for the analysis of these additional events.

#### **APCC** score

The API preclinical cognitive composite (APCC) test score is defined as a weighted sum of the following test items:

- Raven's Progressive Matrices sum of subset items A2, A4, A8 & B1-B6 (0-9)
- MMSE:
  - Orientation to Time (0-5)
  - Orientation to Place (0-5)
- RBANS (Subtest raw scores):
  - List Recall (0-10)
  - Story Recall (0-12)
  - Coding (0-89)
  - Line Orientation (0-20)

The range of the APCC test score is from 0 to 100 where higher scores in the APCC correspond to a better cognitive performance. The APCC will be derived based on the test items using the below formula and weights:

APCC test score = 1.360×RBANS List Recall + 1.100×RBANS Story Recall +1.390×Raven's Progressive Matrices (subset items A2, A4, A8, B1-B6) + 0.321×RBANS Coding + 0.510×RBANS Line Orientation + 2.140×MMSE Orientation to Place + 2.240×MMSE Orientation to Time.

#### 2.5.2 Statistical hypothesis, model, and method of analysis

Except from the primary objective on the TTE endpoint, the other primary objective (for APCC) aimed to evaluate effects of CAD106 versus Placebo by comparing changes from baseline to Month 60. Due to the early termination of CAD106, no data have been collected at Month 60. Only very few participants have provided data on active treatment with CAD106 beyond one year of follow-up. Hence, the originally planned inferential and model based statistical analyses cannot be performed and are no longer applicable.

The subgroup of Amyloid level will be applied to all the efficacy (except for TTE) endpoints:

• Amyloid level (A+/A-). Definition of Amyloid level is in Section 2.7.

#### Time to event (MCI due to AD or dementia due to AD)

#### **Tables**

Time to Event analysis using Kaplan Meier approach will be presented for time to MCI due to AD or Dementia due to AD (events as per protocol) and for time to first change in diagnostic classification (this is an event regardless of confirmation and adjudication) from cognitively

unimpaired by the investigator. The Kaplan-Meier estimates of the cumulative event rate for each treatment group will be summarized and plotted. To calculate the proportion of participants with events, number of participants at risk will be used as the denominator. "Participant at risk" at a specific time point is defined as the number of participants in the study without an event at up to that time point.

These analyses will only be performed if there are at least five such events.

In addition, the number and percentage of the additional situations (Section 2.5.1) defined events overall (not by visit) will be summarized by treatment group.

#### **APCC** score

#### **Tables**

The APCC test score and the seven components (listed above in <u>Section 2.5.1</u>) will be summarized on the SAF by visit as well as last assessment. Last assessment is defined as the last assessment post baseline.

#### **Figures**

- Plot of raw values for APCC over time (including baseline and all post-baseline visits) with smoothing curve
- For APCC, effect sizes of change from baseline as well as 80% confidence intervals (CIs) for the effect size will be reported. The effect size (and CI) of change from baseline will be calculated for following post-baseline visits: Week 26 and Week 52, Week 78, Week 104, TEC, and EoS and last assessment.

The effect size will follow the Cohen's d formula: The raw mean to standard deviation ratio, not model based mean to standard deviation ratio. The effect size will be calculated as the difference between active and placebo in mean change from baseline divided by the pooled standard deviation of the change. Effect sizes and CIs will be calculated (active versus placebo).

#### Derivation of study specific effect size d and corresponding CI

BL = Baseline value; PBL= Post baseline value;

SD = Standard deviation; SE = Standard error;  $n_1$  = Sample size group 1;  $n_2$  sample size group 2;  $S_1^2$  = Variance group 1;  $S_2^2$  = Variance group 2

Numerator: Mean change from BL to PBL active – mean change from BL to PBL control

Denominator: pooled SD defined as

$$SD_{pooled} = \sqrt{\frac{(n_1 - 1)S_1^2 + (n_2 - 1)S_2^2}{n_1 + n_2 - 2}}$$

Where the groups are given by factor treatment (active versus control).

The confidence interval can be derived using the formula proposed by Hunter and Schmidt 2004 and Nakagawa and Cuthill (2007):

$$CI: d \pm z * SE(d)$$

Where z is the 10% Quantile of the normal distribution in case of the 80% CI. The SE(d) is calculated as

$$SE_d = \sqrt{\frac{(n_1 + n_2 - 1)}{(n_1 + n_2 - 3)} \left[ \left( \frac{4}{n_1 + n_2} \right) \left( 1 + \frac{d^2}{8} \right) \right]}$$

### 2.5.3 Handling of missing values/censoring/discontinuations

# Time to event (MCI due to AD or dementia due to AD) and Time to first change in diagnosis classification

In general, an observation will be censored if no event has been observed at the TTE analysis cut-off date. The censoring date will be defined as the last date (before cut-off date) where the TTE endpoint has been assessed.

The censoring date for each participant that did not have an event (i.e., a confirmed diagnosis) is defined as follows:

- 1. For participants ongoing in the study without a confirmed diagnosis at the time of the cutoff: the last day of a diagnosis assessment (the previous visit where a diagnosis assessment occurred prior to the cut-off date).
- 2. For participants who permanently discontinued from the study prior to the cut-off: The last day of a diagnosis assessment prior to study discontinuation.
- 3. For participants who had their last diagnosis assessment prior to randomization (i.e. during screening epoch) or do not have any diagnosis assessment post randomization, their randomization date will be used as censoring date.

Note: For Time to MCI due to AD or dementia due to AD, the cut-off date will be 15 April 2020. For Time to First change in diagnosis classification, the cut-off date will be database lock date.

Further details on derivation of events and censoring will be added to the programming document specifications (PDS).

#### Other primary efficacy endpoint variable (APCC)

Due to the early termination of the trial, analyses of primary efficacy variable APCC will in general be based on observed cases only, i.e. there will be no imputation of missing data. Exception in primary efficacy variable APCC applies to missing data in subtests of Raven's matrices included in the primary efficacy variable APCC. Missing values for the subtests of Raven's matrices of the APCC may be imputed using the imputation rule defined in Appendix 5.1.3.3.1.

#### 2.5.4 Supportive analyses

Not applicable.

### 2.6 Analysis of the key secondary objective

#### 2.6.1 Key secondary endpoint

The key secondary endpoint variable is Clinical Dementia Rating Scale Sum of Boxes (CDR-SOB).

#### Clinical Dementia Rating (CDR) global and Sum of Boxes (CDR-SOB)

The CDR is obtained through semi-structured interviews of participants and informants, and cognitive functioning is rated in six domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a 5-point scale of functioning as follows: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). The CDR global score ranges from zero to three, with greater scores indicating greater disease severity. The CDR-SOB is defined as the sum of the ratings from the six domains, ranging from 0 to 18 with a minimum increment of 0.5. A higher CDR-SOB score indicates greater disease severity.

#### 2.6.2 Statistical hypothesis, model, and method of analysis

The key secondary objective aimed to evaluate effects of CAD106 versus Placebo by comparing changes from baseline to Month 60. Due to the early termination of CAD106, no data have been collected at Month 60. Only very few participants have provided data on active treatment with CAD106 beyond one year of follow-up. Hence, the originally planned inferential and model based statistical analyses cannot be performed and are no longer applicable.

The subgroup of Amyloid level will be applied to all the efficacy (except for TTE) endpoints:

• Amyloid level (A+/A-). Definition of Amyloid level is in <u>Section 2.7</u>.

#### **Tables**

CDR-SOB and CDR global will be summarized on the SAF.

#### 2.6.3 Handling of missing values/censoring/discontinuations

Due to early termination of the trial, analyses of CDR-SOB will be based on observed cases only, i.e. there will be no imputation of missing data.

### 2.7 Analysis of secondary and other efficacy objective(s)

#### 2.7.1 Secondary and other efficacy endpoints

#### **RBANS Total score and Index scores**

The RBANS is comprised of the following five neurocognitive domains, with associated subtests used for Index scores:

- Immediate Memory List Learning and Story Memory (IMI)
- Visuospatial/Constructional Figure Copy and Line Orientation
- Language Picture Naming and Semantic Fluency
- Attention Digit Span and Coding
- Delayed Memory List Recognition and Sum of (List Recall, , Story Recall, and Figure Recall; DMI)

The RBANS generates age-adjusted index scores for five neurocognitive domains, which are used to calculate a Total Scale Index score using norm tables for each Index scores in Appendix 5.8. The algorithm (by vendor) to derive index scores is based on the current actual age of the participant. For longitudinal analyses, this approach creates artificial variability. As a consequence, the derived data for index scores will not be used in the analyses, but will be derived from source data using the age at screening for adjustment for all assessments. The algorithm to derive the Index scores using age at baseline will be described in the programming specifications (PDS) of this study.

A higher RBANS score indicates better cognitive function.

#### Mini Mental State Examination (MMSE)

The MMSE is a brief, practical clinician reported outcome that examines cognitive status (Folstein et al., 1975). It evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, and the ability to create a sentence and copy two intersecting pentagons. The test consists of five domains (orientation, registration, attention, recall, and language) with a total score ranging from zero to 30. A higher score indicates better cognitive function. The five sub scores as well as the total score will be recorded.

#### **Raven's Progressive Matrices**

Raven's Progressive Matrices (<u>Raven et al 2000</u>) is a non-verbal, multiple choice measure of general ability and reasoning using a visual modality. It was designed to be culturally nonbiased, as neither language nor academic skills are required to answer items successfully.

Although all components of the Raven's Progressive Matrices Set A and Set B will be assessed, in order to calculate the APCC test score, only a subset of items from Sets A and B will be used (items A2, A4, A8, B1-B6), with a range from zero to nine.





#### **Everyday Cognition scale (ECog-Participant and ECog-Informant)**

The ECog scale measures cognitively-relevant everyday abilities and is comprised of 39 items covering six cognitively-relevant domains: Everyday Memory, Everyday Language, Everyday Visuospatial Abilities, Everyday Planning, Everyday Organization, and Everyday Divided Attention (Farias et al 2008). Within each domain, the ability to perform a specific task is rated on a five-point scale ranging from: 1) no difficulty, 2) mild difficulty, 3) moderate difficulty, 4) severe difficulty, or 5) unable to do. The scale has 2 versions one for patient (PRO) and one for informant (study partner).

The total score for the 39 items ranges from 39 to 195, with greater scores indicating worse daily function.

#### Volumetric MRI

Screening (baseline) volumetric measurements are performed using FreeSurfer software. This leads to reference volumes for whole brain, ventricles, hippocampus, and intra-cranial.

Volumetric data will be available for the following regions:

- intra-cranial volume (ICV),
- total/whole brain,
- left/right hippocampus,
- lateral ventricles.

In order to assess atrophy rate, volumetric MRI images from follow-up time points are compared to those from screening, using the boundary shift integral (BSI) technique in selected brain regions. The technique determines the total volume through which the boundaries of a given cerebral structure have moved, and hence, it aims at quantifying the amount of change in these selected brain regions. The output of the method is a change from baseline in volume (atrophy).

Volume changes in the following regions of interest (ROI) will be reported:

- whole brain,
- hippocampus (sum of left and right),
- lateral ventricles (left and right).

Data provided by vender will be:

- Baseline volume (absolute volume)
- Post-baseline atrophy from baseline

As the absolute volume for post-baseline visits is not provided directly by vender. Post-baseline volume will be derived using baseline volume and atrophy.

#### Biomarkers in Cerebrospinal Fluid (CSF)

The following AD related markers in CSF are analyzed:

- total-tau and phospho-tau (p-tau)
- $A\beta 1-40$  and  $A\beta 1-42$

#### Biomarkers in blood:

- Plasma Abeta-40
- Serum Light Chain Neurofilaments (NFL)

Values below the lower limit of quantification (LLOQ) will be set to LLOQ/2 for statistical analysis, values above upper limit of quantification (ULOQ) will be imputed with ULOQ. LLOQ and ULOQ value may differ across samples according to the dilution factor applied in the specific sample. For statistical analysis, the sample specific LLOQ and ULOQ value should be used.

#### Positron Emission Tomography (PET) Standard Uptake Value Ratio (SUVR)

Across the three F<sup>18</sup> amyloid binding radiotracers used Florbetapir (FBP), Florbetaben (FBB) and Flutemetamol (Flute): Centiloids using the agreed formulae

For participants who consent to the voluntary AD-related imaging biomarker evaluations, regional activity concentration and the cortical Standardized Uptake Value (SUV) are measured based on the following brain regions of interest (ROIs):

- Parietal cortex
- Posterior cingulate or Precuneus
- Medial orbitofrontal cortex
- Anterior cingulate
- Temporal cortex

and the whole cerebellum as reference region.

Data for regional activity concentration will not be reported.

Neocortical composite is the composite score of other individual ROIs with whole cerebellum is the reference region, and will be summarized for Cohort I. The *global* cortical amyloid load will be derived as the unweighted average cortical Standardized Uptake Value Ratio (SUVR) between the cortical ROIs and the reference region.

#### Standardized Uptake Value Ratio (SUVR) values

For Amyloid PET, the baseline load obtained from different tracers (florbetapir (FBP), flutemetamol (Flute) and florbetaben (FBB)) will be converted to a standardized Centiloid scale. The conversion equation for each tracer has been obtained following a non standard analysis method (AVID method) based on level-1 (GAAIN, Klunk et al. Centiloid values) and level-2 (InVicro Centiloid values) as documented in the Image Analysis charter from InVicro:

$$CL = 183.00 * SUVr_{FBP} - 176.97$$
  
 $CL = 123.90 * SUVr_{Flute} - 114.86$   
 $CL = 156.06 * SUVr_{FBB} - 148.132$ 

The reference is Klunk et al., 2015. The % change in SUVR will be calculated as

$$\%Change = \frac{(SUVR_{FU} - SUVR_{BL})}{SUVR_{BL}} \times 100\%$$

with SUVR<sub>BL</sub> as the baseline value and SUVR<sub>FU</sub> the SUVR value at follow-up visit.

#### Analysis of positive/negative amyloid levels

Amyloid level (positive/negative) is measured at screening by two methods:

- CSF collection via Lumbar puncture
- Brain Amyloid PET radiotracers (amyloid PET: SUVr)

The studies allow either method for determination of amyloid level. CSF samples are collected and analyzed using selected validated assay. The cut-off value to determine the amyloid level as positive/negative will depend on the assay selected. The criteria for positive amyloid level in CSF is based on pTau/Ab42 ratio. The criteria for positive amyloid PET will follow specifications for the specific radiotracer used. Following Table 2-1 describes the cutoffs for both methods.

Centiloid value  $\geq$  24.33 is considered as A+ regardless of tracer type. This value is roughly equivalent to a florbetapir SUVR of 1.17. The definition of Amyloid positivity based on Centiloid cut-off is equivalent to SUVr approach, though scales are different.

Table 2-1 Amyloid Level Stratification Criteria

| Metho | ods | Positive(A+) | Negative(A-) |
|---|---|---|---|
| CSF | | • Elecsys ratio p-Tau/ Aβ1-42> 0.024 | • Elecsys ratio p-Tau/ Aβ1-42≤ 0.024 |
| | | AND | OR |
| | | • Elecsys Aβ1-42≤ 1700.0 pg/ml (upper limit of the measuring range) | , |
| PET | Florbetapir (FBP) | SUVr_FBP ≥ 1.1 | SUVr_FBP < 1.1 |
| | Flutemetamol (Flute) | SUVr Flute ≥ 1.123 | SUVr Flute < 1.123 |

| Florbetaben (FBB) | SUVr FBB ≥ 1.105 | SUVr FBB <1.105 |
|-------------------|------------------|-----------------|

Analysis of Amyloid levels will be derived as Positive/Negative as described in Table 2-1 above. However, in the database, eligibility result for Amyloid status will be Elevated/Not-Elevated as provided by vendor. The Amyloid status flag is as reference only. For reporting and other publication exercise, the flag of Amyloid level (Positive/Negative) derived using the criteria above will be used.

#### A-beta-specific antibody titers for immunogenicity

The immune response based on antibody titer data will be performed in patients receiving CAD106.

A $\beta$ -antibody response is measured by determination of A $\beta$ -specific IgG titers in serum using enzyme-linked immunosorbent assay (ELISA) methods.

 $A\beta$ -IgG titers will be determined in serum at scheduled visits from Screening up to End of Study.  $A\beta$ -IgG titers measurement will be performed prior to the investigational drug injection (samples taken pre-dose) at scheduled visits.

#### 2.7.2 Statistical hypothesis, model, and method of analysis

The subgroup of Amyloid level will be applied to all the efficacy (except for TTE) endpoints:

• Amyloid level (A+/A-). Definition of Amyloid level is in <u>Section 2.7</u>.

#### **RBANS Total score and Index scores**

#### **Tables**

RBANS total score and RBANS Index scores will be summarized on the SAF by visit as well as last assessment.

#### **Figures**

- For RBANS total and RBANS index scores, effect sizes of change from baseline as well as 80% confidence intervals (CIs) for the effect size will be reported using Cohen's D as described in <a href="Section 2.5.2">Section 2.5.2</a>. The effect size (and CI) of change from baseline will be calculated for following post-baseline visits: Week 26 and Week 52, Week 78, Week 104, TEC, and EoS and last assessment.
- Plot of raw values for RBANS Total over time (including baseline and all post-baseline visits) with smoothing curve

#### **MMSE**

#### **Tables**

MMSE total score and the sub-scores on each of the five domains (orientation, registration, attention, recall, and language) will be summarized on the SAF by visit as well as last assessment.

#### **Raven's Progressive Matrices**

Raven's total score (sum of all items from Sets A and B) and the sub-score included in the APCC (sum of items A2, A4, A8, B1-B6) will be summarized on the SAF by visit as well as last assessment.

#### **Everyday Cognition scale (ECog-Subject and ECog-Informant)**

#### **Tables**

**Tables** 

ECog total score will be summarized on the SAF by visit as well as last assessment.

#### **Volumetric MRI**

#### **Tables**

Summary statistics for absolute change and percent change from Baseline to time point will be provided. All statistics will be based on the total volume, i.e. the sum of the respective left and right volumes as applicable.

Raw volumes, as well as changes, % changes, annualized changes, and annualized % changes from baseline will be summarized by visit as well as last assessment. Last assessment is defined as the last volMRI assessment post baseline. Calculation of annualized percent change from BL:

Individual patient annualized percentage change from BL in volMRI is calculated as (percentage change per patient / time interval (in days)  $\times$  365.25. Time interval will be derived as (date of current MRI assessment – date of baseline MRI assessment + 1).

Calculation of annualized change from BL:

Individual patient annualized change from BL in volMRI is calculated as (change per patient / time interval (in days) × 365.25. Time interval will be derived as (date of current MRI assessment – date of baseline MRI assessment + 1).

All biomarker data will be summarized by visit as applicable as well as last assessment. **Biomarkers in CSF** 

#### **Tables**

CSF Biomarkers will be summarized for baseline visit. Post baseline CSF biomarker will only be listed due to limited data.

#### Listings

For participants with post baseline CSF Biomarkers, baseline and post-baseline data will be listed.

#### Biomarkers in blood: serum Light Chain Neurofilaments (NFL)

#### **Tables**

Available measurements for NFL from serum will be summarized for actual values as well as for change from baseline.

Additionally, summary statistics will be presented after baseline outlier(s) being excluded. Outlier(s) will be identified based on pooled baseline data across CAD106 and placebo. The following quantities(fences) are needed for identifying outlier(s) in the tails of the distribution:

• lower outer fence: Q1 - 3\*IQ or

• upper outer fence: Q3 + 3\*IQ

Q1 (first quantile), Q3 (third quantile), and IQ (inter quantile: Q3-Q1) are needed for deriving the fences.

#### **Figures**

Box-plots for serum NFL over time by treatment group will be provided based on all available participants and without baseline outlier.

#### Biomarkers in blood: Plasma Abeta-40

#### **Tables**

Available measurements for Plasma Abeta-40 will be summarized for actual values as well as for change from baseline.

#### **Amyloid PET SUVr and Centiloid**

#### **Tables**

SUVr baseline, post-baseline, change, % change, annualized change, and annualized % change will be reported by ligand. Centiloid baseline, post-baseline, change, annualized change will be reported across all three ligands (% change will not be applied to Centiloid).

Post baseline visit includes week 104, TEC and last assessment. Last assessment is defined as the last amyloid PET assessment post baseline, which is pooling week 104 and TEC. For subject(s) who had both week 104 and TEC, the later one will be used to derive last assessment.

Calculation of annualized change from BL for centiloid:

Individual patient annualized change from BL in centiloid is calculated as (absolute change per patient / time interval (in days)  $\times$  365.25. Time interval will be derived as (date of current Amyloid PET assessment – date of baseline Amyloid PET assessment + 1).

#### **Figures**

Boxplot of annualized change in centiloid will be presented for last assessment by treatment group.

Scatter plot of annualized change in centiloids (last assessment) vs Baseline amyloid will be presented by treatment group.

#### Analysis of positive/negative amyloid levels

#### **Tables**

Amyloid levels (Positive/Negative) by method CSF and PET will be summarized as frequencies and percentages.

#### A-beta-specific antibody titers for immunogenicity

Note, the classification of responder status (in protocol) based on titer data up to week 26 is no longer valid because the data shows that titer concentration is still high after week 26. Protocol definition:

The classification of participants into serological responders (SR) and serological non-responders (NR) to CAD106 will be based on the individual CAD106-induced Aβ-specific IgG titer values in serum up to week 26. The classification rules have been developed on available data from previous Phase II studies. Participants of the CAD106 cohort will be classified in the following categories: SR, NR and Placebo. SR will be defined in the following way based on titer assessments: Participants whose Aβ-specific IgG titer in serum is greater than 16 units after 2nd and before 3rd injection AND greater than 3 times the LLOQ (LLOQ=8.93 units as determined in the phase II program, 3\*LLOQ=26.8 units) after the 3rd injection. NR will be participants that do not meet the SR definition.

For completeness, responder status along with other titer parameters will be reported, though it is acknowledged that responder status is not a valid parameter to draw any conclusions in this study.

The following parameters will be calculated:

- Responder status
- Cmax = Maximum Titer Concentration of any post-baseline "on treatment" visit
- Average Peak = Mean (Week 9, Week 15)
- Area under the curve (AUC): starting from baseline (zero concentration) and including all "on treatment" visits.

A visit is classified as "on treatment" if the assessment date is within {last injection date + 180 days}. For AUC calculation, in case of missing data, the following imputation rule will be applied:

- For missing trough values (NOT week 9 or 15), the average of non-missing "on treatment" trough values will be used to impute.
- For missing peak values (Week 9 and 15), no imputation will be done. Only interpolate the values to calculate AUC.

Titer values below the LLOQ were set to 0 for the computation of AUC.

The scheduled Titer assessments to be considered for deriving responder status, and average peak are as follows:

- Week 9 (two weeks after 2nd injection, expected to be a peak value) and Week 13 (before 3rd injection, trough value),
- Week 15 (two weeks after 3rd injection, expected to be a peak value) and Week 26 (before 4th injection, trough value).

The responder status, and average peak will be calculated for all participants having at least one available assessment for either Week 9 or Week 13 and at least one assessment for either Week

15 or Week 26. In case of missing antibody titers data, calculation of responder status, and average peak will follow the rules described in Table 2-2.

Table 2-2 Calculation of summary parameters for immunogenicity

| | | | | <b>5</b> . | • |
|---|---|---|---|---|---|
| Week<br>9 | Week<br>13 | Week<br>15 | Week 26 | Responder status | Average<br>peak |
| X9 | X13 | X15 | X26 | If (X9 > 16 or X13>16) and | Mean(X9,X15) |
| | | | | (X15 > 26.8 or X26>26.8) then SR else NR | |
| X9 | X13 | X15 | | If (X9 > 16 or X13>16) and (X15 > 26.8) then SR else NR | Mean(X9,X15) |
| X9 | X13 | • | X26 | If (X9 > 16 or X13>16) and (X26>26.8) then SR else NR | X9 |
| X9 | | X15 | X26 | If (X9 > 16) and (X15 > 26.8 or X26>26.8) then SR else NR | Mean(X9,X15) |
| - | X13 | X15 | X26 | If (X13>16) and (X15 > 26.8 or X13>26.8) then SR else NR | X15 |
| X9 | • | X15 | • | If (X9 > 16) and (X15 > 26.8) then SR else NR | Mean(X9,X15) |
| - | X13 | X15 | • | If (X13>16) and (X15 > 26.8) then SR else NR | X15 |
| X9 | • | | X26 | If (X9 > 16) and (X26>26.8) then SR else NR | X9 |
| | X13 | | X26 | If (X13>16) and (X26>26.8) then SR else NR | |
| X9 | | | | | X9 |
| | | X15 | | | X15 |
| | X13 | | | | |
| | | | X26 | | |

In all other situations, the above summary parameters will be set to missing.

#### **Tables**

- Summarize the SR/NR using the classification rules in protocol for completeness.
- Summaries by visit of Aβ specific IgG titers in serum, including mean (with 95% confidence intervals), standard deviation, quartiles, and geometric mean.
- Aβ specific IgG titers in serum summary parameters: Cmax, AUC and, average peak including mean (with 95% confidence intervals), standard deviation, quartiles, and geometric mean (with 95% confidence intervals).
- Correlation between annualized change from baseline in centiloid and AUC will be presented using two types of correlation coefficients (Pearson and Spearman) for CAD106 group overall and by amyloid level (A+/A-). For participants with more than one post-baseline PET scan, the later one will be used for correlation calculation.

The annualized change calculation is the same as described in Amyloid PET section.

The confidence intervals for Cmax and average peak will be computed based on the log transform (assuming normal distribution of the log-transformed values). 95% CI will be calculated based on log-transformation and back transformation will yield a confidence interval


on the original scale. For titer concentration data the arithmetic mean and 95% confidence

interval will be computed using raw data (no log-transformation will be performed).

#### **Figures**

- Individual profile plot for serum A-beta IgG antibody titers over time.
- Mean and 95% confidence intervals of Aβ specific IgG titers in serum at each visit for all CAD106.
- Correlation between annualized change from baseline in centiloid and AUC will be presented using scatter plot by amyloid level (A+/A-). Regression lines will be added for two groups: all CAD106 and CAD A+.

#### 2.7.3 Handling of missing values/censoring/discontinuations

Due to the early termination of the trial, analyses of secondary and other efficacy variables will in general be based on observed cases only, i.e. there will be no imputation of missing data. Exception applies to missing data in RBANS Index scores, i.e., missing values for RBANS Index scores may be imputed using the imputation rule defined in Appendix 5.1.3.3.1.

In case of missing antibody titers data, calculation of responder status, average peak, and Cmax will follow the rules described in Table 2-2. Imputation rule for AUC is described in Section 2.7.2.

#### 2.8 Safety analyses

Reporting of safety data will be based on the SAF. Safety assessments will include adverse events, serious adverse events, deaths, laboratory data (hematology, blood chemistry, urinalysis), vital signs, ECG, safety MRI, physical and neurological examination, prospective suicidality assessment, T-cell lymphocyte response and eDiary.

Summary statistics for categorical data will typically include frequencies and percentages.

For safety parameters, the summaries will be based on worst available observation in an analysis window. The analysis window and definition of worst value is present in Appendix 5.7.

#### 2.8.1 Adverse events (AEs)

Treatment-emergent AEs (TEAEs) are events that either started after the first dose of study drug or events present prior to the start of study drug but increased in severity since the first dose. Adverse events reported within 180 days from study drug discontinuation date (i.e., last injection date) will be considered as TEAE. AEs reported more than 180 days after study drug discontinuation will not be considered treatment emergent (non-TEAE).

TEAEs and non-TEAEs will be summarized separately on the SAF.

#### **Tables**

TEAEs, SAEs, deaths and non-TEAEs will be summarized as follows

- TEAEs regardless of relationship to study drug by SOC, PT and maximum severity
- non-TEAEs regardless of relationship to study drug by SOC, and PT

- TEAEs causing study drug discontinuation by SOC, PT and maximum severity
- TEAEs related to study drug by SOC, PT and maximum severity
- TE-SAEs regardless of relationship to study drug by SOC and PT and maximum severity
- TEAEs regardless of relationship study drug, starting within 7 days after an injection by preferred term and treatment

Note: For missing information on AE relationship to study drug, the most conservative approach will be considered: If information on relationship of the AE to study drug is missing, the AE will be considered as related to study drug for reporting TEAEs. Participants with Unknown or Missing AE severity are included in Mild/Moderate Severity category.

The above summaries are generally without exposure adjustment, except from TEAEs by SOC and PT: this summary will be presented with exposure adjustment. The exposure-adjusted incidence rate of adverse events is defined as the number of participants with the adverse event divided by total participant years at risk in the treatment group. The time at risk for each participant will differ for each adverse event. For participants with events, only the time until the first event contributes to the total participant years at risk. For participants who do not experience the event, the time at risk will be calculated using the duration of exposure as defined in Section 2.4.1. The exposure-adjusted incident rate will be summarized per 100 participant years. For participants with multiple occurrences of the same event, the event will be counted only once per participant.

Adverse events will be reported according to the latest MedDRA dictionary version available at the time of database lock.

If a participant reported more than one adverse event within the same PT, the adverse event with the greatest severity will be counted. If a participant reported more than one adverse event within the same primary SOC, the participant will be counted only once with the greatest severity at the SOC level, wherever applicable. Sorting order for the AE summaries will be as follows:

- For summaries by SOC, SOC will be presented in alphabetical order.
- For summaries by SOC and PT, SOC will presented in alphabetical order; PT will be sorted within system organ class in alphabetical order.

#### Listings

All AEs will be listed ordered by country/center/participant and event date. Adverse events of special interest / grouping of AEs

An adverse event of special interest (AESI) is a set of adverse events that are of scientific and medical concern specific to a compound. These groupings are defined using MedDRA terms, SMQs (standardized MedDRA queries), HLGTs (high level group terms), HLT (high level terms) and PTs (preferred terms).

Customized SMQs (Novartis MedDRA queries, NMQ) may also be used. An NMQ is a customized group of search terms which defines a medical concept for which there is no official SMQ available or the available SMQ does not completely fit the need. It may include a combination of single terms and/or an existing SMQ, narrow or broad.
AESIs as specified in the CAD106-specific Development Safety Profiling Plan (DSPP) are grouped in the corresponding Case Retrieval Sheet (eCRS) and analyzed as a specific group along with other risk search terms.

The search criteria for each of the risks and events will be based on MedDRA and will be comprised by the eCRS. The most recent eCRS at the time of database lock will be used to determine the MedDRA search criteria for identification of the adverse events of special interests.

#### **Tables**

Number and percentages of participants with treatment emergent adverse events of special interest by risk and MedDRA levels will be summarized on SAF.

#### **2.8.2** Deaths

#### **Tables**

Deaths regardless of relationship to study drug by SOC and PT will be summarized on the SAF.

## Listings

Deaths will also be listed separately.

#### 2.8.3 Laboratory data

#### **Tables**

Number and percentages of participants with newly occurring or worsening laboratory abnormalities meeting the clinically notable criteria at any time post-baseline visit will be summarized for all parameters as specified in Appendix 5.6 of this document.

For a participant to meet the criterion of a newly occurring clinically notable value, the participant needs to have a baseline value that is not clinically notable for that parameter. For a participant to meet the criterion of a worsening clinically notable value, the participant needs to have a baseline value that is clinically notable and also have a worse post-baseline value. For participants with missing baseline value, any post-baseline notable value will be considered as newly occurring.

For each participant, all available post-baseline laboratory tests will be used to compare with the notable criteria. If at least one of the results, for a particular parameter, exceeds the criteria, the value will be considered as clinically notable abnormal for that parameter. A participant can be counted in both, low and high categories.

The upper limit of normal (ULN) for each parameter is available in the lab dataset. All available post-baseline laboratory tests will be used to compare with the criteria specified in Appendix 5.6. If at least one of the results, for a particular parameter, exceeds the criteria, the value will be considered as notable abnormal for that parameter. To categorize the abnormality, use the worst case within a lab parameter for a participant if multiple abnormality occurrences exist for the same lab parameter.

The laboratory parameters will be reported in SI units.

The number and percentage of participants with newly occurring or worsening liver enzyme abnormalities meeting the clinically notable criteria at any time post-baseline visit as specified in Appendix 5.3 will be summarized.

## Figures

Box-plots for lab parameters of hematology, biochemistry and urinalysis over time by treatment group will be provided:

### 2.8.4 Other safety data

#### 2.8.4.1 ECG

12-lead ECGs will be performed at screening and throughout the study in supine position. The ECG values will be interpreted and analyzed centrally. The QT intervals will be corrected according to the formula by Fridericia:

Fridericia's formula:  $OTcF = OT/RR^{1/3}$ 

#### **Tables**

The number and percentage of participants with newly occurring or worsening clinically notable ECG abnormalities at any time post-baseline visit will be summarized for all parameters as specified in Appendix 5.6.

#### **Figures**

Box plots over time will be presented by ECG parameter and treatment group.

#### **2.8.4.2** Vital signs

#### **Tables**

The number and percentage of participants with clinically notable vital signs abnormalities will be summarized by visit and by time point as applicable. At each visit, vital signs were collected at three time points: pre-dose, 30 min post dose and 60 min post dose including Body Temperature (C), Sitting Diastolic Blood Pressure (mmHg), Sitting Pulse Rate (BEATS/MIN) and Sitting Systolic Blood Pressure (mmHg). The criteria of clinically notable vital signs are provided in Appendix 5.6.

For body temperature, The eDiary were completed on the day of the injection (in the evening) and then over the following 7 days (in case of persisting reactions, the eDiary should be continued up to 14 days). The 7 days self-measurement eDiary will be summarized by visit.

#### 2.8.4.3 Prospective Suicidality Assessment

The Columbia-Suicide Severity Rating Scale (C-SSRS) is a questionnaire that prospectively assesses Suicidal Ideation and Suicidal Behavior. The electronic version, the eC-SSRS will be administered as described in the visit schedule of the study protocols and may also include unscheduled visits. At the first time of administration of the eC-SSRS, a retrospective

assessment of suicidal behavior and ideation will be collected across lifetime. This data will be used to check inclusion/exclusion criteria. At all other scheduled assessments of suicidal behavior and ideation, any occurrence since the last visit will be collected.

The data will be reported for post-baseline period only. The following three periods have been identified to cover lifetime history, the time between collection of lifetime history and start of study drug intake, and the time on study drug (post-baseline).

#### **Tables**

The number and percentage of participants pertaining to each of the categories of suicidal ideation and behaviors will be presented for all visits after baseline visit (including unscheduled).

The summaries will show numbers and percentages of participants who have an answer "yes" to a suicidal behavior or ideation category at any time for post baseline period.

#### Listings

For participants with any assessment that meets the criteria to trigger the recording of an SAE as specified in the study protocols, a full listing will be presented. The criteria for SAE reporting are as follows:

If, at any time, the score is "Yes" on item 4 or item 5 of the Suicidal Ideation section of the C-SSRS or "Yes". All such cases regardless of whether there was an SAE reported or not will be listed.

## 2.8.4.4 Safety MRI

Safety MRI findings will be summarized overall (at any visit) for ARIA-E, ARIA-H and White matter disease findings.

Worsening of white matter disease is defined on the age-related white matter changes rating Scale (ARWMC) which is rated on a 4 point (0-3) scale per region (bilaterally) on the following 5 different brain regions: Frontal Lobe, Parieto-Occipital, Temporal Lobe, Infratentorial area, Basal ganglia. ARWMC composite score is the sum of individual ARWMC scores from the 5 regions and ranges from 0 to 15. The ARWMC composite score will be used to summarize the white matter disease findings. The definitions of the rating scores is shown in the below <u>Table</u> 2-3.

Table 2-3 The ARWMC Rating Scale for MRI

| Score | Definition |
|---|---|
| White matter lesions | |
| 0 | No lesions (including symmetrical, well-defined caps or bands) |
| 1 | Focal lesions |
| 2 | Beginning confluence of lesions |
| 3 | Diffuse involvement of the entire region, with or without involvement of U fibers |
| Basal ganglia lesions | |
| 0 | No lesions |

| Novartis | For business use only | Page 40 |
|----------------|------------------------|-----------------------|
| SAP Addendum 4 | | CAPI15A2201J Cohort I |
| 1 | 1 focal lesion (≥5 mm) | |
| 2 | >1 focal lesion | |

#### **Tables**

3

#### **Tables**

For ARIA-E, the following parameters will be presented

Confluent lesions

• Participants with any new ARIA-E (mild, moderate and severe) since Baseline,

For ARIA-H, the following parameters will be presented

- Participants with > 4 new microhemorrhages or any new macrohemorrhage ≥ 10 mm in diameter since the Baseline MRI assessment

  OR
- Participants with >10 microhemorrhages (new hemosiderin deposits < 10 mm) Or ≥ 2 macrohemorrhages or ≥ 2 areas of superficial siderosis (large area of hemosiderin deposition ≥ 10 mm)

For white matter disease, the following parameters will be presented

• Participants with a white matter disease score increase since Baseline

#### Listings

Detailed safety MRI listings will be produced for participants with new occurrences or worsening (including Other MRI abnormalities) of identified findings.

#### 2.8.4.5 A-beta - and Q-beta-specific T-cell lymphocyte response

T-cell studies are planned as a part of this study on a subset of at least 50 participants in Cohort I (CAD106 or placebo) at selected sites with personnel trained specifically on the collection process. In the Informed consent at these sites, volume of blood to be collected will be adapted correspondingly.

The objective is the characterization of A $\beta$ - and Q $\beta$ -specific IFN- $\gamma$  responses of T-cell lymphocytes following treatment with CAD106 using living peripheral blood mononuclear cells (PBMCs). The randomization ratio in the CAD106 cohort will be 5:3 (active vs. placebo). Hence, a total sample size of n = 50 will result in about 31 participants on CAD106.

Based on an event rate of 6% for meningoencephalitis as seen with AN-1792, (Orgogozo et al 2003), the probability of observing at least one case of A $\beta$ -specific T-cell activation in 31 patients on active treatment, is 85.3%.

To evaluate T-cell response to A $\beta$ 1-42 peptide, to A $\beta$ 1-6 peptide and to Q $\beta$  protein (positive control), specific Enzyme-Linked ImmunoSpot (ELISPOT) assays will be performed on PBMC samples at a central analytical laboratory specialized in such assays.

A specific T-cell proliferation assay will be performed on PBMC samples taken at Screening. T-cell response data on Gamma interferon (IFN- $\gamma$ ) will be generated for the following test antigens:

- Aβ1-6 peptide,
- Aβ1-42 peptide and
- Qβ peptide pool.

Since  $Q\beta$  is the main component of the virus like particle of CAD106,  $Q\beta$ -specific T-cell priming after dosing with CAD106 is expected (positive control). Antigen-specific T-cell responses will be determined by comparing medium control counts with antigen counts for each patient, at each visit where PBMC samples are taken. Cytokine/antigen samples are repeated three times for each patient and visit, as were the medium control samples. At each visit, the test antigens and the medium control are sampled three times each. The antigen-specific T-cell response will be derived as follows for reliable samples:

- for each patient at each visit, the mean cell count for antigen stimulated wells and the corresponding standard deviation based on the three replicates will be calculated for three types of antigens (Mean(R\_j), SD(R\_j) j=1,2,3).
- for each patient at each visit, the mean cell count for medium control wells and the corresponding standard deviation based on the three replicates will be calculated for the IFN-γ cytokine (Mean(C), SD(C)).
- The antigen-specific T-cell response will then be calculated, for each patient at each visit and for three types of antigens, as Mean(R j) SD(R j) (Mean(C) + SD(C)) for j=1,2,3.

#### **Tables**

For each type of antigen (A $\beta$ 1-6 peptide, A $\beta$ 1-42 peptide, and Q $\beta$  peptide pool) the antigenspecific T-cell response and the change from baseline in T-cell response will be summarized by treatment. The raw T-cell response data and the derived parameters will be listed by patient and visit. No inferential statistical analyses will be performed.





# 2.11 Patient-reported outcomes

The analysis for the patient reported outcome ECog is described within the secondary and other efficacy variables Section 2.7, and eCSSRS is described in the safety analysis Section 2.8.

#### 2.12 Biomarkers

The biomarkers are described in secondary and other efficacy variables <u>Section 2.7</u>.



# 2.14 Interim analysis

IA already occurred:

- DMC activities for safety
- Immunogenicity for CAD106

Due to early termination of the studies, other planned IA for CAD106 will not be performed. All interim analyses are described more specifically in the DMC SAP located in CREDI under /CREDI Projects/C/CNP520A/Administrative files/DMC Documents and Analyses/RAP



# 4 Change to protocol specified analyses

SAF definition (defined in <u>Section 2.2</u>) is different from the protocol defined SAF definition.

The following analysis were defined in the protocol but will not be performed due to early termination of the study:

- Primary analysis for both the primary endpoints
- Sensitivity to the primary analysis
- Supportive analysis to primary endpoints
- MMRM model to key secondary endpoint
- MMRM model to secondary efficacy endpoints

• Antibody titer responder status

The following analysis were not defined in the protocol but will be added:

- All the efficacy analysis will be performed on the SAF.
- Effect size for APCC and RBANS will be calculated and presented graphically.
- Subgroup analysis for Amyloid level will be added to all efficacy (except for TTE) and biomarker endpoints.
- Correlation between centiloid (across all three ligands) and AUC of antibody titer data from "on treatment" visits.
- Correlation between brain volume and amyloid.
- Baseline comparability of specific baseline characteristics.
- The unit of CSF biomarker Abeta 40 was incorrectly specified in DTS as "pg/mL". The correct unit should be "ng/mL". The actual values transferred by were in the correct unit "ng/mL", but were mis-specified in the database as "pg/mL". This has been confirmed by vender ( ). The mistake will be taken care of at programming level for CSR that the unit of CSF Abeta 40 will be summarized and reported using "ng/mL". No transformation of the values is needed.
- In the T-cell data, two participants and the time point 701(baseline) and 702(week 9) has been mixed up (inverted). This issue will be taken care by database unlock in Dec 2020.

# 5 Appendix

## 5.1 Imputation rules

## 5.1.1 Study drug

If study treatment end date is missing, then treatment epoch completion date will be considered the last dose date, the rule will be provided in Programming Dataset Specification (PDS) document in details.

### 5.1.2 AE date imputation

Rules for imputing AE end date or start date will be provided in Programming Dataset Specification (PDS) document in details.

## 5.1.3 Concomitant medication date imputation

Rules for imputing the CM end date or start date will be provided in Programming Dataset Specification (PDS) document in details.

### 5.1.3.1 Prior therapies date imputation

Not Applicable.

## 5.1.3.2 Post therapies date imputation

Rules for imputing the post non-drug therapies end date or start date will be provided in Programming Dataset Specification (PDS) document in details.

#### 5.1.3.3 Other imputations

#### 5.1.3.3.1 Missing values from the same latent variable

For subtests that contribute to the same latent construct variable (Table 5-1), the following rule for missing subtests will be applied: When less than or equal to 50% of the related subtests within a constructed latent variable is missing, these missing subtests will be imputed from the remaining subtests contributing to its latent variable, standardized so that each subtest contributes the same weight to the construct as it would have if measured.

Table 5-1 Latent construct variables and their corresponding subtests

| Latent construct variable | Subtests |
|---|---|
| Immediate Memory Index score | List Learning and Story Memory |
| Visuospatial/Constructional Index Score | Figure Copy and Line Orientation |
| Language Index Score | Semantic Fluency and Picture Naming |
| Attention Index Score | Coding and Digital Span |
| Delayed Memory Index Score | List Recall, Story Recall, Figure Recall and List Recognition |
| Raven's matrices contributing to APCC | A2, A4, A8, B1-B6 |

This is done by calculating the total subscale-weight adjusted observed subtests (i), divided by the maximum weight-adjusted values possible for the observed subtests (i). This will provide the proportion to apply to the missing subtest (j) maximum possible value in order to obtain its imputed value as follows:

 $missing \ subtest_{j} \\ = \frac{\sum_{i=1}^{n} (weight_{i} \times observed \ subtest_{i})}{\sum_{i=1}^{n} (weight_{i} \times observed \ subtest \ max_{i})} \times \ missing \ subtest_{j} \ max.$ 

Missing subtests that could not borrow information from observed related subtests and construct variable values which could not be calculated from their underlying observed/imputed values will be regarded as MAR and will not be imputed.

# 5.2 AEs coding/grading

The MedDRA version which will be available at the time of database lock, will be used for the coding purpose of the adverse events.

# 5.3 Laboratory parameters derivations

Table 5-2 Liver Event and Laboratory Trigger Definitions

| | , 55 |
|---|---|
| | Definition/ threshold |
| LIVER LABORATORY | 3×ULN < ALT / AST ≤ 5×ULN |
| TRIGGERS | 1.5×ULN < TBL ≤ 2×ULN |
| LIVER EVENTS | ALT or AST > 5 × ULN |
| | ALP > 2×ULN (in the absence of known bone pathology) |
| | TBL > 2×ULN (in the absence of known Gilbert syndrome) |
| | ALT or AST > 3×ULN and INR > 1.5 |
| | Potential Hy's Law cases (defined as ALT or AST > 3×ULN and TBL > 2×ULN [mainly conjugated fraction] without notable increase in ALP to > 2×ULN) |
| | Any clinical event of jaundice (or equivalent term) |
| | ALT or AST > 3×ULN accompanied# by (general) malaise, fatigue, abdominal pain, nausea, or vomiting, or rash with eosinophilia |
| | Any adverse event potentially indicative of a liver toxicity * |

<sup>\*</sup>These events cover the following: hepatic failure, fibrosis and cirrhosis, and other liver damage related conditions; the non-infectious hepatitis; the benign, malignant and unspecified liver neoplasms.

ALP = alkaline phosphatase; ALT = Alanine aminotransferase; AST = Aspartate aminotransferase TBL: total bilirubin; ULN: upper limit of normal.

<sup>\*</sup>Consider these adverse events in a window from 30 days before the liver event criteria (ALT or AST >  $3 \times ULN$ ) to 30 days after the liver event criteria (ALT or AST >  $3 \times ULN$ ).

| Table 5-3 | Specific r | renal alert | criteria a | and actions |
|-----------|------------|-------------|------------|-------------|
|-----------|------------|-------------|------------|-------------|

| | Definition/ threshold |
|---|---|
| Serum event | Serum creatinine increase 25 – 49% compared to baseline |
| | Acute Kidney Injury: Serum creatinine increase $\geq 50\%$ compared to baseline |
| Urine event | New dipstick proteinuria ≥ 1+ |
| | Albumin- or Protein-creatinine ratio increase ≥ 2-fold |
| | $ACR \ge 30 \text{ mg/g or} \ge 3 \text{ mg/mmol};$ |
| | PCR ≥ 150 mg/g or > 15 mg/mmol |
| | New dipstick glycosuria ≥ 1+ not due to diabetes |
| | New dipstick hematuria ≥ 1+ not due to trauma* |

ACR = Albumin-creatinine ratio; PCR = Protein-creatinine ratio.

#### 5.4 Statistical models

SAS codes for all statistical methodology described in this section will be included as programming note in TFL Shells.

#### 5.4.1 Primary analysis

### Kaplan Meier approach for TTE

The Kaplan-Meier estimates of the survival functions for each treatment will be plotted. The plot will include the number of participants at risk for each treatment group at pre-specified time points. Median time to event and quartiles including 95% confidence intervals, if estimable, will be provided for each treatment group using the SAS procedure LIFETEST. The confidence intervals will be based on log-log transformation. For each treatment group and time interval: participants at risk, participants with event, participants with event divided by participants at risk, cumulative participants with event and cumulative event probability including 95% confidence interval will be provided.

#### 5.5 Rule of exclusion criteria of analysis sets

The important protocol deviations are defined in below Table 5-4 with deviation ID, deviation code and it's corresponding text description.

Rule of exclusion criteria from analysis sets due to important protocol deviations (if any) will be included prior to database lock in a separate document in CREDI.

The Non-PD criteria for exclusion from analysis sets is explained in below Table 5-5.

<sup>\*</sup>Consider adverse event (injury) in a window from 30 days before the hematuria criteria.

# Table 5-4 Deviation codes description

| Deviation code | Text description | Deviation ID |
|----------------|-------------------------------------------|--------------|
| 1 | SELECTION CRITERIA NOT MET | INCLXX |
| ı | SELECTION CRITERIA NOT WET | EXCLXX |
| 2 | PARTICIPANT NOT WITHDRAWN AS PER PROTOCOL | WITHXX |
| 4 | TREATMENT DEVIATION | TRTXX |
| 5 | PROHIBITED CONCOMITANT MEDICATION | COMDXX |
| 998 | OTHER | OTHXX |

## Table 5-5 Participant Classification

| Analysis Set | PD ID that | Non-PD criteria that cause |
|---|---|---|
| | cause patients to be excluded | patients to be excluded |
| Screened Set | NA | Not having informed consent; |
| | | Not having screening epoch disposition page |
| RAS | NA | Not randomized |
| SAF | NA | No double-blind study drug taken |

# 5.6 Notable and abnormality criteria

# Table 5-6 Clinically notable criteria for vital signs

| Vital Sign Variable | Notable Criteria |
|-----------------------|----------------------------------------------------|
| Pulse (beats/min) | > 120bpm or Increase of ≥15 bpm from baseline |
| | or |
| | < 50bpm or Decrease of ≥15 bpm from baseline |
| Systolic BP (mmHg) | >180 mm Hg or Increase of ≥20 mm Hg from baseline |
| | Or |
| | < 90 mm Hg or Decrease of ≥ 20 mm Hg from baseline |
| Diastolic BP (mmHg) | > 105 mmHg or Increase of ≥ 15 mm Hg from baseline |
| | Or |
| | < 50 mmHg or Decrease of ≥ 15 mm Hg from baseline |
| Body weight (kg) | Decrease ≥ 7% from baseline weight |
| | Increase ≥ 7% from baseline weight |
| Body Temperature (°C) | High: >=38 °C |

## Table 5-7 Clinically notable criteria for selected hematology tests

| | SI units | | US or other units | |
|---|---|---|---|---|
| Laboratory parameter | Lower bound | Upper bound | Lower bound | Upper bound |
| Hemoglobin | 70 (g/L) | 200 (g/L) | 7 (g/dL) | 20 (g/dL) |
| White Cell count | 2 (x10 <sup>9</sup> /L) | 30 (x10 <sup>9</sup> /L) | 2 (x10 <sup>3</sup> /uL) | 30 (x10 <sup>3</sup> /uL) |

| | SI units | | US or other units | |
|---|---|---|---|---|
| Laboratory parameter | Lower bound | Upper bound | Lower bound | Upper bound |
| Platelets | 50 (x10 <sup>9</sup> /L) | 1000<br>(x10 <sup>9</sup> /L) | 50 (x10 <sup>3</sup> /uL) | 1000 x10 <sup>3</sup> /uL) |

# Table 5-8 Clinically notable criteria for selected blood chemistry tests

| Table 5-6 | Cillically Hotab | ie Criteria ioi Seie | cted blood chen | ilistry tests |
|---|---|---|---|---|
| | SI units | | US or other units | 3 |
| Laboratory parameter | Lower bound | Upper bound | Lower bound | Upper bound |
| Sodium | 125 (mmol/L) | 155 (mmol/L) | 125 (mmol/L) | 155 (mmol/L) |
| Potassium | 3 (mmol/L) | 6 (mmol/L) | 3 (mmol/L) | 6 (mmol/L) |
| Calcium | 1.5 (mmol/L) | 3 (mmol/L) | 6 (mg/dL) | 12 (mg/dL) |
| Magnesium | 0.4 (mmol/L) | 1.2 (mmol/L) | 1 (mg/dL) | 3 (mg/dL) |
| Bilirubin (Total) | - | 41 (umol/L) | - | 2.4 (mg/dL) |
| AST | - | > 3×ULN | - | > 3×ULN |
| ALT | - | > 3×ULN | - | > 3×ULN |
| Alkaline<br>Phosphatase<br>(Male) | - | > 2×ULN | - | > 2×ULN |
| Alkaline<br>Phosphatase<br>(Female) | - | > 2×ULN | - | > 2×ULN |
| Creatinine | - | increase 25 –<br>49% compared<br>to baseline | - | increase 25 – 49% compared to baseline |
| | | increase ≥ 50% compared to baseline | | increase ≥ 50% compared to baseline |

# Table 5-9 ECG Abnormality Ranges

| | Abnormality Flags |
|-----------------------------------------|----------------------|
| ECG Parameter | Absolute |
| PR interval | > 250 msec |
| QRS Interval | > 140 msec |
| OT-F lest-mark | >= 500 msec (All) |
| QTcF Interval (Fridericia's correction) | >= 450 msec (Male) |
| (Trideficial & Correction) | >= 470 msec (Female) |

| | Abnormality Flags |
|-------------------------|-------------------|
| ECG Parameter | Absolute |
| QT change from baseline | >60 msec |

# 5.7 Analysis windows rules

Table 5-10 Raven's, MMSE and CDR, ECog

| | | Analysis | window* | |
|---|---|---|---|---|
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 301 | Baseline (Day 1) | -1 | 1 | Baseline |
| 302 | | | | |
| 303 | | | | |
| 304 | | | | |
| 305 | | | | |
| 306 | Week 26 (Day 182) | 2 | 272 | Week 26 |
| 307 | | | | |
| 308 | Week 52 (Day 364) | 273 | 454 | Week 52 |
| 309 | | | | |
| 310 | Week 78 (Day 546) | 455 | 636 | Week 78 |
| 311 | | | | |
| 312 | Week 104 (Day 728) | 637 | 818 | Week 104 |
| 313 | | | | |
| 314 | Week 130 (Day 910) | 819 | 1000 | Week 130 |
| 315 | | | | |
| 316 | Week 156 (Day 1092) | 1001 | 1182 | Week 156 |
| 317 | | | | |
| 318 | Week 182 (Day 1274) | 1183 | 1364 | Week 182 |
| 319 | | | | |
| 320 | Week 208 (Day 1456) | 1365 | 1546 | Week 208 |
| 321 | | | | |
| 322 | Week 234 (Day 1638) | 1547 | 1728 | Week 234 |
| 323 | | | | |
| 324 | Week 260 (Day 1820) | 1729 | 1910 | Week 260 |
| 325 | | | | |
| 326 | Week 286 (Day 2002) | 1911 | 2092 | Week 286 |
| 327 | | | | |
| 328 | Week 312 (Day 2184) | 2093 | 2274 | Week 312 |
| 329 | | | | |

| | | Analysis | window* | |
|---|---|---|---|---|
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 330 | Week 338 (Day 2366) | 2275 | 2456 | Week 338 |
| 331 | | | | |
| 332 | Week 364 (Day 2548) | 2457 | 2638 | Week 364 |
| 333 | | | | |
| 334 | Week 390 (Day 2730) | 2639 | 2820 | Week 390 |
| 335 | | | | |
| 336 | Week 416 (Day 2912) | 2821 | Until EOS | Week 416 |

# Table 5-11 RBANS,

| | | Analysis | window* | |
|---|---|---|---|---|
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 301 | Baseline (Day 1) | -1 | 1 | Baseline |
| 302 | | | | |
| 303 | | | | |
| 304 | Week 13 (Day 91) | 2 | 136 | Week 13 |
| 305 | | | | |
| 306 | Week 26 (Day 182) | 137 | 272 | Week 26 |
| 307 | | | | |
| 308 | Week 52 (Day 364) | 273 | 454 | Week 52 |
| 309 | | | | |
| 310 | Week 78 (Day 546) | 455 | 636 | Week 78 |
| 311 | | | | |
| 312 | Week 104 (Day 728) | 637 | 818 | Week 104 |
| 313 | | | | |
| 314 | Week 130 (Day 910) | 819 | 1000 | Week 130 |
| 315 | | | | |
| 316 | Week 156 (Day 1092) | 1001 | 1182 | Week 156 |
| 317 | | | | |
| 318 | Week 182 (Day 1274) | 1183 | 1364 | Week 182 |
| 319 | | | | |
| 320 | Week 208 (Day 1456) | 1365 | 1546 | Week 208 |
| 321 | | | | |
| 322 | Week 234 (Day 1638) | 1547 | 1728 | Week 234 |
| 323 | | | | |
| 324 | Week 260 (Day 1820) | 1729 | 1910 | Week 260 |
| 325 | | | | |
| 326 | Week 286 (Day 2002) | 1911 | 2092 | Week 286 |
| 327 | | | | |
| 328 | Week 312 (Day 2184) | 2093 | 2274 | Week 312 |

| | | Analysis | window* | |
|---|---|---|---|---|
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 329 | | | | |
| 330 | Week 338 (Day 2366) | 2275 | 2456 | Week 338 |
| 331 | | | | |
| 332 | Week 364 (Day 2548) | 2457 | 2638 | Week 364 |
| 333 | | | | |
| 334 | Week 390 (Day 2730) | 2639 | 2820 | Week 390 |
| 335 | | | | |
| 336 | Week 416 (Day 2912) | 2821 | Until EOS | Week 416 |

 Table 5-12
 Physical / Neurological exams, ECG, laboratory tests

| | | Analysis | window* | |
|---|---|---|---|---|
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 301 | Baseline (Day 1) | -1 | 1 | Baseline |
| 302 | | | | |
| 303 | | | | |
| 304 | Week 13 (Day 91) | 2 | 136 | Week 13 |
| 305 | | | | |
| 306 | Week 26 (Day 182) | 137 | 272 | Week 26 |
| 307 | | | | |
| 308 | Week 52 (Day 364) | 273 | 454 | Week 52 |
| 309 | | | | |
| 310 | Week 78 (Day 546) | 455 | 636 | Week 78 |
| 311 | | | | |
| 312 | Week 104 (Day 728) | 637 | 818 | Week 104 |
| 313 | | | | |
| 314 | Week 130 (Day 910) | 819 | 1000 | Week 130 |
| 315 | | | | |
| 316 | Week 156 (Day 1092) | 1001 | 1182 | Week 156 |
| 317 | | | | |
| 318 | Week 182 (Day 1274) | 1183 | 1364 | Week 182 |
| 319 | | | | |
| 320 | Week 208 (Day 1456) | 1365 | 1546 | Week 208 |
| 321 | | | | |
| 322 | Week 234 (Day 1638) | 1547 | 1728 | Week 234 |
| 323 | | | | |
| 324 | Week 260 (Day 1820) | 1729 | 1910 | Week 260 |
| 325 | | | | |
| 326 | Week 286 (Day 2002) | 1911 | 2092 | Week 286 |
| 327 | | | | |
| 328 | Week 312 (Day 2184) | 2093 | 2274 | Week 312 |
| 329 | | | | |
| 330 | Week 338 (Day 2366) | 2275 | 2456 | Week 338 |
| 331 | | | | |
| 332 | Week 364 (Day 2548) | 2457 | 2638 | Week 364 |
| 333 | | | | |
| 334 | Week 390 (Day 2730) | 2639 | 2820 | Week 390 |
| 335 | | | | |
| 336 | Week 416 (Day 2912) | 2821 | Until EOS | Week 416 |

| | | Analysis | window* | |
|---|---|---|---|---|
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 004 | D 11 (D 4) | | 4 | B " |
| 301 | Baseline (Day 1) | -1 | 1 | Baseline |
| 302 | | | | |
| 303 | | | | |
| 304 | | | | |
| 305 | | | | |
| 306 | Week 26 (Day 182) | 2 | 272 | Week 26 |
| 307 | | | | |
| 308 | Week 52 (Day 364) | 273 | 545 | Week 52 |
| 309 | | | | |
| 310 | | | | |
| 311 | | | | |
| 312 | Week 104 (Day 728) | 546 | 909 | Week 104 |
| 313 | | | | |
| 314 | | | | |
| 315 | | | | |
| 316 | Week 156 (Day 1092) | 910 | 1273 | Week 156 |
| 317 | | | | |
| 318 | | | | |
| 319 | | | | |
| 320 | Week 208 (Day 1456) | 1274 | 1637 | Week 208 |
| 321 | | | | |
| 322 | | | | |
| 323 | | | | |
| 324 | Week 260 (Day 1820) | 1638 | 2001 | Week 260 |
| 325 | , | | | |
| 326 | | | | |
| 327 | | | | |
| 328 | Week 312 (Day 2184) | 2002 | 2365 | Week 312 |
| 329 | ( - , , | - | | |
| 330 | | | | |
| 331 | | | | |
| 332 | Week 364 (Day 2548) | 2366 | 2729 | Week 364 |
| 333 | (Buj 2010) | | | 1700.00 |
| 334 | | | | |
| 335 | | | | |
| 336 | Week 416 (Day 2912) | 2730 | Until EOS | Week 416 |
| 000 | **CCN +10 (Day 2312) | 2100 | Jilli LOO | **CCN T10 |

Table 5-14 Vital signs

| Table 5-14 | vitai sigiis | | | |
|---|---|---|---|---|
| | | Analysis | window* | |
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 301 | Baseline (Day 1) | -1 | 1 | Baseline |
| 302 | Week 7 (Day 49) | 2 | 69 | Week 7 |
| 303 | | | | |
| 304 | Week 13 (Day 91) | 70 | 136 | Week 13 |
| 305 | | | | |
| 306 | Week 26 (Day 182) | 137 | 272 | Week 26 |
| 307 | | | | |
| 308 | Week 52 (Day 364) | 273 | 454 | Week 52 |
| 309 | | | | |
| 310 | Week 78 (Day 546) | 455 | 636 | Week 78 |
| 311 | | | | |
| 312 | Week 104 (Day 728) | 637 | 818 | Week 104 |
| 313 | | | | |
| 314 | Week 130 (Day 910) | 819 | 1000 | Week 130 |
| 315 | | | | |
| 316 | Week 156 (Day 1092) | 1001 | 1182 | Week 156 |
| 317 | | | | |
| 318 | Week 182 (Day 1274) | 1183 | 1364 | Week 182 |
| 319 | | | | |
| 320 | Week 208 (Day 1456) | 1365 | 1546 | Week 208 |
| 321 | | | | |
| 322 | Week 234 (Day 1638) | 1547 | 1728 | Week 234 |
| 323 | | | | |
| 324 | Week 260 (Day 1820) | 1729 | 1910 | Week 260 |
| 325 | | | | |
| 326 | Week 286 (Day 2002) | 1911 | 2092 | Week 286 |
| 327 | | | | |
| 328 | Week 312 (Day 2184) | 2093 | 2274 | Week 312 |
| 329 | | | | |
| 330 | Week 338 (Day 2366) | 2275 | 2456 | Week 338 |
| 331 | | | | |
| 332 | Week 364 (Day 2548) | 2457 | 2638 | Week 364 |
| 333 | | | | |
| 334 | Week 390 (Day 2730) | 2639 | 2820 | Week 390 |
| 335 | | | | |
| 336 | Week 416 (Day 2912) | 2821 | Until EOS | Week 416 |

# Table 5-15 Injections of CAD106

| | | Analysis | window* | |
|---|---|---|---|---|
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 301 | Baseline (Day 1) | -1 | 1 | Baseline |
| 302 | Week 7 (Day 49) | 2 | 90 | Week 7 |
| 303 | | | | |
| 304 | Week 13 (Day 91) | 91 | 181 | Week 13 |
| 305 | | | | |
| 306 | Week 26 (Day 182) | 182 | 272 | Week 26 |
| 307 | Week 39 (Day 273) | 273 | 363 | Week 39 |
| 308 | Week 52 (Day 364) | 364 | 727 | Week 52 |
| 309 | | | | |
| 310 | | | | |
| 311 | | | | |
| 312 | Week 104 (Day 728) | 728 | 1091 | Week 104 |
| 313 | | | | |
| 314 | | | | |
| 315 | | | | |
| 316 | Week 156 (Day 1092) | 1092 | 1455 | Week 156 |
| 317 | | | | |
| 318 | | | | |
| 319 | | | | |
| 320 | Week 208 (Day 1456) | 1456 | Until EOS | Week 208 |

| Table 5-16 | Antibody response | | | |
|---|---|---|---|---|
| | | Analysis | window* | |
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 301 | Baseline (Day 1) | -1 | 1 | Baseline |
| 302 | | | | |
| 303 | Week 9 (Day 63) | 2 | 63 | Week 9 |
| 304 | Week 13 (Day 91) | 64 | 91 | Week 13 |
| 305 | Week 15 (Day 105) | 92 | 105 | Week 15 |
| 306 | Week 26 (Day 182) | 106 | 182 | Week 26 |
| 307 | Week 39 (Day 273) | 183 | 273 | Week 39 |
| 308 | Week 52 (Day 364) | 274 | 364 | Week 52 |
| 309 | Week 65 (Day 455) | 365 | 455 | Week 65 |
| 310 | Week 78 (Day 546) | 456 | 546 | Week 78 |
| 311 | Week 91 (Day 637) | 547 | 637 | Week 91 |
| 312 | Week 104 (Day 728) | 638 | 728 | Week 104 |
| 313 | | | | |
| 314 | Week 130 (Day 910) | 729 | 910 | Week 130 |
| 315 | | | | |
| 316 | Week 156 (Day 1092) | 911 | 1092 | Week 156 |
| 317 | | | | |
| 318 | Week 182 (Day 1274) | 1093 | 1274 | Week 182 |
| 319 | | | | |
| 320 | Week 208 (Day 1456) | 1275 | 1456 | Week 208 |
| 321 | | | | |
| 322 | Week 234 (Day 1638) | 1457 | 1638 | Week 234 |
| 323 | | | | |
| 324 | Week 260 (Day 1820) | 1639 | 1820 | Week 260 |
| 325 | | | | |
| 326 | Week 286 (Day 2002) | 1821 | 2002 | Week 286 |
| 327 | | | | |
| 328 | Week 312 (Day 2184) | 2003 | 2184 | Week 312 |
| 329 | | | | |
| 330 | Week 338 (Day 2366) | 2185 | 2366 | Week 338 |
| 331 | | | | |
| 332 | Week 364 (Day 2548) | 2367 | 2548 | Week 364 |
| 333 | | | | |
| 334 | Week 390 (Day 2730) | 2549 | 2730 | Week 390 |
| 335 | | | | |
| 336 | Week 416 (Day 2912) | 2731 | 2912 | Week 416 |

# **Analyses not by Analysis windows**

The following domains will not be analyzed by analysis window, but according to the scheduled visit and/or visit day as applicable. Analysis windows will not be provided for these.

- Amyloid PET
- Tau PET
- •
- CSF biomarkers
- Blood biomarkers (Serum/Plasma)
- Drug administration
- C-SSRS
- T-cell responses
- Antibody Titer

## 5.8 RBANS Index tables

The RBANS index scores are obtained from the following five age adjusted tables corresponding to the respective total subtest scores.

Table 5-17 Immediate Memory Index Score Equivalents of Subtest Raw Score

| | | | Story | Story Memory Total Score | | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 |
| | | 0 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 1 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 2 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 3 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 4 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 5 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 6 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 7 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 8 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 9 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 10 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 11 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 12 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| | | 13 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| ؈ | | 14 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| Score | | 15 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| la<br>Se | | 16 | 49 | 49 | 49 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 69 | 76 | 78 | 83 | 83 | 83 | 83 | 83 | 87 | 94 | 100 |
| Total | | 17 | 49 | 49 | 49 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 69 | 76 | 78 | 83 | 83 | 83 | 83 | 83 | 87 | 94 | 100 |
| ing | -59 | 18 | 53 | 53 | 53 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 73 | 78 | 81 | 85 | 85 | 85 | 85 | 85 | 90 | 97 | 103 |
| Learning | 50-59 | 19 | 53 | 53 | 53 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 73 | 78 | 81 | 85 | 85 | 85 | 85 | 85 | 90 | 97 | 103 |
| t Le | Ages | 20 | 53 | 53 | 53 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 73 | 78 | 81 | 85 | 85 | 85 | 85 | 85 | 90 | 97 | 103 |
| List | ¥ | 21 | 57 | 57 | 57 | 57 | 57 | 61 | 61 | 61 | 65 | 65 | 69 | 69 | 73 | 76 | 76 | 81 | 83 | 87 | 87 | 87 | 87 | 87 | 94 | 100 | 106 |

| Novartis | For business use only | Page 59 |
|----------------|-----------------------|------------------------|
| SAP Addendum 4 | | CAPI015A2201J Cohort I |

| | 22 | 61 | 61 | 61 | 61 | 61 | 65 | 65 | 65 | 69 | 69 | 73 | 73 | 76 | 78 | 78 | 83 | 85 | 90 | 90 | 90 | 90 | 90 | 97 | 103 | 109 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 23 | 61 | 61 | 61 | 61 | 61 | 65 | 65 | 65 | 69 | 69 | 73 | 73 | 76 | 78 | 78 | 83 | 85 | 90 | 90 | 90 | 90 | 90 | 97 | 103 | 109 |
| | 24 | 65 | 65 | 65 | 65 | 65 | 69 | 69 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 81 | 85 | 87 | 94 | 94 | 94 | 94 | 94 | 100 | 106 | 112 |
| | 25 | 69 | 69 | 69 | 69 | 69 | 73 | 73 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 83 | 87 | 90 | 97 | 97 | 97 | 97 | 97 | 103 | 109 | 114 |
| | 26 | 73 | 73 | 73 | 73 | 73 | 76 | 76 | 76 | 78 | 78 | 81 | 81 | 83 | 85 | 85 | 90 | 94 | 100 | 100 | 100 | 100 | 100 | 106 | 112 | 117 |
| | 27 | 76 | 76 | 76 | 76 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 87 | 87 | 94 | 97 | 103 | 103 | 103 | 103 | 103 | 109 | 114 | 120 |
| | 28 | 76 | 76 | 76 | 76 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 87 | 87 | 94 | 97 | 103 | 103 | 103 | 103 | 103 | 109 | 114 | 120 |
| | 29 | 78 | 78 | 78 | 78 | 78 | 81 | 81 | 81 | 83 | 83 | 85 | 85 | 87 | 90 | 90 | 97 | 100 | 106 | 106 | 106 | 106 | 106 | 112 | 117 | 123 |
| | 30 | 81 | 81 | 81 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 94 | 100 | 103 | 109 | 109 | 109 | 109 | 109 | 114 | 120 | 126 |
| | 31 | 81 | 81 | 81 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 94 | 100 | 103 | 109 | 109 | 109 | 109 | 109 | 114 | 120 | 126 |
| | 32 | 81 | 81 | 81 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 94 | 100 | 103 | 109 | 109 | 109 | 109 | 109 | 114 | 120 | 126 |
| | 33 | 83 | 83 | 83 | 83 | 83 | 85 | 85 | 85 | 87 | 87 | 90 | 90 | 94 | 97 | 97 | 103 | 106 | 112 | 112 | 112 | 112 | 112 | 117 | 123 | 129 |
| | 34 | 85 | 85 | 85 | 85 | 85 | 87 | 87 | 87 | 90 | 90 | 94 | 94 | 97 | 100 | 100 | 106 | 109 | 114 | 114 | 114 | 114 | 114 | 120 | 126 | 132 |
| | 35 | 87 | 87 | 87 | 87 | 87 | 90 | 90 | 90 | 94 | 94 | 97 | 97 | 100 | 103 | 103 | 109 | 112 | 117 | 117 | 117 | 117 | 117 | 123 | 129 | 136 |
| | 36 | 87 | 87 | 87 | 87 | 87 | 90 | 90 | 90 | 94 | 94 | 97 | 97 | 100 | 103 | 103 | 109 | 112 | 117 | 117 | 117 | 117 | 117 | 123 | 129 | 136 |
| | 37 | 90 | 90 | 90 | 90 | 90 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 103 | 106 | 106 | 112 | 114 | 120 | 120 | 120 | 120 | 120 | 126 | 132 | 140 |
| | 38 | 94 | 94 | 94 | 94 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 109 | 114 | 117 | 123 | 123 | 123 | 123 | 123 | 129 | 136 | 144 |
| | 39 | 97 | 97 | 97 | 97 | 97 | 100 | 100 | 100 | 103 | 103 | 106 | 106 | 109 | 112 | 112 | 117 | 120 | 126 | 126 | 126 | 126 | 126 | 132 | 140 | 148 |
| | 40 | 100 | 100 | 100 | 100 | 100 | 103 | 103 | 103 | 106 | 106 | 109 | 109 | 112 | 114 | 114 | 120 | 123 | 129 | 129 | 129 | 129 | 129 | 136 | 144 | 152 |
| | 0 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | 1 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | 2 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | 3 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | 4 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | 5 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | 6 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| • | 7 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| 69 - | 8 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| 09 9 | 9<br>10 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53<br>53 | 53 | 57<br>57 | 61 | 61 | 69<br>69 | 73 | 78<br>79 | 78<br>79 | 78<br>79 | 78<br>78 | 78<br>78 | 83 | 87 | 94 |
| ges | 11 | 44 | 40 | 40<br>44 | 40 | 40 | 44<br>49 | 44<br>49 | 44<br>49 | 49<br>53 | 49<br>53 | 57 | 53<br>57 | 57<br>61 | 61<br>65 | 61<br>65 | 73 | 73<br>76 | 78<br>81 | 78<br>81 | 78<br>81 | 81 | 81 | 83<br>85 | 90 | 97 |
| ⋖ | | 44 | 44 | 44 | ++ | 44 | 43 | 43 | 45 | 55 | 55 | 51 | 31 | UI | 05 | 05 | 13 | 70 | 01 | 01 | 01 | ΟI | 01 | 00 | 90 | 31 |

| Novartis | For business use only | Page 60 |
|----------------|-----------------------|------------------------|
| SAP Addendum 4 | | CAPI015A2201J Cohort I |

| | 12 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 13 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| | 14 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| | 15 | 49 | 49 | 49 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 69 | 76 | 78 | 83 | 83 | 83 | 83 | 83 | 87 | 94 | 100 |
| | 16 | 49 | 49 | 49 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 69 | 76 | 78 | 83 | 83 | 83 | 83 | 83 | 87 | 94 | 100 |
| | 17 | 49 | 49 | 49 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 69 | 76 | 78 | 83 | 83 | 83 | 83 | 83 | 87 | 94 | 100 |
| | 18 | 53 | 53 | 53 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 73 | 78 | 81 | 85 | 85 | 85 | 85 | 85 | 90 | 97 | 103 |
| | 19 | 53 | 53 | 53 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 73 | 78 | 81 | 85 | 85 | 85 | 85 | 85 | 90 | 97 | 103 |
| | 20 | 53 | 53 | 53 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 73 | 78 | 81 | 85 | 85 | 85 | 85 | 85 | 90 | 97 | 103 |
| | 21 | 57 | 57 | 57 | 57 | 57 | 61 | 61 | 61 | 65 | 65 | 69 | 69 | 73 | 76 | 76 | 81 | 83 | 87 | 87 | 87 | 87 | 87 | 94 | 100 | 106 |
| | 22 | 61 | 61 | 61 | 61 | 61 | 65 | 65 | 65 | 69 | 69 | 73 | 73 | 76 | 78 | 78 | 83 | 85 | 90 | 90 | 90 | 90 | 90 | 97 | 103 | 109 |
| | 23 | 61 | 61 | 61 | 61 | 61 | 65 | 65 | 65 | 69 | 69 | 73 | 73 | 76 | 78 | 78 | 83 | 85 | 90 | 90 | 90 | 90 | 90 | 97 | 103 | 109 |
| | 24 | 65 | 65 | 65 | 65 | 65 | 69 | 69 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 81 | 85 | 87 | 94 | 94 | 94 | 94 | 94 | 100 | 106 | 112 |
| | 25 | 69 | 69 | 69 | 69 | 69 | 73 | 73 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 83 | 87 | 90 | 97 | 97 | 97 | 97 | 97 | 103 | 109 | 114 |
| | 26 | 73 | 73 | 73 | 73 | 73 | 76 | 76 | 76 | 78 | 78 | 81 | 81 | 83 | 85 | 85 | 90 | 94 | 100 | 100 | 100 | 100 | 100 | 106 | 112 | 117 |
| | 27 | 76 | 76 | 76 | 76 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 87 | 87 | 94 | 97 | 103 | 103 | 103 | 103 | 103 | 109 | 114 | 120 |
| | 28 | 78 | 78 | 78 | 78 | 78 | 81 | 81 | 81 | 83 | 83 | 85 | 85 | 87 | 90 | 90 | 97 | 100 | 106 | 106 | 106 | 106 | 106 | 112 | 117 | 123 |
| | 29 | 78 | 78 | 78 | 78 | 78 | 81 | 81 | 81 | 83 | 83 | 85 | 85 | 87 | 90 | 90 | 97 | 100 | 106 | 106 | 106 | 106 | 106 | 112 | 117 | 123 |
| | 30 | 81 | 81 | 81 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 94 | 100 | 103 | 109 | 109 | 109 | 109 | 109 | 114 | 120 | 126 |
| | 31 | 81 | 81 | 81 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 94 | 100 | 103 | 109 | 109 | 109 | 109 | 109 | 114 | 120 | 126 |
| | 32 | 81 | 81 | 81 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 94 | 100 | 103 | 109 | 109 | 109 | 109 | 109 | 114 | 120 | 126 |
| | 33 | 83 | 83 | 83 | 83 | 83 | 85 | 85 | 85 | 87 | 87 | 90 | 90 | 94 | 97 | 97 | 103 | 106 | 112 | 112 | 112 | 112 | 112 | 117 | 123 | 129 |
| | 34 | 85 | 85 | 85 | 85 | 85 | 87 | 87 | 87 | 90 | 90 | 94 | 94 | 97 | 100 | 100 | 106 | 109 | 114 | 114 | 114 | 114 | 114 | 120 | 126 | 132 |
| | 35 | 87 | 87 | 87 | 87 | 87 | 90 | 90 | 90 | 94 | 94 | 97 | 97 | 100 | 103 | 103 | 109 | 112 | 117 | 117 | 117 | 117 | 117 | 123 | 129 | 136 |
| | 36 | 90 | 90 | 90 | 90 | 90 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 103 | 106 | 106 | 112 | 114 | 120 | 120 | 120 | 120 | 120 | 126 | 132 | 140 |
| | 37 | 94 | 94 | 94 | 94 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 109 | 114 | 117 | 123 | 123 | 123 | 123 | 123 | 129 | 136 | 144 |
| | 38 | 94 | 94 | 94 | 94 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 109 | 114 | 117 | 123 | 123 | 123 | 123 | 123 | 129 | 136 | 144 |
| | 39 | 97 | 97 | 97 | 97 | 97 | 100 | 100 | 100 | 103 | 103 | 106 | 106 | 109 | 112 | 112 | 117 | 120 | 126 | 126 | 126 | 126 | 126 | 132 | 140 | 148 |
| | 40 | 100 | 100 | 100 | 100 | 100 | 103 | 103 | 103 | 106 | 106 | 109 | 109 | 112 | 114 | 114 | 120 | 123 | 129 | 129 | 129 | 129 | 129 | 136 | 144 | 152 |
| D 4 | • | 40 | 40 | 40 | 40 | 4.4 | 40 | 40 | 40 | 50 | 50 | | | 04 | 0.5 | 00 | 70 | 70 | 70 | 70 | 70 | 0.4 | 00 | 0.7 | 00 | 0.4 |
| Ages | 0 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |

| <br> | | | | | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 1 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 2 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 3 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 4 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 5 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 6 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 7 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 8 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 9 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 10 | 44 | 44 | 44 | 44 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 73 | 76 | 76 | 81 | 81 | 81 | 83 | 85 | 90 | 94 | 97 |
| | 11 | 44 | 44 | 44 | 44 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 73 | 76 | 76 | 81 | 81 | 81 | 83 | 85 | 90 | 94 | 97 |
| | 12 | 44 | 44 | 44 | 44 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 73 | 76 | 76 | 81 | 81 | 81 | 83 | 85 | 90 | 94 | 97 |
| | 13 | 44 | 44 | 44 | 44 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 73 | 76 | 76 | 81 | 81 | 81 | 83 | 85 | 90 | 94 | 97 |
| | 14 | 49 | 49 | 49 | 49 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 76 | 78 | 78 | 83 | 83 | 83 | 85 | 87 | 94 | 97 | 100 |
| | 15 | 49 | 49 | 49 | 49 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 76 | 78 | 78 | 83 | 83 | 83 | 85 | 87 | 94 | 97 | 100 |
| | 16 | 53 | 53 | 53 | 53 | 57 | 61 | 61 | 61 | 65 | 65 | 69 | 69 | 73 | 76 | 78 | 81 | 81 | 85 | 85 | 85 | 87 | 90 | 97 | 100 | 103 |
| | 17 | 53 | 53 | 53 | 53 | 57 | 61 | 61 | 61 | 65 | 65 | 69 | 69 | 73 | 76 | 78 | 81 | 81 | 85 | 85 | 85 | 87 | 90 | 97 | 100 | 103 |
| | 18 | 57 | 57 | 57 | 57 | 61 | 65 | 65 | 65 | 69 | 69 | 73 | 73 | 76 | 78 | 81 | 83 | 83 | 87 | 87 | 87 | 90 | 94 | 100 | 103 | 106 |
| | 19 | 61 | 61 | 61 | 61 | 65 | 69 | 69 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 85 | 85 | 90 | 90 | 90 | 94 | 97 | 103 | 106 | 109 |
| | 20 | 61 | 61 | 61 | 61 | 65 | 69 | 69 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 85 | 85 | 90 | 90 | 94 | 97 | 100 | 106 | 109 | 112 |
| | 21 | 65 | 65 | 65 | 65 | 69 | 73 | 73 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 85 | 87 | 87 | 94 | 94 | 94 | 97 | 100 | 106 | 109 | 112 |
| | 22 | 65 | 65 | 65 | 65 | 69 | 73 | 73 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 85 | 87 | 87 | 94 | 94 | 94 | 97 | 100 | 106 | 109 | 112 |
| | 23 | 69 | 69 | 69 | 69 | 73 | 76 | 76 | 76 | 78 | 78 | 81 | 81 | 83 | 85 | 87 | 90 | 90 | 97 | 97 | 97 | 100 | 103 | 109 | 112 | 114 |
| | 24 | 73 | 73 | 73 | 73 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 87 | 90 | 94 | 94 | 100 | 100 | 100 | 103 | 106 | 112 | 114 | 117 |
| | 25 | 73 | 73 | 73 | 73 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 87 | 90 | 94 | 94 | 100 | 100 | 100 | 103 | 106 | 112 | 114 | 117 |
| | 26 | 76 | 76 | 76 | 76 | 78 | 81 | 81 | 81 | 83 | 83 | 85 | 85 | 87 | 90 | 94 | 97 | 97 | 103 | 103 | 103 | 106 | 109 | 114 | 117 | 120 |
| | 27 | 78 | 78 | 78 | 78 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 97 | 100 | 100 | 106 | 106 | 106 | 109 | 112 | 117 | 120 | 123 |
| | 28 | 78 | 78 | 78 | 78 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 97 | 100 | 100 | 106 | 106 | 106 | 109 | 112 | 117 | 120 | 123 |
| | 29 | 81 | 81 | 81 | 81 | 83 | 85 | 85 | 85 | 87 | 87 | 90 | 90 | 94 | 97 | 100 | 103 | 103 | 109 | 109 | 109 | 112 | 114 | 120 | 123 | 126 |
| | 30 | 81 | 81 | 81 | 81 | 83 | 85 | 85 | 85 | 87 | 87 | 90 | 90 | 94 | 97 | 100 | 103 | 103 | 109 | 109 | 109 | 112 | 114 | 120 | 123 | 126 |
| | 31 | 83 | 83 | 83 | 83 | 85 | 87 | 87 | 87 | 90 | 90 | 94 | 94 | 97 | 100 | 103 | 106 | 106 | 112 | 112 | 112 | 114 | 117 | 123 | 126 | 129 |
| | 32 | 85 | 85 | 85 | 85 | 87 | 90 | 90 | 90 | 94 | 94 | 97 | 97 | 100 | 103 | 106 | 109 | 109 | 114 | 114 | 114 | 117 | 120 | 126 | 129 | 132 |

| Novartis | For business use only | Page 62 |
|----------------|-----------------------|------------------------|
| SAP Addendum 4 | | CAPI015A2201J Cohort I |

| | | 1 | | 1 | | 1 | 1 | | | 1 | 1 | 1 | 1 | | 1 | | 1 | 1 | | | 1 | 1 | 1 | 1 | 1 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 33 | 87 | 87 | 87 | 87 | 90 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 103 | 106 | 109 | 112 | 112 | 117 | 117 | 117 | 120 | 123 | 129 | 132 | 136 |
| | 34 | 87 | 87 | 87 | 87 | 90 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 103 | 106 | 109 | 112 | 112 | 117 | 117 | 117 | 120 | 123 | 129 | 132 | 136 |
| | 35 | 90 | 90 | 90 | 90 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 112 | 114 | 114 | 120 | 120 | 120 | 123 | 126 | 132 | 136 | 140 |
| | 36 | 90 | 90 | 90 | 90 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 112 | 114 | 114 | 120 | 120 | 120 | 123 | 126 | 132 | 136 | 140 |
| | 37 | 94 | 94 | 94 | 94 | 97 | 100 | 100 | 100 | 103 | 103 | 106 | 106 | 109 | 112 | 114 | 117 | 117 | 123 | 123 | 123 | 126 | 129 | 136 | 140 | 144 |
| | 38 | 97 | 97 | 97 | 97 | 100 | 103 | 103 | 103 | 106 | 106 | 109 | 109 | 112 | 114 | 117 | 120 | 120 | 126 | 126 | 126 | 129 | 132 | 140 | 144 | 148 |
| | 39 | 97 | 97 | 97 | 97 | 100 | 103 | 103 | 103 | 106 | 106 | 109 | 109 | 112 | 114 | 117 | 120 | 120 | 126 | 126 | 126 | 129 | 132 | 140 | 144 | 148 |
| | 40 | 100 | 100 | 100 | 100 | 103 | 106 | 106 | 106 | 109 | 109 | 112 | 112 | 114 | 117 | 120 | 123 | 123 | 129 | 129 | 129 | 132 | 136 | 144 | 148 | 152 |
| | 0 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | 1 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | 2 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | 3 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | 4 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | 5 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | 6 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | 7 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | 8 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | 9 | 44 | 44 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 85 | 85 | 87 | 90 | 94 | 97 |
| | 10 | 44 | 44 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 85 | 85 | 87 | 90 | 94 | 97 |
| | 11 | 44 | 44 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 85 | 85 | 87 | 90 | 94 | 97 |
| | 12 | 44 | 44 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 85 | 85 | 87 | 90 | 94 | 97 |
| | 13 | 49 | 49 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 76 | 78 | 78 | 81 | 81 | 83 | 85 | 87 | 87 | 90 | 94 | 97 | 100 |
| | 14 | 49 | 49 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 76 | 78 | 78 | 81 | 81 | 83 | 85 | 87 | 87 | 90 | 94 | 97 | 100 |
| | 15 | 53 | 53 | 57 | 57 | 61 | 61 | 61 | 65 | 65 | 69 | 69 | 73 | 78 | 81 | 81 | 83 | 83 | 85 | 87 | 90 | 90 | 94 | 97 | 100 | 103 |
| | 16 | 57 | 57 | 61 | 61 | 65 | 65 | 65 | 69 | 69 | 73 | 73 | 76 | 81 | 83 | 83 | 85 | 85 | 87 | 90 | 94 | 94 | 97 | 100 | 103 | 106 |
| | 17 | 61 | 61 | 65 | 65 | 69 | 69 | 69 | 73 | 73 | 76 | 76 | 78 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 97 | 97 | 100 | 103 | 106 | 109 |
| | 18 | 61 | 61 | 65 | 65 | 69 | 69 | 69 | 73 | 73 | 76 | 76 | 78 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 97 | 97 | 100 | 103 | 106 | 109 |
| | 19 | 65 | 65 | 69 | 69 | 73 | 73 | 73 | 76 | 76 | 78 | 78 | 81 | 85 | 87 | 87 | 90 | 90 | 94 | 97 | 100 | 100 | 103 | 106 | 109 | 112 |
| 68 | 20 | 69 | 69 | 73 | 73 | 76 | 76 | 76 | 78 | 78 | 81 | 81 | 83 | 87 | 90 | 90 | 94 | 94 | 97 | 100 | 103 | 103 | 106 | 109 | 112 | 114 |
| 80-89 | 21 | 73 | 73 | 76 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 90 | 94 | 94 | 97 | 97 | 100 | 103 | 106 | 106 | 109 | 112 | 114 | 117 |
| S | 22 | 73 | 73 | 76 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 90 | 94 | 94 | 97 | 97 | 100 | 103 | 106 | 106 | 109 | 112 | 114 | 117 |
| Ag | 23 | 76 | 76 | 78 | 78 | 81 | 81 | 81 | 83 | 83 | 85 | 85 | 87 | 94 | 97 | 97 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 114 | 117 | 120 |

| _ | | | | | | | | | | | | | | | | | | | | | | | 1 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 24 | 78 | 78 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 112 | 112 | 114 | 117 | 120 | 123 |
| | 25 | 78 | 78 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 112 | 112 | 114 | 117 | 120 | 123 |
| | 26 | 81 | 81 | 83 | 83 | 85 | 85 | 85 | 87 | 87 | 90 | 90 | 94 | 100 | 103 | 103 | 106 | 106 | 109 | 112 | 114 | 114 | 117 | 120 | 123 | 126 |
| | 27 | 83 | 83 | 85 | 85 | 87 | 87 | 87 | 90 | 90 | 94 | 94 | 97 | 103 | 106 | 106 | 109 | 109 | 112 | 114 | 117 | 117 | 120 | 123 | 126 | 129 |
| | 28 | 83 | 83 | 85 | 85 | 87 | 87 | 87 | 90 | 90 | 94 | 94 | 97 | 103 | 106 | 106 | 109 | 109 | 112 | 114 | 117 | 117 | 120 | 123 | 126 | 129 |
| | 29 | 85 | 85 | 87 | 87 | 90 | 90 | 90 | 94 | 94 | 97 | 97 | 100 | 106 | 109 | 109 | 112 | 112 | 114 | 117 | 120 | 120 | 123 | 126 | 129 | 132 |
| | 30 | 85 | 85 | 87 | 87 | 90 | 90 | 90 | 94 | 94 | 97 | 97 | 100 | 106 | 109 | 109 | 112 | 112 | 114 | 117 | 120 | 120 | 123 | 126 | 129 | 132 |
| | 31 | 87 | 87 | 90 | 90 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 103 | 109 | 112 | 112 | 114 | 114 | 117 | 120 | 123 | 123 | 126 | 129 | 132 | 136 |
| | 32 | 87 | 87 | 90 | 90 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 103 | 109 | 112 | 112 | 114 | 114 | 117 | 120 | 123 | 123 | 126 | 129 | 132 | 136 |
| | 33 | 90 | 90 | 94 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 112 | 114 | 114 | 117 | 117 | 120 | 123 | 126 | 126 | 129 | 132 | 136 | 140 |
| | 34 | 90 | 90 | 94 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 112 | 114 | 114 | 117 | 117 | 120 | 123 | 126 | 126 | 129 | 132 | 136 | 140 |
| | 35 | 94 | 94 | 97 | 97 | 100 | 100 | 100 | 103 | 103 | 106 | 106 | 109 | 114 | 117 | 117 | 120 | 120 | 123 | 126 | 129 | 129 | 132 | 136 | 140 | 144 |
| | 36 | 94 | 94 | 97 | 97 | 100 | 100 | 100 | 103 | 103 | 106 | 106 | 109 | 114 | 117 | 117 | 120 | 120 | 123 | 126 | 129 | 129 | 132 | 136 | 140 | 144 |
| | 37 | 97 | 97 | 100 | 100 | 103 | 103 | 103 | 106 | 106 | 109 | 109 | 112 | 117 | 120 | 120 | 123 | 123 | 126 | 129 | 132 | 132 | 136 | 140 | 144 | 148 |
| | 38 | 97 | 97 | 100 | 100 | 103 | 103 | 103 | 106 | 106 | 109 | 109 | 112 | 117 | 120 | 120 | 123 | 123 | 126 | 129 | 132 | 132 | 136 | 140 | 144 | 148 |
| | 39 | 100 | 100 | 103 | 103 | 106 | 106 | 106 | 109 | 109 | 112 | 112 | 114 | 120 | 123 | 123 | 126 | 126 | 129 | 132 | 136 | 136 | 140 | 144 | 148 | 152 |
| | 40 | 100 | 100 | 103 | 103 | 106 | 106 | 106 | 109 | 109 | 112 | 112 | 114 | 120 | 123 | 123 | 126 | 126 | 129 | 132 | 136 | 136 | 140 | 144 | 148 | 152 |

Table 5-18 Visuospatial/Constructional Index Score Equivalents of Subtest Raw Scores

| | | | Line ( | Orienta | tion To | tal Sc | ore | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 |
| | | 0 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| <u>=</u> | | 1 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| Total | | 2 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| py l | | 3 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| Cop | | 4 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| ် လ | _ | 5 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| igu | 0-59 | 6 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| 证 | )S S( | 7 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | Age | 8 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |

| | | | Line ( | Orienta | tion To | tal Sc | ore | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 |
| | | 9 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 10 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 11 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 12 | 53 | 53 | 53 | 53 | 53 | 53 | 56 | 56 | 58 | 60 | 62 | 62 | 64 | 66 | 66 | 69 | 72 | 75 | 81 | 84 | 87 |
| | | 13 | 56 | 56 | 56 | 56 | 56 | 56 | 58 | 58 | 60 | 62 | 64 | 64 | 66 | 69 | 69 | 72 | 75 | 78 | 84 | 87 | 89 |
| | | 14 | 58 | 58 | 58 | 58 | 58 | 58 | 60 | 60 | 62 | 64 | 66 | 66 | 69 | 72 | 72 | 75 | 78 | 81 | 87 | 89 | 92 |
| | | 15 | 60 | 60 | 60 | 60 | 60 | 60 | 62 | 62 | 64 | 66 | 69 | 69 | 72 | 75 | 75 | 78 | 81 | 84 | 89 | 92 | 96 |
| | | 16 | 62 | 62 | 62 | 62 | 62 | 62 | 64 | 64 | 66 | 69 | 72 | 72 | 75 | 78 | 78 | 81 | 84 | 87 | 92 | 96 | 100 |
| | | 17 | 66 | 66 | 66 | 66 | 66 | 66 | 69 | 69 | 72 | 75 | 78 | 78 | 81 | 84 | 84 | 87 | 89 | 92 | 100 | 102 | 105 |
| | | 18 | 72 | 72 | 72 | 72 | 72 | 72 | 75 | 75 | 78 | 81 | 84 | 84 | 87 | 89 | 89 | 92 | 96 | 100 | 105 | 109 | 112 |
| | | 19 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 78 | 81 | 84 | 87 | 87 | 89 | 92 | 92 | 96 | 100 | 102 | 109 | 112 | 116 |
| | | 20 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 84 | 87 | 89 | 92 | 92 | 96 | 100 | 100 | 102 | 105 | 109 | 116 | 121 | 126 |
| | | | Line C | Orienta | tion To | tal Sc | ore | | | | | | | | | | | | | | | | |
| | | 1 | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 |
| | | 0 | 50 | <b>1</b> 50 | <b>2</b> 50 | 50 | 50 | 50 | 53 | 56 | 56 | 58 | 60 | <b>11</b> 60 | 62 | 64 | 64 | 66 | 69 | 72 | <b>18</b> 78 | 81 | 84 |
| | | 1 | 50<br>50 | 50<br>50 | 50<br>50 | 50<br>50 | 50<br>50 | 50<br>50 | 53<br>53 | 56<br>56 | 56<br>56 | 58<br>58 | 60<br>60 | 60<br>60 | 62<br>62 | 64<br>64 | 64<br>64 | 66<br>66 | 69<br>69 | 72<br>72 | 78<br>78 | 81<br>81 | 84<br>84 |
| | | 1 2 | 50<br>50<br>50 | 50<br>50<br>50 | 50<br>50<br>50 | 50<br>50<br>50 | 50<br>50<br>50 | 50<br>50<br>50 | 53<br>53<br>53 | 56<br>56<br>56 | 56<br>56<br>56 | 58<br>58<br>58 | 60<br>60<br>60 | 60<br>60<br>60 | 62<br>62<br>62 | 64<br>64<br>64 | 64<br>64<br>64 | 66<br>66<br>66 | 69<br>69<br>69 | 72<br>72<br>72 | 78<br>78<br>78 | 81<br>81<br>81 | 84<br>84<br>84 |
| | | 1 2 3 | 50<br>50<br>50<br>50 | 50<br>50<br>50<br>50 | 50<br>50<br>50<br>50 | 50<br>50<br>50<br>50 | 50<br>50<br>50<br>50 | 50<br>50<br>50<br>50 | 53<br>53<br>53<br>53 | 56<br>56<br>56<br>56 | 56<br>56<br>56<br>56 | 58<br>58<br>58<br>58 | 60<br>60<br>60 | 60<br>60<br>60 | 62<br>62<br>62<br>62 | 64<br>64<br>64<br>64 | 64<br>64<br>64<br>64 | 66<br>66<br>66 | 69<br>69<br>69 | 72<br>72<br>72<br>72 | 78<br>78<br>78<br>78 | 81<br>81<br>81<br>81 | 84<br>84<br>84<br>84 |
| Đ | | 1 2 3 4 | 50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50 | 53<br>53<br>53<br>53<br>53 | 56<br>56<br>56<br>56<br>56 | 56<br>56<br>56<br>56<br>56 | 58<br>58<br>58<br>58<br>58 | 60<br>60<br>60<br>60 | 60<br>60<br>60<br>60 | 62<br>62<br>62<br>62<br>62 | 64<br>64<br>64<br>64 | 64<br>64<br>64<br>64<br>64 | 66<br>66<br>66<br>66 | 69<br>69<br>69<br>69 | 72<br>72<br>72<br>72<br>72<br>72 | 78<br>78<br>78<br>78<br>78 | 81<br>81<br>81<br>81<br>81 | 84<br>84<br>84<br>84<br>84 |
| core | | 1 2 3 | 50<br>50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50 | 53<br>53<br>53<br>53<br>53<br>53 | 56<br>56<br>56<br>56<br>56<br>56 | 56<br>56<br>56<br>56<br>56<br>56 | 58<br>58<br>58<br>58<br>58<br>58 | 60<br>60<br>60 | 60<br>60<br>60 | 62<br>62<br>62<br>62<br>62<br>62 | 64<br>64<br>64<br>64 | 64<br>64<br>64<br>64<br>64<br>64 | 66<br>66<br>66 | 69<br>69<br>69 | 72<br>72<br>72<br>72 | 78<br>78<br>78<br>78 | 81<br>81<br>81<br>81 | 84<br>84<br>84<br>84<br>84<br>84 |
| al Score | | 1<br>2<br>3<br>4<br>5 | 50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50<br>50 | 53<br>53<br>53<br>53<br>53 | 56<br>56<br>56<br>56<br>56 | 56<br>56<br>56<br>56<br>56 | 58<br>58<br>58<br>58<br>58 | 60<br>60<br>60<br>60<br>60 | 60<br>60<br>60<br>60<br>60 | 62<br>62<br>62<br>62<br>62 | 64<br>64<br>64<br>64<br>64 | 64<br>64<br>64<br>64<br>64 | 66<br>66<br>66<br>66<br>66 | 69<br>69<br>69<br>69<br>69 | 72<br>72<br>72<br>72<br>72<br>72<br>72 | 78<br>78<br>78<br>78<br>78<br>78 | 81<br>81<br>81<br>81<br>81 | 84<br>84<br>84<br>84<br>84 |
| Total Score | | 1<br>2<br>3<br>4<br>5<br>6 | 50 | 50<br>50<br>50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50<br>50<br>50 | 50<br>50<br>50<br>50<br>50<br>50<br>50 | 53 | 56<br>56<br>56<br>56<br>56<br>56<br>56 | 56<br>56<br>56<br>56<br>56<br>56<br>56 | 58<br>58<br>58<br>58<br>58<br>58<br>58 | 60<br>60<br>60<br>60<br>60<br>60 | 60<br>60<br>60<br>60<br>60<br>60 | 62 | 64<br>64<br>64<br>64<br>64<br>64<br>64 | 64<br>64<br>64<br>64<br>64<br>64<br>64 | 66<br>66<br>66<br>66<br>66<br>66 | 69<br>69<br>69<br>69<br>69<br>69 | 72 | 78<br>78<br>78<br>78<br>78<br>78<br>78 | 81<br>81<br>81<br>81<br>81<br>81 | 84<br>84<br>84<br>84<br>84<br>84 |
| Total | | 1<br>2<br>3<br>4<br>5<br>6<br>7 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 56 | 58 | 60<br>60<br>60<br>60<br>60<br>60<br>60 | 60<br>60<br>60<br>60<br>60<br>60<br>60 | 62 | 64<br>64<br>64<br>64<br>64<br>64<br>64 | 64 | 66<br>66<br>66<br>66<br>66<br>66<br>66 | 69<br>69<br>69<br>69<br>69<br>69<br>69 | 72 | 78 | 81<br>81<br>81<br>81<br>81<br>81<br>81 | 84<br>84<br>84<br>84<br>84<br>84<br>84 |
| Total | 6 | 1<br>2<br>3<br>4<br>5<br>6<br>7<br>8 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69<br>69<br>69<br>69<br>69<br>69<br>69 | 72 | 78 | 81 | 84 |
| Copy Total | 69-09 | 1<br>2<br>3<br>4<br>5<br>6<br>7<br>8 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| Total | ges 60-69 | 1<br>2<br>3<br>4<br>5<br>6<br>7<br>8<br>9 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |

| | | | Line C | Orienta | tion To | tal Sc | ore | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 |
| | | 14 | 58 | 58 | 58 | 58 | 58 | 58 | 60 | 62 | 62 | 64 | 66 | 66 | 69 | 72 | 72 | 75 | 78 | 81 | 87 | 89 | 92 |
| | | 15 | 60 | 60 | 60 | 60 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 69 | 72 | 75 | 75 | 78 | 81 | 84 | 89 | 92 | 96 |
| | | 16 | 62 | 62 | 62 | 62 | 62 | 62 | 64 | 66 | 66 | 69 | 72 | 72 | 75 | 78 | 78 | 81 | 84 | 87 | 92 | 96 | 100 |
| | | 17 | 66 | 66 | 66 | 66 | 66 | 66 | 69 | 72 | 72 | 75 | 78 | 78 | 81 | 84 | 84 | 87 | 89 | 92 | 100 | 102 | 105 |
| | | 18 | 72 | 72 | 72 | 72 | 72 | 72 | 75 | 78 | 78 | 81 | 84 | 84 | 87 | 89 | 89 | 92 | 96 | 100 | 105 | 109 | 112 |
| | | 19 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 81 | 84 | 87 | 87 | 89 | 92 | 92 | 96 | 100 | 102 | 109 | 112 | 116 |
| | | 20 | 84 | 84 | 84 | 84 | 84 | 84 | 87 | 89 | 89 | 92 | 96 | 96 | 100 | 102 | 102 | 105 | 109 | 112 | 121 | 126 | 131 |
| | | 0 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 1 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 2 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 3 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 4 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 5 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 6 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 7 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 8 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 9 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 10 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | | 11 | 53 | 53 | 53 | 53 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 62 | 64 | 66 | 66 | 69 | 72 | 75 | 81 | 84 | 87 |
| | | 12 | 56 | 56 | 56 | 56 | 56 | 56 | 58 | 60 | 62 | 62 | 64 | 64 | 66 | 69 | 69 | 72 | 75 | 78 | 84 | 87 | 89 |
| | | 13 | 58 | 58 | 58 | 58 | 58 | 58 | 60 | 62 | 64 | 64 | 66 | 66 | 69 | 72 | 72 | 75 | 78 | 81 | 87 | 89 | 92 |
| | | 14 | 58 | 58 | 58 | 58 | 58 | 58 | 60 | 62 | 64 | 64 | 66 | 66 | 69 | 72 | 72 | 75 | 78 | 81 | 87 | 89 | 92 |
| | | 15 | 60 | 60 | 60 | 60 | 60 | 60 | 62 | 64 | 66 | 66 | 69 | 69 | 72 | 75 | 75 | 78 | 81 | 84 | 89 | 92 | 96 |
| | | 16 | 64 | 64 | 64 | 64 | 64 | 64 | 66 | 69 | 72 | 72 | 75 | 75 | 78 | 81 | 81 | 84 | 87 | 89 | 96 | 100 | 102 |
| | 6 | 17 | 69 | 69 | 69 | 69 | 69 | 69 | 72 | 75 | 78 | 78 | 81 | 81 | 84 | 87 | 87 | 89 | 92 | 96 | 102 | 105 | 109 |
| | 70-7 | 18 | 72 | 72 | 72 | 72 | 72 | 72 | 75 | 78 | 81 | 81 | 84 | 84 | 87 | 89 | 89 | 92 | 96 | 100 | 105 | 109 | 112 |
| | ges 7 | 19 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 87 | 87 | 89 | 89 | 92 | 96 | 96 | 100 | 102 | 105 | 112 | 116 | 121 |
| ļ | Ag | 20 | 84 | 84 | 84 | 84 | 84 | 84 | 87 | 89 | 92 | 92 | 96 | 96 | 100 | 102 | 102 | 105 | 109 | 112 | 121 | 126 | 131 |

| | | Line ( | Orienta | tion To | tal Sc | ore | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 |
| | 0 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 1 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 2 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 3 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 4 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 5 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 6 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 7 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 8 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 9 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 10 | 53 | 53 | 53 | 53 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 62 | 64 | 66 | 66 | 72 | 75 | 81 | 84 | 87 | 89 |
| | 11 | 53 | 53 | 53 | 53 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 62 | 64 | 66 | 66 | 72 | 75 | 81 | 84 | 87 | 89 |
| | 12 | 56 | 56 | 56 | 56 | 56 | 58 | 58 | 60 | 62 | 62 | 64 | 64 | 66 | 69 | 69 | 75 | 78 | 84 | 87 | 89 | 92 |
| | 13 | 58 | 58 | 58 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 66 | 69 | 72 | 72 | 78 | 81 | 87 | 89 | 92 | 96 |
| | 14 | 60 | 60 | 60 | 60 | 60 | 62 | 62 | 64 | 66 | 66 | 69 | 69 | 72 | 75 | 75 | 81 | 84 | 89 | 92 | 96 | 100 |
| | 15 | 62 | 62 | 62 | 62 | 62 | 64 | 64 | 66 | 69 | 69 | 72 | 72 | 75 | 78 | 78 | 84 | 87 | 92 | 96 | 100 | 102 |
| 68 | 16 | 66 | 66 | 66 | 66 | 66 | 69 | 69 | 72 | 75 | 75 | 78 | 78 | 81 | 84 | 84 | 89 | 92 | 100 | 102 | 105 | 109 |
| 80-89 | 17 | 72 | 72 | 72 | 72 | 72 | 75 | 75 | 78 | 81 | 81 | 84 | 84 | 87 | 89 | 89 | 96 | 100 | 105 | 109 | 112 | 116 |
| Ages | 18 | 75 | 75 | 75 | 75 | 75 | 78 | 78 | 81 | 84 | 84 | 87 | 87 | 89 | 92 | 92 | 100 | 102 | 109 | 112 | 116 | 121 |
| Αĉ | 19 | 78 | 78 | 78 | 78 | 78 | 81 | 81 | 84 | 87 | 87 | 89 | 89 | 92 | 96 | 96 | 102 | 105 | 112 | 116 | 121 | 126 |
| | 20 | 84 | 84 | 84 | 84 | 84 | 87 | 87 | 89 | 92 | 92 | 96 | 96 | 100 | 102 | 102 | 109 | 112 | 121 | 126 | 131 | 136 |

Table 5-19 Language Index Score Equivalents of Subtest Raw Scores

| Picture Naming Total Score | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9–10 |
| nan<br>c<br>enc<br>otal | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| Sen<br>tit<br>Flue<br>A Ag | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |

| | Picture Namir | Picture Naming Total Score | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9–10 |
| 2 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| 3 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| 4 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| 5 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| 6 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| 7 | 44 | 44 | 44 | 44 | 44 | 47 | 51 | 54 | 60 | 75 |
| 8 | 44 | 44 | 44 | 44 | 44 | 47 | 51 | 54 | 60 | 75 |
| 9 | 47 | 47 | 47 | 47 | 47 | 51 | 54 | 57 | 64 | 79 |
| 10 | 47 | 47 | 47 | 47 | 47 | 51 | 54 | 57 | 64 | 79 |
| 11 | 47 | 47 | 47 | 47 | 47 | 51 | 54 | 57 | 64 | 79 |
| 12 | 51 | 51 | 51 | 51 | 51 | 54 | 57 | 60 | 68 | 82 |
| 13 | 51 | 51 | 51 | 51 | 51 | 54 | 57 | 60 | 68 | 82 |
| 14 | 54 | 54 | 54 | 54 | 54 | 57 | 60 | 64 | 71 | 84 |
| 15 | 57 | 57 | 57 | 57 | 57 | 60 | 64 | 68 | 75 | 87 |
| 16 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 71 | 79 | 90 |
| 17 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 71 | 79 | 90 |
| 18 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 75 | 83 | 94 |
| 19 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 75 | 83 | 94 |
| 20 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 79 | 87 | 97 |
| 21 | 71 | 71 | 71 | 71 | 71 | 75 | 79 | 83 | 90 | 99 |
| 22 | 71 | 71 | 71 | 71 | 71 | 75 | 79 | 83 | 90 | 99 |
| 23 | 75 | 75 | 75 | 75 | 75 | 79 | 83 | 87 | 92 | 102 |
| 24 | 75 | 75 | 75 | 75 | 75 | 79 | 83 | 87 | 92 | 102 |
| 25 | 79 | 79 | 79 | 79 | 79 | 83 | 87 | 90 | 94 | 105 |
| 26 | 83 | 83 | 83 | 83 | 83 | 87 | 90 | 92 | 96 | 109 |
| 27 | 83 | 83 | 83 | 83 | 83 | 87 | 90 | 92 | 96 | 109 |
| 28 | 87 | 87 | 87 | 87 | 87 | 90 | 92 | 94 | 100 | 113 |
| 29 | 87 | 87 | 87 | 87 | 87 | 90 | 92 | 94 | 100 | 113 |

| | | Picture Na | ming Total Scor | e | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9–10 |
| | 30 | 90 | 90 | 90 | 90 | 90 | 92 | 94 | 96 | 102 | 117 |
| | 31 | 92 | 92 | 92 | 92 | 92 | 94 | 96 | 100 | 104 | 120 |
| | 32 | 92 | 92 | 92 | 92 | 92 | 94 | 96 | 100 | 104 | 120 |
| | 33 | 94 | 94 | 94 | 94 | 94 | 96 | 100 | 102 | 108 | 124 |
| | 34 | 96 | 96 | 96 | 96 | 96 | 100 | 102 | 104 | 112 | 127 |
| | 35 | 100 | 100 | 100 | 100 | 100 | 102 | 104 | 108 | 116 | 131 |
| | 36+ | 100 | 100 | 100 | 100 | 100 | 102 | 104 | 108 | 116 | 131 |
| | | | <b>.</b> | • | <u>'</u> | | 1 | | | <b>.</b> | <u>'</u> |
| | 0 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 74 |
| | 1 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 74 |
| | 2 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 74 |
| | 3 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 74 |
| | 4 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 74 |
| | <u>5</u> | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 74 |
| | 6 | 44 | 44 | 44 | 44 | 44 | 47 | 51 | 54 | 60 | 78 |
| | 7 | 44 | 44 | 44 | 44 | 44 | 47 | 51 | 54 | 60 | 78 |
| | 8 | 44 | 44 | 44 | 44 | 44 | 47 | 51 | 54 | 60 | 78 |
| 59-0 | 9 | 47 | 47 | 47 | 47 | 47 | 51 | 54 | 57 | 64 | 82 |
| Ages 60-69 | 10 | 47 | 47 | 47 | 47 | 47 | 51 | 54 | 57 | 64 | 82 |
| Age | 11 | 47 | 47 | 47 | 47 | 47 | 51 | 54 | 57 | 64 | 82 |
| | 12 | 51 | 51 | 51 | 51 | 51 | 54 | 57 | 60 | 68 | 85 |
| | 13 | 51 | 51 | 51 | 51 | 51 | 54 | 57 | 60 | 68 | 85 |
| | 14 | 54 | 54 | 54 | 54 | 54 | 57 | 60 | 64 | 71 | 87 |
| | 15 | 57 | 57 | 57 | 57 | 57 | 60 | 64 | 68 | 75 | 90 |
| | 16 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 71 | 79 | 92 |
| | 17 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 71 | 79 | 92 |
| | 18 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 75 | 83 | 96 |
| | 19 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 75 | 83 | 96 |
| | 20 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 79 | 87 | 98 |

| | | Picture Nam | ning Total Score | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9–10 |
| | 21 | 71 | 71 | 71 | 71 | 71 | 75 | 79 | 83 | 90 | 101 |
| | 22 | 71 | 71 | 71 | 71 | 71 | 75 | 79 | 83 | 90 | 101 |
| | 23 | 75 | 75 | 75 | 75 | 75 | 79 | 83 | 87 | 92 | 104 |
| | 24 | 75 | 75 | 75 | 75 | 75 | 79 | 83 | 87 | 92 | 104 |
| | 25 | 79 | 79 | 79 | 79 | 79 | 83 | 87 | 90 | 94 | 108 |
| | 26 | 83 | 83 | 83 | 83 | 83 | 87 | 90 | 92 | 96 | 111 |
| | 27 | 87 | 87 | 87 | 87 | 87 | 90 | 92 | 94 | 100 | 116 |
| | 28 | 87 | 87 | 87 | 87 | 87 | 90 | 92 | 94 | 100 | 116 |
| | 29 | 90 | 90 | 90 | 90 | 90 | 92 | 94 | 96 | 102 | 120 |
| | 30 | 90 | 90 | 90 | 90 | 90 | 92 | 94 | 96 | 102 | 120 |
| | 31 | 94 | 94 | 94 | 94 | 94 | 96 | 100 | 102 | 108 | 127 |
| | 32 | 94 | 94 | 94 | 94 | 94 | 96 | 100 | 102 | 108 | 127 |
| | 33 | 94 | 94 | 94 | 94 | 94 | 96 | 100 | 102 | 108 | 127 |
| | 34 | 96 | 96 | 96 | 96 | 96 | 100 | 102 | 104 | 112 | 130 |
| | 35 | 100 | 100 | 100 | 100 | 100 | 102 | 104 | 108 | 116 | 134 |
| | 36+ | 100 | 100 | 100 | 100 | 100 | 102 | 104 | 108 | 116 | 134 |
| | 0 | 40 | 40 | 40 | 40 | 40 | 47 | 47 | 51 | 57 | 74 |
| | 1 | 40 | 40 | 40 | 40 | 40 | 47 | 47 | 51 | 57 | 74 |
| | 2 | 40 | 40 | 40 | 40 | 40 | 47 | 47 | 51 | 57 | 74 |
| | 3 | 40 | 40 | 40 | 40 | 40 | 47 | 47 | 51 | 57 | 74 |
| 79 | 4 | 40 | 40 | 40 | 40 | 40 | 47 | 47 | 51 | 57 | 74 |
| Ages 70-79 | <u>5</u> | 40 | 40 | 40 | 40 | 40 | 47 | 47 | 51 | 57 | 74 |
| ges | 6 | 44 | 44 | 44 | 44 | 44 | 51 | 51 | 54 | 60 | 78 |
| ĕ | 7 | 44 | 44 | 44 | 44 | 44 | 51 | 51 | 54 | 60 | 78 |
| | 8 | 47 | 47 | 47 | 47 | 47 | 54 | 54 | 57 | 64 | 82 |
| | 9 | 47 | 47 | 47 | 47 | 47 | 54 | 54 | 57 | 64 | 82 |
| | 10 | 51 | 51 | 51 | 51 | 51 | 57 | 57 | 60 | 68 | 85 |
| | 11 | 51 | 51 | 51 | 51 | 51 | 57 | 57 | 60 | 68 | 85 |

| | | Picture Nar | ming Total Scor | re | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| _ | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9–10 |
| | 12 | 54 | 54 | 54 | 54 | 54 | 60 | 60 | 64 | 71 | 88 |
| | 13 | 54 | 54 | 54 | 54 | 54 | 60 | 60 | 64 | 71 | 88 |
| | 14 | 57 | 57 | 57 | 57 | 57 | 64 | 64 | 68 | 75 | 90 |
| | 15 | 60 | 60 | 60 | 60 | 60 | 68 | 68 | 71 | 79 | 92 |
| | 16 | 60 | 60 | 60 | 60 | 60 | 68 | 68 | 71 | 79 | 92 |
| | 17 | 64 | 64 | 64 | 64 | 64 | 71 | 71 | 75 | 83 | 96 |
| | 18 | 64 | 64 | 64 | 64 | 64 | 71 | 71 | 75 | 83 | 96 |
| | 19 | 68 | 68 | 68 | 68 | 68 | 75 | 75 | 79 | 87 | 99 |
| | 20 | 71 | 71 | 71 | 71 | 71 | 79 | 79 | 83 | 90 | 101 |
| | 21 | 75 | 75 | 75 | 75 | 75 | 83 | 83 | 87 | 92 | 105 |
| | 22 | 75 | 75 | 75 | 75 | 75 | 83 | 83 | 87 | 92 | 105 |
| | 23 | 79 | 79 | 79 | 79 | 79 | 87 | 87 | 90 | 94 | 108 |
| | 24 | 79 | 79 | 79 | 79 | 79 | 87 | 87 | 90 | 94 | 108 |
| | 25 | 83 | 83 | 83 | 83 | 83 | 90 | 90 | 92 | 96 | 112 |
| | 26 | 83 | 83 | 83 | 83 | 83 | 90 | 90 | 92 | 96 | 112 |
| | 27 | 87 | 87 | 87 | 87 | 87 | 92 | 92 | 94 | 100 | 117 |
| | 28 | 90 | 90 | 90 | 90 | 90 | 94 | 94 | 96 | 102 | 120 |
| | 29 | 92 | 92 | 92 | 92 | 92 | 96 | 96 | 100 | 104 | 124 |
| | 30 | 92 | 92 | 92 | 92 | 92 | 96 | 96 | 100 | 104 | 124 |
| | 31 | 94 | 94 | 94 | 94 | 94 | 100 | 100 | 102 | 108 | 128 |
| | 32 | 94 | 94 | 94 | 94 | 94 | 100 | 100 | 102 | 108 | 128 |
| | 33 | 96 | 96 | 96 | 96 | 96 | 102 | 102 | 104 | 112 | 131 |
| | 34 | 100 | 100 | 100 | 100 | 100 | 104 | 104 | 108 | 116 | 134 |
| | 35 | 100 | 100 | 100 | 100 | 100 | 104 | 104 | 108 | 116 | 134 |
| | 36+ | 100 | 100 | 100 | 100 | 100 | 104 | 104 | 108 | 116 | 134 |
| | | | | | • | • | | • | | • | • |
| -08 | 0 | 40 | 40 | 40 | 40 | 40 | 47 | 51 | 54 | 57 | 76 |
| Ages<br>89 | 1 | 40 | 40 | 40 | 40 | 40 | 47 | 51 | 54 | 57 | 76 |

| | Picture Na | aming Total Scor | e | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9–10 |
| 3 | 40 | 40 | 40 | 40 | 40 | 47 | 51 | 54 | 57 | 76 |
| 4 | 40 | 40 | 40 | 40 | 40 | 47 | 51 | 54 | 57 | 76 |
| <u>5</u> | 44 | 44 | 44 | 44 | 44 | 51 | 54 | 57 | 60 | 80 |
| 6 | 44 | 44 | 44 | 44 | 44 | 51 | 54 | 57 | 60 | 80 |
| 7 | 44 | 44 | 44 | 44 | 44 | 51 | 54 | 57 | 60 | 80 |
| 8 | 47 | 47 | 47 | 47 | 47 | 54 | 57 | 60 | 64 | 83 |
| 9 | 51 | 51 | 51 | 51 | 51 | 57 | 60 | 64 | 68 | 86 |
| 10 | 51 | 51 | 51 | 51 | 51 | 57 | 60 | 64 | 68 | 86 |
| 11 | 54 | 54 | 54 | 54 | 54 | 60 | 64 | 68 | 71 | 89 |
| 12 | 57 | 57 | 57 | 57 | 57 | 64 | 68 | 71 | 75 | 92 |
| 13 | 57 | 57 | 57 | 57 | 57 | 64 | 68 | 71 | 75 | 92 |
| 14 | 60 | 60 | 60 | 60 | 60 | 68 | 71 | 75 | 79 | 95 |
| 15 | 64 | 64 | 64 | 64 | 64 | 71 | 75 | 79 | 83 | 97 |
| 16 | 68 | 68 | 68 | 68 | 68 | 75 | 79 | 83 | 87 | 99 |
| 17 | 71 | 71 | 71 | 71 | 71 | 79 | 83 | 87 | 90 | 103 |
| 18 | 71 | 71 | 71 | 71 | 71 | 79 | 83 | 87 | 90 | 103 |
| 19 | 75 | 75 | 75 | 75 | 75 | 83 | 87 | 90 | 92 | 107 |
| 20 | 79 | 79 | 79 | 79 | 79 | 87 | 90 | 92 | 94 | 110 |
| 21 | 83 | 83 | 83 | 83 | 83 | 90 | 92 | 94 | 96 | 113 |
| 22 | 87 | 87 | 87 | 87 | 87 | 92 | 94 | 96 | 100 | 117 |
| 23 | 90 | 90 | 90 | 90 | 90 | 94 | 96 | 100 | 102 | 122 |
| 24 | 90 | 90 | 90 | 90 | 90 | 94 | 96 | 100 | 102 | 122 |
| 25 | 92 | 92 | 92 | 92 | 92 | 96 | 100 | 102 | 104 | 125 |
| 26 | 92 | 92 | 92 | 92 | 92 | 96 | 100 | 102 | 104 | 125 |
| 27 | 94 | 94 | 94 | 94 | 94 | 100 | 102 | 104 | 108 | 129 |
| 28 | 94 | 94 | 94 | 94 | 94 | 100 | 102 | 104 | 108 | 129 |
| 29 | 94 | 94 | 94 | 94 | 94 | 100 | 102 | 104 | 108 | 129 |
| 30 | 96 | 96 | 96 | 96 | 96 | 102 | 104 | 108 | 112 | 133 |
| 31 | 96 | 96 | 96 | 96 | 96 | 102 | 104 | 108 | 112 | 133 |
| 32 | 96 | 96 | 96 | 96 | 96 | 102 | 104 | 108 | 112 | 133 |

| Novartis | For business use only | Page 72 |
|----------------|-----------------------|------------------------|
| SAP Addendum 4 | | CAPI015A2201J Cohort I |

| | Picture Naming Total Score | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9–10 |
| 33 | 100 | 100 | 100 | 100 | 100 | 104 | 108 | 112 | 116 | 137 |
| 34 | 100 | 100 | 100 | 100 | 100 | 104 | 108 | 112 | 116 | 137 |
| 35 | 100 | 100 | 100 | 100 | 100 | 104 | 108 | 112 | 116 | 137 |
| 36+ | 100 | 100 | 100 | 100 | 100 | 104 | 108 | 112 | 116 | 137 |
Table 5-20
 Attention Index Score Equivalents of Subtest Raw Scores

| | | | Digit \$ | Span To | otal Sco | re | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| | | 0 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 1 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 2 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 3 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 4 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 5 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 6 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 7 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 8 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 9 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 10 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 11 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 12 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| | | 13 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| | | 14 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| | | 15 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| | | 16 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| | | 17 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| <u>Je</u> | | 18 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| Scc | | 19 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |
| <u>a</u> | တ္ | 20 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |
| Coding Total Score | 50-59 | 21 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |
| ding | 3S & | 22 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |
| Co | Ages | 23 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |

| 24 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 25 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |
| 26 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 75 | 82 | 85 | 88 | 91 | 94 | 97 | 100 |
| 27 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 75 | 82 | 85 | 88 | 91 | 94 | 97 | 100 |
| 28 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 75 | 82 | 85 | 88 | 91 | 94 | 97 | 100 |
| 29 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 75 | 82 | 85 | 88 | 91 | 94 | 97 | 100 |
| 30 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 75 | 82 | 85 | 88 | 91 | 94 | 97 | 100 |
| 31 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 72 | 79 | 85 | 88 | 91 | 94 | 97 | 100 | 103 |
| 32 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 72 | 79 | 85 | 88 | 91 | 94 | 97 | 100 | 103 |
| 33 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 72 | 79 | 85 | 88 | 91 | 94 | 97 | 100 | 103 |
| 34 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 75 | 82 | 88 | 91 | 94 | 97 | 100 | 103 | 106 |
| 35 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 75 | 82 | 88 | 91 | 94 | 97 | 100 | 103 | 106 |
| 36 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 75 | 82 | 88 | 91 | 94 | 97 | 100 | 103 | 106 |
| 37 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 79 | 85 | 91 | 94 | 97 | 100 | 103 | 106 | 109 |
| 38 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 79 | 85 | 91 | 94 | 97 | 100 | 103 | 106 | 109 |
| 39 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 79 | 85 | 91 | 94 | 97 | 100 | 103 | 106 | 109 |
| 40 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 79 | 85 | 91 | 94 | 97 | 100 | 103 | 106 | 109 |
| 41 | 64 | 64 | 64 | 64 | 68 | 72 | 75 | 79 | 82 | 88 | 94 | 97 | 100 | 103 | 106 | 109 | 112 |
| 42 | 64 | 64 | 64 | 64 | 68 | 72 | 75 | 79 | 82 | 88 | 94 | 97 | 100 | 103 | 106 | 109 | 112 |
| 43 | 68 | 68 | 68 | 68 | 72 | 75 | 79 | 82 | 85 | 91 | 97 | 100 | 103 | 106 | 109 | 112 | 115 |
| 44 | 68 | 68 | 68 | 68 | 72 | 75 | 79 | 82 | 85 | 91 | 97 | 100 | 103 | 106 | 109 | 112 | 115 |
| 45 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 88 | 94 | 100 | 103 | 106 | 109 | 112 | 115 | 118 |
| 46 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 88 | 94 | 100 | 103 | 106 | 109 | 112 | 115 | 118 |
| 47 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 88 | 94 | 100 | 103 | 106 | 109 | 112 | 115 | 118 |
| 48 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 88 | 94 | 100 | 103 | 106 | 109 | 112 | 115 | 118 |
| 49 | 75 | 75 | 75 | 75 | 79 | 82 | 85 | 88 | 91 | 97 | 103 | 106 | 109 | 112 | 115 | 118 | 122 |
| 50 | 75 | 75 | 75 | 75 | 79 | 82 | 85 | 88 | 91 | 97 | 103 | 106 | 109 | 112 | 115 | 118 | 122 |

| 51 | 79 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 94 | 100 | 106 | 109 | 112 | 115 | 118 | 122 | 125 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 52 | 79 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 94 | 100 | 106 | 109 | 112 | 115 | 118 | 122 | 125 |
| 53 | 79 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 94 | 100 | 106 | 109 | 112 | 115 | 118 | 122 | 125 |
| 54 | 82 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 97 | 103 | 109 | 112 | 115 | 118 | 122 | 125 | 128 |
| 55 | 82 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 97 | 103 | 109 | 112 | 115 | 118 | 122 | 125 | 128 |
| 56 | 82 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 97 | 103 | 109 | 112 | 115 | 118 | 122 | 125 | 128 |
| 57 | 85 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 100 | 106 | 112 | 115 | 118 | 122 | 125 | 128 | 132 |
| 58 | 85 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 100 | 106 | 112 | 115 | 118 | 122 | 125 | 128 | 132 |
| 59 | 85 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 100 | 106 | 112 | 115 | 118 | 122 | 125 | 128 | 132 |
| 60 | 85 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 100 | 106 | 112 | 115 | 118 | 122 | 125 | 128 | 132 |
| 61 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 103 | 109 | 115 | 118 | 122 | 125 | 128 | 132 | 135 |
| 62 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 103 | 109 | 115 | 118 | 122 | 125 | 128 | 132 | 135 |
| 63 | 91 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 106 | 112 | 118 | 122 | 125 | 128 | 132 | 135 | 138 |
| 64 | 91 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 106 | 112 | 118 | 122 | 125 | 128 | 132 | 135 | 138 |
| 65 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 115 | 122 | 125 | 128 | 132 | 135 | 138 | 142 |
| 66 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 115 | 122 | 125 | 128 | 132 | 135 | 138 | 142 |
| 67 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 115 | 122 | 125 | 128 | 132 | 135 | 138 | 142 |
| 68 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 118 | 125 | 128 | 132 | 135 | 138 | 142 | 146 |
| 69 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 118 | 125 | 128 | 132 | 135 | 138 | 142 | 146 |
| 70 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 118 | 125 | 128 | 132 | 135 | 138 | 142 | 146 |
| 71 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 118 | 125 | 128 | 132 | 135 | 138 | 142 | 146 |
| 72 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 73 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 74 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 75 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 76 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 77 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |

| Texas Texa | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 80 | | 78 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 81 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 83 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 84 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 85 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 85 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 86 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 86 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 86 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 87 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 87 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 88 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 88 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 89 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 89 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 89 100 100 100 100 403 46 49 53 60 64 72 75 79 85 88 91 91 14 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 44 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 55 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 55 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 66 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 66 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 66 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 77 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 71 80 40 | | 79 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| Record 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 | | 80 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 83 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 84 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 85 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 86 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 87 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 88 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 89 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 89 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 89 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 1 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 2 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 3 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 4 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 5 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 6 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 7 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 7 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 43 46 49 5 | | 81 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 84 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 85 100 100 100 100 100 100 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 86 100 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 87 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 88 100 100 100 103 106 109 112 115 122 128 132 135 138 <td< td=""><td></td><td>82</td><td>100</td><td>100</td><td>100</td><td>100</td><td>103</td><td>106</td><td>109</td><td>112</td><td>115</td><td>122</td><td>128</td><td>132</td><td>135</td><td>138</td><td>142</td><td>146</td><td>150</td></td<> | | 82 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| S5 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 | | 83 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 86 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 87 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 88 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 89 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 97 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 97 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 97 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 97 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 97 100 10 | | 84 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 87 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 88 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 89 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 100 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 100 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 100 | | 85 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 88 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 89 100 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 10 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 11 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 11 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 11 40 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 11 | | 86 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 89 100 100 100 100 103 106 109 112 115 122 128 132 135 138 142 146 150 0 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 2 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 3 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 5 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 5 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 6 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 7 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 8 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 8 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 9 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 9 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 12 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 | | 87 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 0 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 2 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 3 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 4 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 5 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 6 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 7 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 8 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 9 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 9 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 40 53 66 64 88 75 79 82 88 91 94 11 43 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 | | 88 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 1 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 3 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 5 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 6 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 6 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 6 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 7 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 7 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 8 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 8 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 | | 89 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| 2 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 3 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 4 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 5 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 6 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 7 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 8 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 8 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 9 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 9 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 12 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 | | 0 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 3 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 4 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 5 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 6 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 7 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 8 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 9 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 9 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 12 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 14 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 | | 1 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 4 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 6 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 7 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 81 8 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 8 8 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 8 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 | | 2 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 5 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 7 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 8 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 8 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 9 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 60 64 68 75 79 82 88 91 94 94 12 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 13 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 | | 3 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 6 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 7 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 8 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 9 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 13 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 | | 4 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 7 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 8 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 9 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 13 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 | | 5 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 8 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 91 9 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 12 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 14 43 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 14 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 14 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 | | 6 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 9 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 12 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 13 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 | | 7 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 10 40 40 40 40 43 46 49 53 60 64 72 75 79 85 88 91 91 11 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 12 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 13 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 14 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 14 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 14 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 | | 8 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 11 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 12 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 13 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 | | 9 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 12 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 13 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 14 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 14 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94 | | 10 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 12 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94<br>13 43 43 43 43 46 49 53 56 64 68 75 79 82 88 91 94 94<br>14 43 43 43 44 45 49 53 56 64 68 75 79 82 88 91 94 94 | <b>o</b> | 11 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 13 43 43 43 44 45 45 45 56 64 68 75 79 82 88 91 94 94 14 43 43 43 44 45 49 53 56 64 68 75 79 82 88 91 94 94 | 9-0 | 12 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 14 43 43 43 44 49 53 56 64 68 75 79 82 88 91 94 94 | 9 88 | 13 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| | Agé | 14 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |

| <br>• | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 15 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 16 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 17 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 18 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 19 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 20 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 21 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 22 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 23 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 24 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 25 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 26 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 27 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 28 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 75 | 79 | 85 | 88 | 91 | 97 | 100 | 103 | 103 |
| 29 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 75 | 79 | 85 | 88 | 91 | 97 | 100 | 103 | 103 |
| 30 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 75 | 79 | 85 | 88 | 91 | 97 | 100 | 103 | 103 |
| 31 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 75 | 79 | 85 | 88 | 91 | 97 | 100 | 103 | 103 |
| 32 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 33 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 34 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 35 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 36 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 37 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 38 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 39 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 40 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 41 | 64 | 64 | 64 | 64 | 68 | 72 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |

| <u> </u> | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 42 | 64 | 64 | 64 | 64 | 68 | 72 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |
| | 43 | 68 | 68 | 68 | 68 | 72 | 75 | 79 | 82 | 88 | 91 | 97 | 100 | 103 | 109 | 112 | 115 | 115 |
| | 44 | 68 | 68 | 68 | 68 | 72 | 75 | 79 | 82 | 88 | 91 | 97 | 100 | 103 | 109 | 112 | 115 | 115 |
| | 45 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| | 46 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| | 47 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| | 48 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| | 49 | 75 | 75 | 75 | 75 | 79 | 82 | 85 | 88 | 94 | 97 | 103 | 106 | 109 | 115 | 118 | 122 | 122 |
| | 50 | 79 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 97 | 100 | 106 | 109 | 112 | 118 | 122 | 125 | 125 |
| | 51 | 79 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 97 | 100 | 106 | 109 | 112 | 118 | 122 | 125 | 125 |
| | 52 | 82 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 100 | 103 | 109 | 112 | 115 | 122 | 125 | 128 | 128 |
| | 53 | 82 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 100 | 103 | 109 | 112 | 115 | 122 | 125 | 128 | 128 |
| | 54 | 85 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 103 | 106 | 112 | 115 | 118 | 125 | 128 | 132 | 132 |
| | 55 | 85 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 103 | 106 | 112 | 115 | 118 | 125 | 128 | 132 | 132 |
| | 56 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 106 | 109 | 115 | 118 | 122 | 128 | 132 | 135 | 135 |
| | 57 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 106 | 109 | 115 | 118 | 122 | 128 | 132 | 135 | 135 |
| | 58 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 106 | 109 | 115 | 118 | 122 | 128 | 132 | 135 | 135 |
| | 59 | 91 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 109 | 112 | 118 | 122 | 125 | 132 | 135 | 138 | 138 |
| | 60 | 91 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 109 | 112 | 118 | 122 | 125 | 132 | 135 | 138 | 138 |
| | 61 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| | 62 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| | 63 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| | 64 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| | 65 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| | 66 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| | 67 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| | 68 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |

| | 69 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 70 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 71 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 72 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 73 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 74 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 75 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 76 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 77 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 78 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 79 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 80 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 81 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 82 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 83 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 84 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 85 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 86 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 87 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 88 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 89 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 92-02 | 0 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 02 | 1 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| Ages | 2 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| Ĭ ₹ | 3 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | 4 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | 5 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |

| <br> | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 6 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 7 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 8 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 9 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 10 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 11 | 43 | 43 | 43 | 46 | 49 | 53 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 12 | 43 | 43 | 43 | 46 | 49 | 53 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 13 | 43 | 43 | 43 | 46 | 49 | 53 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 14 | 43 | 43 | 43 | 46 | 49 | 53 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 15 | 43 | 43 | 43 | 46 | 49 | 53 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 16 | 43 | 43 | 43 | 46 | 49 | 53 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 17 | 46 | 46 | 46 | 49 | 53 | 56 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 18 | 46 | 46 | 46 | 49 | 53 | 56 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 19 | 46 | 46 | 46 | 49 | 53 | 56 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 20 | 49 | 49 | 49 | 53 | 56 | 60 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 21 | 49 | 49 | 49 | 53 | 56 | 60 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 22 | 49 | 49 | 49 | 53 | 56 | 60 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 23 | 53 | 53 | 53 | 56 | 60 | 64 | 64 | 68 | 75 | 79 | 85 | 88 | 91 | 97 | 100 | 103 | 103 |
| 24 | 53 | 53 | 53 | 56 | 60 | 64 | 64 | 68 | 75 | 79 | 85 | 88 | 91 | 97 | 100 | 103 | 103 |
| 25 | 56 | 56 | 56 | 60 | 64 | 68 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 26 | 56 | 56 | 56 | 60 | 64 | 68 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 27 | 56 | 56 | 56 | 60 | 64 | 68 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 28 | 60 | 60 | 60 | 64 | 68 | 72 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 29 | 60 | 60 | 60 | 64 | 68 | 72 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 30 | 60 | 60 | 60 | 64 | 68 | 72 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 31 | 60 | 60 | 60 | 64 | 68 | 72 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 32 | 64 | 64 | 64 | 68 | 72 | 75 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |

| 33 | 64 | 64 | 64 | 68 | 72 | 75 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 34 | 64 | 64 | 64 | 68 | 72 | 75 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |
| 35 | 64 | 64 | 64 | 68 | 72 | 75 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |
| 36 | 64 | 64 | 64 | 68 | 72 | 75 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |
| 37 | 68 | 68 | 68 | 72 | 75 | 79 | 79 | 82 | 88 | 91 | 97 | 100 | 103 | 109 | 112 | 115 | 115 |
| 38 | 68 | 68 | 68 | 72 | 75 | 79 | 79 | 82 | 88 | 91 | 97 | 100 | 103 | 109 | 112 | 115 | 115 |
| 39 | 68 | 68 | 68 | 72 | 75 | 79 | 79 | 82 | 88 | 91 | 97 | 100 | 103 | 109 | 112 | 115 | 115 |
| 40 | 72 | 72 | 72 | 75 | 79 | 82 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| 41 | 72 | 72 | 72 | 75 | 79 | 82 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| 42 | 72 | 72 | 72 | 75 | 79 | 82 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| 43 | 75 | 75 | 75 | 79 | 82 | 85 | 85 | 88 | 94 | 97 | 103 | 106 | 109 | 115 | 118 | 122 | 122 |
| 44 | 75 | 75 | 75 | 79 | 82 | 85 | 85 | 88 | 94 | 97 | 103 | 106 | 109 | 115 | 118 | 122 | 122 |
| 45 | 75 | 75 | 75 | 79 | 82 | 85 | 85 | 88 | 94 | 97 | 103 | 106 | 109 | 115 | 118 | 122 | 122 |
| 46 | 79 | 79 | 79 | 82 | 85 | 88 | 88 | 91 | 97 | 100 | 106 | 109 | 112 | 118 | 122 | 125 | 125 |
| 47 | 79 | 79 | 79 | 82 | 85 | 88 | 88 | 91 | 97 | 100 | 106 | 109 | 112 | 118 | 122 | 125 | 125 |
| 48 | 82 | 82 | 82 | 85 | 88 | 91 | 91 | 94 | 100 | 103 | 109 | 112 | 115 | 122 | 125 | 128 | 128 |
| 49 | 82 | 82 | 82 | 85 | 88 | 91 | 91 | 94 | 100 | 103 | 109 | 112 | 115 | 122 | 125 | 128 | 128 |
| 50 | 82 | 82 | 82 | 85 | 88 | 91 | 91 | 94 | 100 | 103 | 109 | 112 | 115 | 122 | 125 | 128 | 128 |
| 51 | 85 | 85 | 85 | 88 | 91 | 94 | 94 | 97 | 103 | 106 | 112 | 115 | 118 | 125 | 128 | 132 | 132 |
| 52 | 85 | 85 | 85 | 88 | 91 | 94 | 94 | 97 | 103 | 106 | 112 | 115 | 118 | 125 | 128 | 132 | 132 |
| 53 | 85 | 85 | 85 | 88 | 91 | 94 | 94 | 97 | 103 | 106 | 112 | 115 | 118 | 125 | 128 | 132 | 132 |
| 54 | 88 | 88 | 88 | 91 | 94 | 97 | 97 | 100 | 106 | 109 | 115 | 118 | 122 | 128 | 132 | 135 | 135 |
| 55 | 88 | 88 | 88 | 91 | 94 | 97 | 97 | 100 | 106 | 109 | 115 | 118 | 122 | 128 | 132 | 135 | 135 |
| 56 | 88 | 88 | 88 | 91 | 94 | 97 | 97 | 100 | 106 | 109 | 115 | 118 | 122 | 128 | 132 | 135 | 135 |
| 57 | 91 | 91 | 91 | 94 | 97 | 100 | 100 | 103 | 109 | 112 | 118 | 122 | 125 | 132 | 135 | 138 | 138 |
| 58 | 91 | 91 | 91 | 94 | 97 | 100 | 100 | 103 | 109 | 112 | 118 | 122 | 125 | 132 | 135 | 138 | 138 |
| 59 | 91 | 91 | 91 | 94 | 97 | 100 | 100 | 103 | 109 | 112 | 118 | 122 | 125 | 132 | 135 | 138 | 138 |

| 60 | 91 | 91 | 91 | 94 | 97 | 100 | 100 | 103 | 109 | 112 | 118 | 122 | 125 | 132 | 135 | 138 | 138 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 61 | 94 | 94 | 94 | 97 | 100 | 103 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| 62 | 94 | 94 | 94 | 97 | 100 | 103 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| 63 | 94 | 94 | 94 | 97 | 100 | 103 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| 64 | 97 | 97 | 97 | 100 | 103 | 106 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| 65 | 97 | 97 | 97 | 100 | 103 | 106 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| 66 | 97 | 97 | 97 | 100 | 103 | 106 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| 67 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 68 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 69 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 70 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 71 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 72 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 73 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 74 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 75 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 76 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 77 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 78 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 79 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 80 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 81 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 82 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 83 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 84 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 85 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 86 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |

| | 87 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 88 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 89 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 0 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| | 1 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| | 2 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| | 3 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| | 4 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| | 5 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| | 6 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| | 7 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| | 8 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| | 9 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| | 10 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 72 | 75 | 82 | 85 | 88 | 91 | 91 | 94 | 97 |
| | 11 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 72 | 75 | 82 | 85 | 88 | 91 | 91 | 94 | 97 |
| | 12 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 72 | 75 | 82 | 85 | 88 | 91 | 91 | 94 | 97 |
| | 13 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 72 | 75 | 82 | 85 | 88 | 91 | 91 | 94 | 97 |
| | 14 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 72 | 75 | 82 | 85 | 88 | 91 | 91 | 94 | 97 |
| | 15 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 72 | 75 | 82 | 85 | 88 | 91 | 91 | 94 | 97 |
| | 16 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 75 | 79 | 85 | 88 | 91 | 94 | 94 | 97 | 100 |
| | 17 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 75 | 79 | 85 | 88 | 91 | 94 | 94 | 97 | 100 |
| | 18 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 75 | 79 | 85 | 88 | 91 | 94 | 94 | 97 | 100 |
| | 19 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 79 | 82 | 88 | 91 | 94 | 97 | 97 | 100 | 103 |
| 0 | 20 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 79 | 82 | 88 | 91 | 94 | 97 | 97 | 100 | 103 |
| 8-0 | 21 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 79 | 82 | 88 | 91 | 94 | 97 | 97 | 100 | 103 |
| ges 80-89 | 22 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 72 | 82 | 85 | 91 | 94 | 97 | 100 | 100 | 103 | 106 |
| Age | 23 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 72 | 82 | 85 | 91 | 94 | 97 | 100 | 100 | 103 | 106 |

| · | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 24 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 75 | 85 | 88 | 94 | 97 | 100 | 103 | 103 | 106 | 109 |
| | 25 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 75 | 85 | 88 | 94 | 97 | 100 | 103 | 103 | 106 | 109 |
| | 26 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 75 | 85 | 88 | 94 | 97 | 100 | 103 | 103 | 106 | 109 |
| | 27 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 79 | 88 | 91 | 97 | 100 | 103 | 106 | 106 | 109 | 112 |
| | 28 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 79 | 88 | 91 | 97 | 100 | 103 | 106 | 106 | 109 | 112 |
| | 29 | 64 | 64 | 64 | 68 | 72 | 75 | 79 | 82 | 91 | 94 | 100 | 103 | 106 | 109 | 109 | 112 | 115 |
| | 30 | 64 | 64 | 64 | 68 | 72 | 75 | 79 | 82 | 91 | 94 | 100 | 103 | 106 | 109 | 109 | 112 | 115 |
| | 31 | 68 | 68 | 68 | 72 | 75 | 79 | 82 | 85 | 94 | 97 | 103 | 106 | 109 | 112 | 112 | 115 | 118 |
| | 32 | 68 | 68 | 68 | 72 | 75 | 79 | 82 | 85 | 94 | 97 | 103 | 106 | 109 | 112 | 112 | 115 | 118 |
| | 33 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 88 | 97 | 100 | 106 | 109 | 112 | 115 | 115 | 118 | 122 |
| | 34 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 88 | 97 | 100 | 106 | 109 | 112 | 115 | 115 | 118 | 122 |
| | 35 | 75 | 75 | 75 | 79 | 82 | 85 | 88 | 91 | 100 | 103 | 109 | 112 | 115 | 118 | 118 | 122 | 125 |
| | 36 | 75 | 75 | 75 | 79 | 82 | 85 | 88 | 91 | 100 | 103 | 109 | 112 | 115 | 118 | 118 | 122 | 125 |
| | 37 | 75 | 75 | 75 | 79 | 82 | 85 | 88 | 91 | 100 | 103 | 109 | 112 | 115 | 118 | 118 | 122 | 125 |
| | 38 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 94 | 103 | 106 | 112 | 115 | 118 | 122 | 122 | 125 | 128 |
| | 39 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 94 | 103 | 106 | 112 | 115 | 118 | 122 | 122 | 125 | 128 |
| | 40 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 97 | 106 | 109 | 115 | 118 | 122 | 125 | 125 | 128 | 132 |
| | 41 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 97 | 106 | 109 | 115 | 118 | 122 | 125 | 125 | 128 | 132 |
| | 42 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 100 | 109 | 112 | 118 | 122 | 125 | 128 | 128 | 132 | 135 |
| | 43 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 100 | 109 | 112 | 118 | 122 | 125 | 128 | 128 | 132 | 135 |
| | 44 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 103 | 112 | 115 | 122 | 125 | 128 | 132 | 132 | 135 | 138 |
| | 45 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 103 | 112 | 115 | 122 | 125 | 128 | 132 | 132 | 135 | 138 |
| | 46 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 106 | 115 | 118 | 125 | 128 | 132 | 135 | 135 | 138 | 142 |
| | 47 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 106 | 115 | 118 | 125 | 128 | 132 | 135 | 135 | 138 | 142 |
| | 48 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 106 | 115 | 118 | 125 | 128 | 132 | 135 | 135 | 138 | 142 |
| | 49 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 118 | 122 | 128 | 132 | 135 | 138 | 138 | 142 | 146 |
| | 50 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 118 | 122 | 128 | 132 | 135 | 138 | 138 | 142 | 146 |

| <b>-</b> 4 | 0.4 | 0.4 | 0.4 | 0.7 | 400 | 400 | 400 | 400 | 440 | 400 | 400 | 400 | 405 | 400 | 400 | 440 | 140 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 51 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 118 | 122 | 128 | 132 | 135 | 138 | 138 | 142 | 146 |
| 52 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 118 | 122 | 128 | 132 | 135 | 138 | 138 | 142 | 146 |
| 53 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 122 | 125 | 132 | 135 | 138 | 142 | 142 | 146 | 150 |
| 54 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 122 | 125 | 132 | 135 | 138 | 142 | 142 | 146 | 150 |
| 55 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 122 | 125 | 132 | 135 | 138 | 142 | 142 | 146 | 150 |
| 56 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 122 | 125 | 132 | 135 | 138 | 142 | 142 | 146 | 150 |
| 57 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 122 | 125 | 132 | 135 | 138 | 142 | 142 | 146 | 150 |
| 58 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 59 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 60 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 61 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 62 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 63 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 64 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 65 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 66 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 67 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 68 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 69 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 70 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 71 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 72 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 73 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 74 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 75 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 76 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 77 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| L ' ' | | | | | .00 | | | | | 120 | .00 | | | 1 10 | 1.10 | 100 | ٠٠. |

| Novartis | For business use only | Page 86 |
|----------------|-----------------------|------------------------|
| SAP Addendum 4 | | CAPI015A2201J Cohort I |

| 78 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 79 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 80 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 81 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 82 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 83 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 84 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 85 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 86 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 87 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 88 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 89 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |

Table 5-21 Delayed Memory Index Score Equivalents of Subtest Raw Scores

| | | | List | Recog | gnition | n Tota | Scor | <b>e</b> | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19–<br>20 |
| | | 0 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| | | 1 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| | | 2 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| | | 3 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| | | 4 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| | | 5 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| | | 6 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| | | 7 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| ore | | 8 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 48 | 52 | 52 | 56 | 64 | 80 |
| Score | | 9 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 48 | 52 | 52 | 56 | 64 | 80 |
| Total | | 10 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 52 | 56 | 56 | 60 | 68 | 82 |
| | | 11 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 52 | 56 | 56 | 60 | 68 | 82 |
| nre | | 12 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 52 | 56 | 56 | 60 | 68 | 82 |
| Fig | | 13 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 56 | 60 | 60 | 64 | 71 | 85 |
| ry/ | | 14 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 56 | 60 | 60 | 64 | 71 | 85 |
| of List/Story/ Figure | | 15 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 60 | 60 | 64 | 64 | 68 | 75 | 88 |
| ist/; | -59 | 16 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 64 | 68 | 68 | 71 | 78 | 91 |
| of L | <del>2</del> 0-4 | 17 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 64 | 68 | 68 | 71 | 78 | 91 |
| m c | səb | 18 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 64 | 68 | 68 | 71 | 78 | 91 |
| Sum | Ag | 19 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 64 | 68 | 68 | 71 | 78 | 91 |

| | | List | Reco | nitior | 1 Tota | l Scor | е | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19-<br>20 |
| | 20 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 64 | 68 | 68 | 71 | 78 | 91 |
| = | 21 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 68 | 71 | 71 | 75 | 81 | 94 |
| | 22 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 68 | 71 | 71 | 75 | 81 | 94 |
| | 23 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 68 | 71 | 71 | 75 | 81 | 94 |
| | 24 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 68 | 71 | 71 | 75 | 81 | 94 |
| _ | 25 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 71 | 75 | 75 | 78 | 84 | 97 |
| | 26 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 71 | 75 | 75 | 78 | 84 | 97 |
| | 27 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 75 | 78 | 78 | 81 | 86 | 99 |
| | 28 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 75 | 78 | 78 | 81 | 86 | 99 |
| _ | 29 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 78 | 81 | 81 | 84 | 88 | 101 |
| | 30 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 78 | 81 | 81 | 84 | 88 | 101 |
| | 31 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 81 | 84 | 84 | 86 | 91 | 105 |
| | 32 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 81 | 84 | 84 | 86 | 91 | 105 |
| | 33 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 84 | 86 | 86 | 88 | 94 | 108 |
| | 34 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 84 | 86 | 86 | 88 | 94 | 108 |
| | 35 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 86 | 88 | 88 | 91 | 97 | 111 |
| - | 36 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 88 | 88 | 91 | 91 | 94 | 100 | 115 |
| | 37 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 91 | 94 | 94 | 97 | 102 | 119 |
| | 38 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 91 | 94 | 94 | 97 | 102 | 119 |
| | 39 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 94 | 97 | 97 | 100 | 104 | 124 |
| | 40 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 94 | 97 | 97 | 100 | 104 | 124 |
| | 41 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 102 | 108 | 127 |
| | 42 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 100 | 100 | 102 | 102 | 104 | 112 | 131 |
| Ag | 0 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |

| | List | Recog | nitior | n Tota | l Scor | е | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19-<br>20 |
| 1 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| 2 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| 3 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| 4 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| 5 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| 6 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| 7 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 52 | 60 | 64 | 81 |
| 8 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 52 | 60 | 64 | 81 |
| 9 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 52 | 60 | 64 | 81 |
| 10 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 56 | 56 | 64 | 68 | 84 |
| 11 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 56 | 56 | 64 | 68 | 84 |
| 12 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 56 | 56 | 64 | 68 | 84 |
| 13 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 60 | 60 | 60 | 68 | 71 | 86 |
| 14 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 60 | 60 | 60 | 68 | 71 | 86 |
| 15 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 60 | 64 | 64 | 64 | 71 | 75 | 89 |
| 16 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 68 | 68 | 75 | 78 | 92 |
| 17 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 68 | 68 | 75 | 78 | 92 |
| 18 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 68 | 68 | 75 | 78 | 92 |
| 19 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 71 | 78 | 81 | 95 |
| 20 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 71 | 78 | 81 | 95 |
| 21 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 71 | 78 | 81 | 95 |
| 22 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 71 | 78 | 81 | 95 |
| 23 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 75 | 75 | 81 | 84 | 98 |
| 24 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 75 | 75 | 81 | 84 | 98 |

| | | List | Recog | gnition | n Tota | l Scor | е | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19-<br>20 |
| | 25 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 75 | 75 | 81 | 84 | 98 |
| | 26 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 78 | 78 | 84 | 86 | 100 |
| | 27 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 78 | 78 | 84 | 86 | 100 |
| | 28 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 81 | 81 | 86 | 88 | 102 |
| | 29 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 81 | 81 | 86 | 88 | 102 |
| | 30 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 81 | 81 | 86 | 88 | 102 |
| | 31 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 84 | 84 | 88 | 91 | 106 |
| | 32 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 84 | 84 | 88 | 91 | 106 |
| | 33 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 86 | 86 | 86 | 91 | 94 | 110 |
| | 34 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 88 | 88 | 94 | 97 | 112 |
| | 35 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 88 | 88 | 94 | 97 | 112 |
| | 36 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 88 | 91 | 91 | 91 | 97 | 100 | 116 |
| | 37 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 94 | 94 | 100 | 102 | 121 |
| | 38 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 94 | 94 | 100 | 102 | 121 |
| | 39 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 97 | 97 | 97 | 102 | 104 | 126 |
| | 40 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 97 | 97 | 97 | 102 | 104 | 126 |
| | 41 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 97 | 100 | 100 | 100 | 104 | 108 | 129 |
| | 42 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 100 | 102 | 102 | 102 | 108 | 112 | 133 |
| L | 0 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 52 | 56 | 60 | 79 |
| L | 1 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 52 | 56 | 60 | 79 |
| 62 | 2 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 52 | 56 | 60 | 79 |
| Ages 70-79 | 3 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 52 | 56 | 60 | 79 |
| es | 4 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 52 | 56 | 60 | 79 |
| Ag | 5 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 56 | 60 | 64 | 82 |

| | List | Recog | gnitio | n Tota | l Scor | е | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19-<br>20 |
| 6 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 56 | 60 | 64 | 82 |
| 7 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 56 | 60 | 64 | 82 |
| 8 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 56 | 60 | 64 | 82 |
| 9 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 56 | 60 | 64 | 68 | 85 |
| 10 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 56 | 60 | 64 | 68 | 85 |
| 11 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 56 | 60 | 64 | 68 | 85 |
| 12 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 60 | 60 | 64 | 68 | 71 | 87 |
| 13 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 60 | 60 | 64 | 68 | 71 | 87 |
| 14 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 60 | 64 | 64 | 68 | 71 | 75 | 90 |
| 15 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 68 | 71 | 75 | 78 | 93 |
| 16 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 68 | 71 | 75 | 78 | 93 |
| 17 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 68 | 71 | 75 | 78 | 93 |
| 18 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 75 | 78 | 81 | 95 |
| 19 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 75 | 78 | 81 | 95 |
| 20 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 75 | 78 | 81 | 95 |
| 21 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 75 | 78 | 81 | 84 | 98 |
| 22 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 75 | 78 | 81 | 84 | 98 |
| 23 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 78 | 81 | 84 | 86 | 101 |
| 24 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 78 | 81 | 84 | 86 | 101 |
| 25 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 78 | 81 | 84 | 86 | 101 |
| 26 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 81 | 84 | 86 | 88 | 103 |
| 27 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 81 | 84 | 86 | 88 | 103 |
| 28 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 84 | 86 | 88 | 91 | 107 |
| 29 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 84 | 86 | 88 | 91 | 107 |

| | | List | Recog | nition | Total | Score | 9 | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19–<br>20 |
| | 30 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 86 | 86 | 88 | 91 | 94 | 110 |
| | 31 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 86 | 86 | 88 | 91 | 94 | 110 |
| | 32 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 88 | 91 | 94 | 97 | 113 |
| | 33 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 88 | 91 | 94 | 97 | 113 |
| | 34 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 88 | 91 | 91 | 94 | 97 | 100 | 117 |
| | 35 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 88 | 91 | 91 | 94 | 97 | 100 | 117 |
| | 36 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 94 | 97 | 100 | 102 | 122 |
| | 37 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 94 | 97 | 100 | 102 | 122 |
| | 38 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 94 | 97 | 100 | 102 | 122 |
| | 39 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 97 | 97 | 100 | 102 | 104 | 127 |
| | 40 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 97 | 100 | 100 | 102 | 104 | 108 | 130 |
| | 41 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 100 | 102 | 102 | 104 | 108 | 112 | 134 |
| | 42 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 102 | 104 | 104 | 108 | 112 | 115 | 137 |
| | 0 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 52 | 52 | 56 | 64 | 80 |
| | 1 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 52 | 52 | 56 | 64 | 80 |
| | 2 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 56 | 56 | 60 | 68 | 82 |
| | 3 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 56 | 56 | 60 | 68 | 82 |
| | 4 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 56 | 56 | 60 | 68 | 82 |
| | 5 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 60 | 60 | 64 | 71 | 85 |
| | 6 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 60 | 60 | 64 | 71 | 85 |
| 83 | 7 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 60 | 60 | 64 | 71 | 85 |
| 80-89 | 8 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 60 | 64 | 64 | 68 | 75 | 88 |
| Ages | 9 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 60 | 64 | 64 | 68 | 75 | 88 |
| Ag | 10 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 68 | 71 | 78 | 90 |

| | Lis | t Reco | gnitio | n Tota | l Scor | е | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19–<br>20 |
| - | <b>1</b> 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 68 | 71 | 78 | 90 |
| • | <b>2</b> 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 68 | 71 | 78 | 90 |
| | <b>3</b> 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 71 | 71 | 75 | 81 | 93 |
| | <b>4</b> 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 71 | 71 | 75 | 81 | 93 |
| | <b>5</b> 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 75 | 75 | 78 | 84 | 96 |
| | <b>6</b> 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 75 | 75 | 78 | 84 | 96 |
| | <b>7</b> 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 78 | 78 | 81 | 86 | 98 |
| | <b>8</b> 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 78 | 78 | 81 | 86 | 98 |
| | 9 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 81 | 81 | 84 | 88 | 101 |
| 2 | <b>10</b> 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 81 | 81 | 84 | 88 | 101 |
| 1 | 2 <b>1</b> 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 81 | 81 | 84 | 88 | 101 |
| 2 | <b>2</b> 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 84 | 84 | 86 | 91 | 104 |
| 2 | <b>3</b> 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 84 | 84 | 86 | 91 | 104 |
| 2 | 4 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 84 | 84 | 86 | 91 | 104 |
| 1 | <b>.5</b> 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 86 | 86 | 88 | 94 | 107 |
| 1 | <b>16</b> 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 86 | 86 | 88 | 94 | 107 |
| 2 | ? <b>7</b> 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 86 | 86 | 88 | 94 | 107 |
| 2 | <b>8</b> 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 86 | 88 | 88 | 91 | 97 | 110 |
| <u> :</u> | <b>9</b> 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 86 | 88 | 88 | 91 | 97 | 110 |
| <u> </u> | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 91 | 91 | 94 | 100 | 114 |
| <u>;</u> | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 91 | 91 | 94 | 100 | 114 |
| <u>;</u> | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 91 | 91 | 94 | 100 | 114 |
| <u>;</u> | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 88 | 91 | 94 | 94 | 97 | 102 | 119 |
| | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 88 | 91 | 94 | 94 | 97 | 102 | 119 |

| | List | Recog | nition | Total | Score | е | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19-<br>20 |
| 35 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 97 | 100 | 104 | 123 |
| 36 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 97 | 100 | 104 | 123 |
| 37 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 97 | 100 | 100 | 102 | 108 | 126 |
| 38 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 97 | 100 | 100 | 102 | 108 | 126 |
| 39 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 97 | 100 | 102 | 102 | 104 | 112 | 131 |
| 40 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 97 | 100 | 102 | 102 | 104 | 112 | 131 |
| 41 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 100 | 102 | 104 | 104 | 108 | 115 | 134 |
| 42 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 102 | 104 | 108 | 108 | 112 | 119 | 137 |

The RBANS Total scores (Total Scale of Index scores) corresponds to the Sum of Index scores in the table below.

Table 5-22 Total Scale Index Score Equivalents of Sum of Index Scores

| Sum of Index<br>Scores | Total Scale<br>of Index<br>Scores | Percentiles | Sum of<br>Index<br>Scores | Total<br>Scale of<br>Index<br>Scores | Percentiles | Sum of Index<br>Scores | Total<br>Scale of<br>Index<br>Scores | Percentiles |
|---|---|---|---|---|---|---|---|---|
| 200–207 | 40 | <0.1 | 427–430 | 81 | 10 | 574–576 | 122 | 93 |
| 208–215 | 41 | <0.1 | 431–435 | 82 | 12 | 577–580 | 123 | 94 |
| 216–223 | 42 | <0.1 | 436–440 | 83 | 13 | 581–583 | 124 | 95 |
| 224–231 | 43 | <0.1 | 441–444 | 84 | 14 | 584–586 | 125 | 95 |
| 232–239 | 44 | <0.1 | 445–449 | 85 | 16 | 587–588 | 126 | 96 |
| 240–247 | 45 | <0.1 | 450–454 | 86 | 18 | 589–591 | 127 | 96 |

| Sum of Index<br>Scores | Total Scale<br>of Index<br>Scores | Percentiles | Sum of<br>Index<br>Scores | Total<br>Scale of<br>Index<br>Scores | Percentiles | Sum of Index<br>Scores | Total<br>Scale of<br>Index<br>Scores | Percentiles |
|---|---|---|---|---|---|---|---|---|
| 248–255 | 46 | <0.1 | 455–458 | 87 | 19 | 592–593 | 128 | 97 |
| 256–263 | 47 | <0.1 | 459–461 | 88 | 21 | 594–596 | 129 | 97 |
| 264–271 | 48 | <0.1 | 462-464 | 89 | 23 | 597–598 | 130 | 98 |
| 272–279 | 49 | <0.1 | 465–468 | 90 | 25 | 599–600 | 131 | 98 |
| 280–287 | 50 | <0.1 | 469–471 | 91 | 27 | 601–602 | 132 | 98 |
| 288–295 | 51 | 0.1 | 472–475 | 92 | 30 | 603–604 | 133 | 99 |
| 296–303 | 52 | 0.1 | 476–479 | 93 | 32 | 605–606 | 134 | 99 |
| 304–311 | 53 | 0.1 | 480–483 | 94 | 34 | 607–608 | 135 | 99 |
| 312–319 | 54 | 0.1 | 484–487 | 95 | 37 | 609–610 | 136 | 99 |
| 320–327 | 55 | 0.1 | 488–490 | 96 | 39 | 611–612 | 137 | 99 |
| 328–330 | 56 | 0.2 | 491–493 | 97 | 42 | 613 | 138 | 99 |
| 331–333 | 57 | 0.2 | 494–496 | 98 | 45 | 614–615 | 139 | 99.5 |
| 334–336 | 58 | 0.3 | 497–499 | 99 | 47 | 616–617 | 140 | 99.6 |
| 337–339 | 59 | 0.3 | 500-505 | 100 | 50 | 618–619 | 141 | 99.7 |
| 340–343 | 60 | 0.4 | 506-509 | 101 | 53 | 620–621 | 142 | 99.7 |
| 344–347 | 61 | 0.5 | 510–513 | 102 | 55 | 622–624 | 143 | 99.8 |
| 348–351 | 62 | 1 | 514–516 | 103 | 58 | 625–628 | 144 | 99.8 |
| 352–355 | 63 | 1 | 517–520 | 104 | 61 | 629–632 | 145 | 99.9 |
| 356–359 | 64 | 1 | 521–523 | 105 | 63 | 633–636 | 146 | 99.9 |
| 360–363 | 65 | 1 | 524-527 | 106 | 66 | 637–639 | 147 | 99.9 |
| 364–367 | 66 | 1 | 528-530 | 107 | 68 | 640–651 | 148 | 99.9 |
| 368–372 | 67 | 1 | 531–533 | 108 | 70 | 652–663 | 149 | 99.9 |
| 373–376 | 68 | 2 | 534-536 | 109 | 73 | 664–675 | 150 | >99.9 |

| Sum of Index<br>Scores | Total Scale<br>of Index<br>Scores | Percentiles | Sum of<br>Index<br>Scores | Total<br>Scale of<br>Index<br>Scores | Percentiles | Sum of Index<br>Scores | Total<br>Scale of<br>Index<br>Scores | Percentiles |
|---|---|---|---|---|---|---|---|---|
| 377–380 | 69 | 2 | 537–539 | 110 | 75 | 676–687 | 151 | >99.9 |
| 381–384 | 70 | 2 | 540-542 | 111 | 77 | 688–699 | 152 | >99.9 |
| 385–387 | 71 | 3 | 543-545 | 112 | 79 | 700–711 | 153 | >99.9 |
| 388–391 | 72 | 3 | 546-548 | 113 | 81 | 712–723 | 154 | >99.9 |
| 392–394 | 73 | 4 | 549-551 | 114 | 82 | 724–735 | 155 | >99.9 |
| 395–398 | 74 | 4 | 552-554 | 115 | 84 | 736–748 | 156 | >99.9 |
| 399–402 | 75 | 5 | 555–556 | 116 | 86 | 749–761 | 157 | >99.9 |
| 403–405 | 76 | 5 | 557–559 | 117 | 87 | 762–774 | 158 | >99.9 |
| 406–409 | 77 | 6 | 560-562 | 118 | 88 | 775–787 | 159 | >99.9 |
| 410–414 | 78 | 7 | 563-566 | 119 | 90 | 788–800 | 160 | >99.9 |
| 415–419 | 79 | 8 | 567–570 | 120 | 91 | | | |
| 420–426 | 80 | 9 | 571–573 | 121 | 92 | | | |

### 6 References

Folstein MF, Folstein SE, McHugh PR (1975) A practical method for grading the cognitive state of patients for the clinician. J. psychiat. Res.; 12:189-98.

Raven JC (2000) Standard Progressive Matrices-1998 Edition, updated 2000. Manual for Standard Progressive Matrices (Section 3): NCS Person, Inc.; San Antonio.

Farias ST, Mungas D, Reed BR, et al (2008) The measurement of everyday cognition (ECog): Scale development and psychometric properties. Neuropsychology; 22(4):531-44.

Klunk et al. The Centiloid Project: Standardizing quantitative amyloid plaque estimation by PET. Alzheimer and Dementia 2015 (11): 1-15.



### Clinical Development

## CNP520A (Cohort II)

#### CAPI015A2201J

# A randomized, double-blind, placebo-controlled, twocohort parallel group study to evaluate the efficacy of CAD106 and CNP520 in participants at risk for the onset of clinical symptoms of Alzheimer's disease

Statistical Analysis Plan (SAP)

Author: Trial Statistician

Document type: SAP Documentation

Document status: Final Addendum 2

Release date: 02-Dec-2020

Number of pages: 100

Property of Novartis
For business use only
May not be used, divulged, published or otherwise disclosed
without the consent of Novartis

## **Document History – Changes compared to previous final version of SAP**

| Date | Time<br>point | Reason for update | Outcome for update | Section and title impacted (Current) |
|---|---|---|---|---|
| 12-<br>Jun-<br>2020 | Prior<br>to<br>DB<br>Lock | Finalizing<br>the<br>Amendment<br>1 | Aligned the analysis and reporting strategy with Generation Study 2, updates from discussions with Clinical team, Stats reporting team, Medical writing team. | |
| 22-<br>Jun-<br>2020 | Prior<br>to<br>DB | Creation of amendment 2 | Updated the derivation of Annualized percent change for Volumetric MRI reporting in section 2.5.2 | |
| | Lock | ck | Added note for handling of missing severity of AE in section 2.8.1 | |
| 23-<br>Jun- | Prior<br>to | Creation of amendment | Updated the typo in "Prior" in Time point column in document history | |
| 2020 | DB<br>Lock | Updated label for "Centiloid "Amyloid PET Centiloid" | Updated label for "Centiloid" to "Amyloid PET Centiloid" | |
| | | | To include MMSE, CDR-SOB and Amyloid PET Centiloid in baseline comparability, the language for baseline comparability paragraph in section 2.3.3 made more generic and flexible | |
| 23-<br>Jul-<br>2020 | Post<br>DB<br>Lock | Creation of addendum 1 | Updated the derivation of Annualized percent change for Volumetric MRI reporting in section 2.5.2 | |
| | | | Updated label for "Centiloid" to "Amyloid PET Centiloid" | |
| | | | To include MMSE, CDR-SOB and Amyloid PET Centiloid in baseline comparability, the language for baseline comparability paragraph in section 2.3.3 made more generic and flexible | |
| | | | Added the need for analysis of Time to first change in diagnosis classification when participants are on treatment, Time to first decrease in RBANS Total Score of >= 14 points when participants are on treatment. | |

| Date | Time<br>point | Reason for update | Outcome for update | Section and title impacted (Current) |
|---|---|---|---|---|
| | | | Updated wording in definition of last on treatment for clarity in section 2.1.1. | |
| | | | Included effect size and CIs for APCC score in section 2.5.1, 2.5.2. | 2.5.1, 2.5.2, |
| | | | Censoring rule clarified for time to first decrease in RBANS >= 14 points in section 2.5.5. | 2.5.5 |
| | | | Minor edits in section 4 | |
| 03-<br>Aug-<br>2020 | Post<br>DB<br>Lock | Creation of addendum 1 | $A\beta 1-42/$ $A\beta 1-40$ ratio added to CSF biomarker reporting in section 2.7.1, 2.7.2. | 2.7.1, 2.7.2 |
| | | | Added a note "summaries of time (in days) of visits that are "last on treatment" and "last off treatment" will be presented in CSR Appendix 16.1.9" in section 2. Added section 5.4.2 for additional SAS outputs in Appendix 5 to be used for CSR Appendix 16.1.9 | |
| 24-<br>Nov-<br>2020 | Post<br>DB<br>Lock | Creation of addendum 2 | Plasma Aβ1-40 summary added to section 2.7.1 under Biomarkers in blood | |
| 27-<br>Nov-<br>2020 | Post<br>DB<br>Lock | Creation of addendum 2 | In section 2.5.1 added additional criteria for change in cognition; improvement (increase) from previous visit by at least 7 points, no change from baseline (change between -6 and 6), no change from previous visit (change between -6 and 6) | |

| Та | | content | 'S | 1 |
|---|---|---|---|---|
| | | | tions | |
| 1 | | | TOHS | |
| 1 | 1.1 | | sign | |
| | 1.1 | 1.1.1 | | |
| | | 1.1.1 | Study Design Summary | |
| | | 1.1.2 | Planned Number of Participants | 10 |
| | | 1.1.4 | Primary Analysis Time Point | |
| | | 1.1.4 | Interim Analyses | |
| | 1.2 | | jectives and endpoints | |
| | 1.2 | 1.2.1 | Primary objectives | |
| | | 1.2.1 | Secondary objectives | |
| | | 1.2.2 | Secondary objectives | 11 |
| 2 | Statia | tical matha | ods | 12 |
| 2 | 2.1 | | lysis general information. | |
| | 2.1 | 2.1.1 | General definitions | |
| | 2.2 | | sets | |
| | 2.2 | 2.2.1 | | |
| | 2.3 | | Group for specific analysis | |
| | 2.3 | 2.3.1 | isposition, demographics and other baseline characteristics Patient disposition | |
| | | 2.3.1 | | _ |
| | | 2.3.3 | Dealtoround and domographic characteristics | |
| | 2.4 | | Background and demographic characteristics | 21 |
| | 2.4 | | nts (study treatment, rescue medication, concomitant therapies, nce) | 22 |
| | | 2.4.1 | Study treatment / compliance | |
| | | 2.4.2 | Prior, concomitant and non-drug therapies | |
| | 2.5 | | of the primary objective | |
| | 2.0 | 2.5.1 | Worsening in cognition and reversibility | |
| | | 2.5.2 | Volumetric MRI | |
| | | 2.5.3 | Primary endpoint | |
| | | 2.5.4 | Statistical hypothesis, model, and method of analysis | |
| | | 2.5.5 | Handling of missing values/censoring/discontinuations | |
| | | 2.5.6 | Supportive analyses | |
| | 2.6 | | of the key secondary objective | |
| | 0 | 2.6.1 | Key secondary endpoint | |
| | | 2.6.2 | Statistical hypothesis, model, and method of analysis | |
| | | 2.6.3 | Handling of missing values/censoring/discontinuations | |

Page 5 CAPI015A2201J

| | 2.7 | Analysi | is of secondary efficacy objective(s) | 30 |
|---|---|---|---|---|
| | | 2.7.1 | Secondary endpoints | 30 |
| | | 2.7.2 | Statistical hypothesis, model, and method of analysis | 33 |
| | | 2.7.3 | Handling of missing values/censoring/discontinuations | 35 |
| | 2.8 | Safety a | analyses | 35 |
| | | 2.8.1 | Adverse events (AEs) | 35 |
| | | 2.8.2 | Deaths | 37 |
| | | 2.8.3 | Laboratory data | 37 |
| | | 2.8.4 | Other safety data | 38 |
| | | | | 40 |
| | | | | 40 |
| | 2.11 | Patient | reported outcomes | 41 |
| | 2.12 | Biomar | kers | 41 |
| | | | | 41 |
| | 2.14 | Interim | analysis | 41 |
| | | | | 41 |
| 4 | Chang | ge to prot | ocol specified analyses | 44 |
| 5 | Appe | ndix | | 44 |
| | 5.1 | Imputat | tion rules | 44 |
| | | 5.1.1 | Study drug | 44 |
| | | 5.1.2 | AE date imputation | 44 |
| | | 5.1.3 | Concomitant medication date imputation | 44 |
| | 5.2 | AEs co | ding/grading | 45 |
| | 5.3 | Laborat | tory parameters derivations | 45 |
| | 5.4 | Statistic | cal models | 47 |
| | | 5.4.1 | Primary analysis | 47 |
| | | 5.4.2 | Additional SAS outputs | 47 |
| | 5.5 | Rule of | exclusion criteria of analysis sets | 48 |
| | 5.6 | Notable | e and abnormality criteria | 49 |
| | 5.7 | Analysi | is windows rules | 51 |
| | 5.8 | RBANS | S Index tables | 60 |
| 6 | Refer | ences | | 98 |

## List of abbreviations

| LIST OF ADDI | eviations |
|--------------|--------------------------------------------------|
| Αβ | Amyloid-beta |
| AD | Alzheimer's Disease |
| AE | Adverse event |
| ALT | Alanine Aminotransferase |
| AmD | Amyloid Disclosure follow up set |
| ANOVA | Analysis of Variance |
| AOPE4 | Apolipoprotein Ε ε4 allele |
| APCC | API Preclinical Composite Cognitive Battery |
| API | Alzheimer's Prevention Initiative |
| APOE | Apolipoprotein E |
| APP | Amyloid Precursor Protein |
| ARIA | Amyloid Related Imaging Abnormalities |
| ARIA-E | Amyloid Related Imaging Abnormality-edema |
| ARIA-H | Amyloid Related Imaging Abnormality-hemorrhages |
| AST | Aspartate Aminotransferase |
| ATC | Anatomic Therapeutic Chemical classification |
| AUC | Area Under the Curve |
| BACE | Beta-site-APP Cleaving Enzyme |
| Bid | bis in diem/twice a day |
| BMI | Body Mass Index |
| BSI | boundary shift integral |
| CDR | Clinical Dementia Rating |
| CDR-SOB | Clinical Dementia Rating Sum of Boxes |
| CFR | US Code of Federal Regulations |
| ChEls | Cholinesterase-Inhibitors |
| CI | Confidence Interval |
| CM | Concomittant Medication |
| CNS | Central Nervous System |
| CRF | Case Report/Record Form (paper or (e)electronic) |
| CSF | Cerebrospinal fluid |
| CSR | Clinical Study report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| СТС | Common Toxicity Criteria |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DDI | Drug-Drug-Interaction |
| DMC | Data Monitoring Committee |
| DMAG | Disclosure Advisory Monitoring Group |
| DNA | Deoxyribonucleic Acid |
| DRM | Dose Regimen Modification |
| ECG | Electrocardiogram |
| ECog | Everyday Cognition scale |
| EDC | Electronic Data Capture |

| EoS | End of Study |
|---|---|
| FAS | Full Analysis Set |
| GCP | Good Clinical Practice |
| GD | Genetic Disclosure follow up set |
| Hb | Hemoglobin |
| HMs | Homozygotes |
| HTs | Heterozygotes |
| IA | Interim Analysis |
| IB | Investigator's Brochure |
| i.m | Intramuscular |
| i.v. | Intravenous |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use |
| IEC | Independent Ethics Committee |
| IgG | Immunoglobulin G |
| IGT-AD | Impact of Genetic Testing for Alzheimer's Disease |
| IRB | Institutional Review Board |
| i.m | Intramuscular |
| IRT | Interactive Response Technology |
| IVR | Interactive Voice Response |
| IWR | Interactive Web Response |
| LDH | Lactate Dehydrogenase |
| LDR | Lower Dose Regimen |
| LFT | Liver Function Test |
| LLOQ | Lower Limit of Quantification |
| LOAD | Late Onset Alzheimer's Disease |
| MAP | Master Analysis Plan |
| MAR | Missing at Random |
| MCI | Mild Cognitive Impairment |
| MedDRA | Medical Dictionary for Drug Regulatory Affairs |
| mSAF | Modified Safety Analysis Set |
| MMSE | Mini-Mental State Examination |
| MMRM | Mixed Model Repeated Measure |
| MRI | Magnetic Resonance Imaging |
| non-HMs | non-Homozygotes, i.e. Heterozygotes or non-carriers |
| NFL | Neurofilaments |
| NYHA | New York Heart Association |
| o.d. | Once Daily |

| 00/550 | |
|---------|--------------------------------------------------------------------|
| OC/RDC | Oracle Clinical/Remote Data Capture |
| OS | Overall Survival |
| p.o. | Oral (per os) |
| PAC | Progression Adjudication Committee |
| PDS | Programming Dataset Specifications |
| PET | Positron Emission Tomography |
| PK | Pharmacokinetics |
| PPS | Per-Protocol Set |
| PPW | Premature Participant Withdrawal |
| PRO | Participant Reported Outcomes |
| PT | Preferred Term |
| q.d. | Quoque die (once each day) |
| Qd | Qua'que di'e / once a day |
| QTcF | Fridericia QT correction formula |
| RAP | Report and Analysis Process |
| RAS | Randomized Analysis Set |
| RBANS | Repeatable Battery for the Assessment of Neuropsychological Status |
| REVEAL | Risk Evaluation & Education for Alzheimer's Disease |
| RNA | Ribonucleic Acid |
| ROI | Region of Interest |
| SAE | Serious Adverse Event |
| SAF | Safety Analysis Set |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analytics System(or Software) |
| SE | Standard Error |
| SMQ | Standardized MedDRA Query |
| SOC | System Organ Class |
| STAI-AD | State Trait Anxiety Inventory for AD |
| SUVR | Standardized Uptake Ratio |
| SD | Standard Deviation |
| TBL | Total Bilirubin |
| TE | Target Engagement |
| TEC | Treatment Epoch Completion |
| TLFs | Tables, Listings and Figures |
| TTE | Time-To-Event |
| ULN | Upper Limit Of Normality |
| WHO-DD | World Health Organization Drug Dictionary |
| γ-GT | Gamma-Glutamyl Transferase |

#### 1 Introduction

This Statistical Analysis Plan (SAP) describes main efficacy and safety analyses of clinical trial CAPI015A2201J for Cohort II. This SAP also describes analysis strategy for the impact of genetic disclosure in a dedicated Section 2.3.2. The study CAPI015A2201J has been terminated prematurely after a regular DMC review in July 2019. Hence, only abbreviated Clinical Study Report (CSR) will be created for this study.

The content of this SAP is based on the final amendment version 6.0 of protocol CAPI015A2201J.

#### 1.1 Study design

#### 1.1.1 Study Design Summary

This study protocol has multiple epochs with two informed consents required:

- 1. Pre-screening Epoch and Genetic Disclosure Follow-up (Informed consent #1)
- 2. Screening, Treatment and Follow-up Epochs (Informed consent #2).

The Pre-screening Epoch includes pre-screening assessments for evaluation of disclosure of APOE genotype to participants; the Genetic Disclosure Follow-up includes assessment telephone calls for all participants who received disclosure of their genotype.

Participants with APOE4 genotype (HMs) can enter the 12 week screening phase during which the pre-study assessments will be performed. The Treatment Epoch follows a randomized, double-blind, placebo-controlled, two-cohort parallel group design in which participants receive one of the investigational treatments or their matching placebo for a planned duration of at least 60 months.

The follow-up epoch is scheduled 26 weeks after last injection of CAD106 for Cohort I and 13 weeks after last dose of CNP520 for Cohort II.



#### 1.1.2 Planned Number of Participants

The trial will involve the assessment of efficacy for two investigational treatments in two separate cohorts, primary analysis will compare each active investigational treatment arm to its matching placebo. For Cohort I, sample sizes of 430 participants in the active treatment arm, CAD106, and 260 in the matching placebo arm are planned; for Cohort II, 390 in the active treatment arm CNP520 and 260 in the corresponding placebo arm are planned. In total, 1340 participants willbe randomized into the study (see Section 3 for the full details of the sample size calculation). This SAP focuses on Cohort II only (CNP520 or placebo).



#### 1.1.4 Primary Analysis Time Point

There are two primary endpoint variables: time to first diagnosis of MCI due to AD or dementia due to AD (TTE), and the APCC test score. TTE will be analyzed only after the target number of events (275 events in the active arm) has been observed. The APCC score is analysed after all participants have completed 60 months follow-up.

#### 1.1.5 Interim Analyses

The main purposes of the planned analyses during the course of the trial are safety monitoring by the DMC and assessment of futility with the potential consequence of discontinuing a futile active treatment arm and the corresponding placebo.

Interim Analyses are planned at various stages throughout the trial.

- 1. Safety monitoring
  - Regular semi-annual evaluation of safety parameters, worsening in cognition as a safety measure together with data allowing risk/benefit assessment to be defined with the DMC
  - Safety monitoring of T-cell activation data of n = 50 participants in Cohort I
- 2. Unblinded futility IA of Immunogenicity of CAD106
- 3. CNS activity based on biomarkers when a pre-defined number of participants reach 24 months.
  - Cerebrospinal fluid (CSF): Aβ (only for CNP520), tau pathology
  - PET imaging data: amyloid,
  - Volumetric MRI (only for CNP520)
- 4. Primary endpoints: Analyses of Primary efficacy parameters (TTE and APCC) when a sufficient number of events are observed to assess futility or stopping due to overwhelming efficacy.

### 1.2 Study objectives and endpoints

#### 1.2.1 Primary objectives

- To demonstrate the effects of CNP520 vs. respective placebo on Time-to-event (TTE), with event defined as a diagnosis of MCI due to AD or dementia due to AD, whichever occurs first during the course of the study,
- To demonstrate the effects of CNP520 vs. respective placebo on cognition as measured by the change from Baseline to Month 60 in the APCC test score.

#### 1.2.2 Secondary objectives

#### Key secondary objective

• To assess the effects of CNP520, vs. respective placebo on global clinical status as measured by the change from Baseline to Month 60 in Clinical Dementia Rating Scale Sum of Boxes (CDR-SOB) score.
# Secondary objectives

- To assess the safety and tolerability of CNP520, vs. respective placebo as measured by adverse events (AEs), and changes in the brain structural MRI, laboratory tests, non-cognitive neurological and psychiatric examinations including the self-reported Columbia Suicide Severity Rating Scale (eC-SSRS), vital signs and electrocardiogram (ECG).
- To assess the effects of CNP520, vs. respective placebo on cognition as measured by changes from Baseline to Month 60 on the Total Scale score and individual neurocognitive domain index scores of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).
- To assess the effects of CNP520, vs. respective placebo on function as measured by the change from Baseline to Month 60 in the Everyday Cognition scale (ECog) total scores reported by the participant and study partner, respectively.
- To assess the effects of CNP520, vs. respective placebo on AD-related biomarkers (amyloid deposition and measures of neurodegeneration) as measured by change from Baseline to Months 24 and 60 in the subset of participants who consent on:
  - amyloid tracer and tau tracer (at the subset of sites with access to tracer and the required imaging capability) obtained using brain positron emission tomography (PET) imaging
  - volumetric MRI measurements, and
  - CSF/blood A $\beta_{40}$ , A $\beta_{42}$ , total tau and phosphorylated tau<sub>181</sub> and NFL levels.
- To assess the effects of CNP520 vs. placebo on cerebral amyloid angiopathy (CAA) as measured by micro-hemorrhages and white matter hyper-intensities on MRI.





# 2 Statistical methods

Due to the early termination of the clinical trial, most of the primary, key secondary and the secondary objectives cannot be addressed with the data collected until termination. The originally planned inferential statistical analyses comparing efficacy readouts at Month 60 across treatment groups will not be conducted, but data collected on primary and secondary variables will be reported descriptively.

All the efficacy and biomarker endpoints except from events and TTE itself will be summarized using descriptive statistics by treatment groups as follows

- Raw values by visit including the "last on treatment", "last off treatment", TEC and the EoS follow-up visit
- Change from baseline by visit including "last on treatment", "last off treatment", TEC and EoS
- Change from "last on treatment" visit to TEC, change from "last on treatment" to "last off treatment", change from "last on treatment" visit to EoS and change from TEC to EoS

Note: Time of "last on treatment" and "last off treatment" will be discussed in CSR statistical Appendix 16.1.9, specifications will be described in the TFL shells document in Section 16.1.9.

All the safety data will be summarized using descriptive statistics by treatment groups.

Analysis of genetic disclosure follow-up will be summarized using descriptive statistics by genotype groups as described in Section 2.3.2.

# 2.1 Data analysis general information

The statistical analysis will be performed by Novartis internal statisticians and programmers.

Unless otherwise stated, summary tables/listings/figures will be presented by treatment group in the respective analysis set. Tables showing only baseline data will also include a total column.

Categorical data will be summarized as frequencies and percentages. Percentages will be calculated as below:

- For population level summaries (like Demographic, AEs, Medical history...etc.), percentages will be calculated using number of participants in each reporting group as the denominator
- For by visit summaries, percentages will be calculated using the number of participants in the analysis set with an assessment at the specified visit as the denominator.

• For specific event based summaries, the denominator will only include the subset of the analysis population of participants at risk at a specific point in time (Kaplan-Meier approach).

Continuous data will be summarized by presenting the number of non-missing observations, mean, standard deviation (SD), median, minimum and maximum, both for raw (absolute) values and for changes from baseline. Summary tables will be presented wherever applicable by visit if not otherwise specified.

Specified parameters of interest will be listed by treatment group, records will be ordered by country/center/participant and time of assessment.

General information on treatment group labels, decimal places and other output related information will be specified in the specification document for tables, figures and listing (TFLs) shells accompanying this analysis plan.

Statistical analysis will be performed using SAS® statistical software (SAS Institute, Cary, NC, USA.) version 9.4 or higher.

#### 2.1.1 General definitions

# **Study Drug**

Study drug refers to CNP520 50 mg, or placebo.

# **Date of First Study Drug Administration (Day 1)**

Day 1 is defined as the first day of randomized study drug administration. All other days will be labelled relative to Day 1. For event dates on or after Day 1, study day for an event date is calculated as (event date – first dose date + 1) which could be Day 2, Day 3 etc. For event dates before Day 1, study day for an event date is calculated as (event date – first dose date), which could be Day -1, Day -2, etc., referring to one day, two days, etc., before Day 1, respectively. Thus, Day -1 is the day preceding Day 1. Day 0 is not defined.

# **Date of Last Study Drug Administration**

The date of last study drug administration is the day of intake of the last dose of study drug.

#### **Baseline**

A baseline value refers to the last (most recent) evaluable measurement prior to Day 1. Typically, baseline values will be the values obtained on the day of randomization. If the Baseline visit is missing or the assessment was not done at Baseline, the last assessment of an earlier visit (scheduled or unscheduled) which is closest to the Baseline visit will be used as Baseline value. In case an assessment is repeated at a later visit during the screening epoch, the latest one will be used as Baseline value.

Note: Assessments at the day of randomization are assumed to have been taken as per protocol, i.e. if the assessment should be performed before dosing, the assessment will be treated as predose as per protocol. Practically, i.e. that the time part of the date/time entry (when collected) will be ignored. Exception: In case there is a protocol deviation or a comment that specifically

indicates that the assessment has been taken post-dose, the assessment will not be handled as pre-dose.

#### Post-baseline

For safety and efficacy evaluations all assessments after Day 1 are defined as post-baseline assessments.

# **Roll-over participants**

Participants from CNP520A2202J study (Generation study 2; GS2) may roll over to be enrolled into API015A2201J study (Generation study 1; GS1). These participants have been genotyped and disclosed in GS2.

Roll-over participants in GS1 have signed the GS1 Informed Consent Form (ICF#1 and ICF#2), and GS1 inclusion/exclusion criteria were verified. The participant received a new subject identifier in GS1. Some of the screening assessments for these participants will be repeated in GS1, and for some assessments, data obtained in GS2 will be re-entered.

Note: For roll-over participants, data collected in GS2 and skipped in GS1 are expected to be mapped (re-entered) from the GS2 to the GS1 database. Hence, there is no programming effort expected to map the data from GS2 to GS1.

# Re-screened participants

Participants who screen-failed due to a temporary condition (e.g. physical, concomitant medications, etc.) or due to administrative reasons may be re-screened after resolution. The participant will receive a new subject identifier at re-screening. The latest screening assessment will be considered for reporting at screening visit. Assessments (like genotype, volumetric MRI, etc.) that are not repeated, will be carried over. This is based on mapping the old subject identifier to the new subject identifier.

In general, all data collected under the old subject identifier is kept after mapping to the new subject identifier. This comprises for instance AEs, vital signs, ECG, and laboratory data. In case of missing values under the new subject identifier, the latest available value from the old subject identifier will be used. In study GS1, the earliest consent date is kept, if the subject is re-screened

#### **Prior and Concomitant Medication**

Prior medication will be defined as any medication taken prior to the first dose of the study drug, irrespective of whether the medication continued into the treatment period.

Any medication administered at least once between Day 1 and end of the study is defined as concomitant medication.

#### **Visit Windows**

In general, by-visit analyses will include data from scheduled as well as un-scheduled visits using visit windows for scheduled visits except for TEC/PPW and EoS. In general, the lower and upper bound of a visit window will be defined as the midpoint between scheduled visits. The visit window rules for efficacy and safety parameters are defined in Appendix 5.7.

For efficacy parameters: In case of competing assessments within a visit window, the assessment value closest to the scheduled visit day will be used. In case of equal distances, the earliest assessment value will be used. Visit window will not be applicable for TEC and EoS.

For safety parameters: In case of competing assessments within a visit window, the worst assessment value within the visit window will be used. This rule also applies for worsening in cognition as a safety measure.

Listings will include all assessments, sorted by date of assessment, flagging unscheduled visits. The listings will include analysis windows and corresponding flags to indicate the assessment's inclusion in the analysis.

# Treatment Epoch Completion (TEC) and End of Study (EoS) and other points in time of interest

TEC is the end of treatment phase visit (i.e., visit 399) that will be completed for all participants after discontinuation of treatment. The same visit will also be completed in case of PPW. PPW is the premature study withdrawal.

EoS is a Follow-up visit scheduled after TEC/PPW, per urgent safety measure (USM) on 11-Jul-2019, and its follow-up letter dated 12-Dec-2019, Modified EoS visits can be scheduled anytime after receipt of this notification but no later than 15-Mar-2020. (i.e. the requirement from 11 July 2019 USM for the 6 month timeframe between modified TEC and mEoS visits is no longer required.)

Participants who were attending study visits (i.e., continuing in the study) but already off-treatment at time of USM were to come for EoS straight (no TEC required).

An assessment will be on treatment if it is before or at last day on study drug + 31 days. The last assessment before or at last day on study drug + 31 days will be referred to as "last on treatment" assessment. The last assessment after last day on study drug + 31 days will be referred to as "last off treatment" assessment. For deriving "last on treatment" or "last off treatment", last assessment date of RBANS will be used. That means, to derive the last on treatment and last off treatment for all the parameters, regardless of their actual assessment dates, RBANS last assessment date will be used as reference date. Note: the "last on treatment" and "last off treatment" flag will be created for each participant at visit level (not at the individual assessment level). If there is missing RBANS assessment at the specific visit, then date of the first day corresponding to that visit (i.e. non-missing assessment of that parameter under consideration) will be used to derive the "last on/off treatment" assessment.

Note: On treatment is a period from first dose to last dose + 31 days

#### For example:

- 1. If a participant has the last dose on 13-Jul-2019, then "on treatment" period would span from first dose to 13-Jul-2019 + 31 days.
- 2. If a participant has the last dose on 09-Apr-2019, then "on treatment" period would span from first dose to 09-Apr-2019 + 31 days.

# 2.2 Analysis sets

The following analysis sets will be used.

The **Randomized analysis set (RAS)** will consist of all participants who received a randomization number, regardless of receiving study medication.

The Safety analysis set (SAF) will consist of all participants who have received study medication.

Note: The above SAF definition is different from the protocol defined SAF definition which restricts to include only those participants in SAF if they have had at least one safety assessment after first dose administration.

The **modified SAF (mSAF)** will consist of all participants of the SAF with at least 3 months exposure duration.

All efficacy analyses (except worsening in cognition and reversibility) and safety analyses will be conducted on the SAF.

In addition, the following sets of participants will be used to understand the composition of analysis sets and disposition of participants.

**Pre-screened set** will consist of all participants completing the Prescreen GD Day 1 visit.

**Screened set** will consist of all participants (HMs only) who sign ICF#2 and proceed into Screening epoch.

# 2.2.1 Group for specific analysis

Analysis of worsening in cognition and assessing reversibility of worsening in cognition will be performed on the mSAF.

# 2.3 Patient disposition, demographics and other baseline characteristics

Summary tables for demographic variables and other baseline characteristics as well as relevant medical history will include a total column in addition to the treatment arms.

The impact of genetic and amyloid disclosure for the participants assessed for genetic disclosure and amyloid disclosure during the screening period will also be reported by genotype groups.

#### 2.3.1 Patient disposition

The number and percentage of participants in each analysis set described above will be presented including all participants that started screening. Primary reason for screen failure will be summarized for all participants.

Participant disposition will be summarized for the RAS showing the flow of participants through the treatment epoch and completing the End of Study disposition page. The disposition summary will show the number and proportion of participants who discontinued treatment epoch and End of Study status along with the reason for discontinuation. The number and proportion of participants with missing End of Study assessment will also be reported. The primary reasons for premature discontinuation of study treatment will also be summarized. Listings will be provided showing the primary reason for premature discontinuation of study and of study treatment.

All the important protocol deviations (PDs) reported during the study will be summarized in the following five categories:

- Selection criteria not met
- Participant not withdrawn as per protocol
- Treatment deviation
- Prohibited concomitant medication
- Other deviations (important deviations that do not fall in the above four categories)

Important PDs are defined as subset of PDs that may significantly impact a subject's rights, safety, and well being or the completeness, accuracy, and/or reliability of the study data. The PD codes to identify the above categories are listed in Table 5-4 in the Appendix.









# 2.3.3 Background and demographic characteristics

The following demographic and baseline variables will be summarized on the SAF. No listings will be provided.

# Demographic variables:

# Continuous variables:

- Age (years)
- Height (cm)
- Weight (kg)
- BMI (kg/m²) will be calculate as (body weight in kilograms) / (height in meters)²
- Volumetric MRI-Whole Brain (cm<sup>3</sup>)
- Volumetric MRI-Hippocampus (cm<sup>3</sup>)
- Amyloid PET Centiloid

# Categorical variables:

- Age group (≤64, 65-69, >70)
- Sex (Male, Female)

- Years of education: <=12 years, 13-16 years, >= 17 years
- BMI (< 25 vs >= 25)
- Race (Caucasian, Black, Asian, Native American, Pacific Islander, Other, Unknown)
- Ethnicity (Hispanic or Latino, Other East Asian, Southeast Asian, South Asian, West Asian, Russian, Japanese, Chinese, Mixed Ethnicity, Other Unknown, Not reported)

# Cognitive scales at baseline

#### Continuous variables:

- MMSE
- RBANS Total score
- Immediate Memory Index
- Delayed Memory Index
- Visiospatial/ Semantic Index
- Language Index
- Attention Index
- CDR-SOB

# Categorical variables:

• CDR Global (Score = 0, Score = 0.5, Score > 0.5)

Comparability of randomized groups (active versus placebo) at baseline will be assessed via Fisher's exact tests for 2x2 tables or the corresponding Freeman-Halton test for general lxk tables  $(l,k \ge 2)$  for the selected categorical variables. If Fisher's exact tests are not estimable (e.g. sample size is too large to calculate the statistic) or not adequate, then Chi-squared tests will be performed. Baseline comparability for selected continuous variables will be assessed using t-tests assuming unequal variances in the two groups (active versus placebo). The tests performed together with the p-value will be reported for each baseline variable that has been investigated for comparability. The selected variables for comparisons will be indicated in the TFL shells.

# **Medical history**

Any condition entered as medical history or current medical conditions at baseline will be coded using the MedDRA dictionary effective at the time of the database lock and summarized by system organ class (SOC) and preferred term (PT) on the SAF. No listing will be provided.

# 2.4 Treatments (study treatment, rescue medication, concomitant therapies, compliance)

# 2.4.1 Study treatment / compliance

The duration of exposure to study drug is defined as the time (in days) from the first study drug administration to last study drug administration + 31 days.

The duration of exposure will be calculated as

(last dose date + 31 days) - first dose date + 1.

Duration of exposure to CNP520 will be summarized as continuous variable (in days) and categorical variable, using categories >=1 day (any exposure), >=3 months, >= 6 months, >=1 year, >=1.5 years.

For each treatment group, the participant-years will be calculated as

(sum of the durations of exposure for all participants in the group)/365.25) and will be summarized.

# 2.4.2 Prior, concomitant and non-drug therapies

The number and percentage of participants receiving concomitant medications will be summarized on the SAF by ATC class and preferred term (according to the latest World Health Organization drug dictionary (WHO-DD) at the time of database lock, including Anatomical Therapeutic Chemical (ATC) classification code).

The number and percentage of participants receiving significant non-drug therapies will be summarized on the SAF by primary system organ class, preferred term (according to the latest MedDRA dictionary version available at the time of database lock).

# 2.5 Analysis of the primary objective

Worsening in cognition triggered early termination of the trial and plan is to describe this as rationale for early termination of the trial in CSR before describing the analysis on primary endpoint, hence the below section describes the worsening in cognition and reversibility before the primary endpoint.

#### 2.5.1 Worsening in cognition and reversibility

Worsening in cognition will be assessed based on RBANS, CDR-SOB and APCC for participants in the mSAF.

#### **Tables**

The number of participants and the frequency of change (and worsening) in cognition of a specific magnitude (absolute change above specific threshold) will be summarized by visit, including TEC, and EoS as well as last assessment on treatment and last assessment off treatment:

- RBANS decrease (total score and Index scores): ≥ 7 points, and ≥ 14 points from baseline, and from previous visit
- RBANS improvement or increase (total score and Index scores): ≥ 7 points from baseline, and from previous visit
- RBANS no change (change between -6 and 6) from baseline, and from previous visit
- CDR-SOB increase: ≥ 0.5 points, ≥ 1.0 point, and ≥ 1.5 points from baseline, and from previous visit
- CDR-SOB improvement (any decrease) from baseline, and from previous visit
- CDR-SOB no change from baseline, and from previous visit

In addition to the "by visit" tabulation, the proportion of participants with a clinically relevant worsening from baseline/previous visit will also be shown for

- Either at Week 13 or Week 26 (not at both) the denominator will be based on participants who have an assessment at both visits;
- Both, at Week 13 and Week 26 the denominator will be based on participants who have an assessment at both visits;
- At any visit out of Week 13 and Week 26 the denominator will be based on participants who have an assessment at at least one of the two visits;
- At Any visit up to and including "last on treatment"—the denominator will be based on participants who have an assessment at any post baseline visit (up to and including "last on treatment" assessment).

For the RBANS total score, RBANS index scores and APCC score, effect sizes of change from baseline as well as 80% confidence intervals (CIs) for the effect size will be reported. The effect size (and CI) of change from baseline will be calculated for following post-baseline visits: Week 13 and Week 26, Week 52, TEC, EoS, last assessment on treatment, and last assessment off treatment. The effect size will follow the *Cohen's d* formula: The raw mean to standard deviation ratio, not model based mean to standard deviation ratio. The effect size will be calculated as the difference between active and placebo in mean change from baseline divided by the pooled standard deviation of the change. Effect sizes and CIs will be calculated (active versus placebo).

# Derivation of study specific effect size d and corresponding CI

BL = Baseline value; PBL= Post baseline value;

SD = Standard deviation; SE = Standard error;  $n_1$  = Sample size group 1;  $n_2$  sample size group 2;  $S_1^2$  = Variance group 1;  $S_2^2$  = Variance group 2

Numerator: Mean change from BL to PBL active – mean change from BL to PBL control

Denominator: pooled SD defined as

$$SD_{pooled} = \sqrt{\frac{(n_1 - 1)S_1^2 + (n_2 - 1)S_2^2}{n_1 + n_2 - 2}}$$

Where the groups are given by factor treatment (active versus control).

The confidence interval can be derived using the formula proposed by Hunter and Schmidt 2004 and Nakagawa and Cuthill (2007):

$$CI: d \pm z * SE(d)$$

Where z is the 10% Quantile of the normal distribution in case of the 80% CI. The SE(d) is calculated as

$$SE_d = \sqrt{\frac{(n_1 + n_2 - 1)}{(n_1 + n_2 - 3)} \left[ \left( \frac{4}{n_1 + n_2} \right) \left( 1 + \frac{d^2}{8} \right) \right]}$$

For CDR-SOB, corresponding confidence intervals for the difference between treatment groups will be provided.

Correlation between changes in RBANS total, APCC score and whole brain, hippocampal volume will be reported (correlation coefficient and R square will be reported by treatment group and visit (including also the last assessment on treatment, last assessment off treatment).

# **Figures**

Graphical presentation (forest plots) of the effect sizes and corresponding confidence intervals for RBANS total, RBANS index scores and APCC score by visit including TEC and EoS, as well as last assessment on treatment and last assessment off treatment.

#### 2.5.2 Volumetric MRI

Screening (baseline) volumetric measurements are performed using FreeSurfer software. This leads to reference volumes for whole brain, ventricles, hippocampus, and intra-cranial.

Volumetric data will be available for the following regions:

- intra-cranial volume (ICV),
- total/whole brain,
- left/right hippocampus,
- lateral ventricles.

In order to assess atrophy rate, volumetric MRI images from follow-up timepoints are compared to those from screening, using the boundary shift integral (BSI) technique in selected brain regions. The technique determines the total volume through which the boundaries of a given cerebral structure have moved, and hence, it aims at quantifying the amount of change in these selected brain regions. The output of the method is a change from baseline in volume (atrophy).

Volume changes in the following regions of interest (ROI) will be reported:

- whole brain,
- hippocampus (sum of left and right),
- lateral ventricles (left and right).

#### **Tables**

Summary statistics for absolute change and percent change from Baseline to timepoint will be provided. All statistics will be based on the total volume, i.e. the sum of the respective left and right volumes as applicable. In addition, the annualized percentage change will be calculated as the mean of individual participant annualized percentage change (percentage change per participant / time interval (in days) between current MRI assessment and date of baseline MRI assessment per participant) x 365.25. Time interval (in days) will be derived as date of current MRI assessment – date of baseline MRI assessment + 1.

Raw volumes, as well as changes, % changes, and annualized % changes from baseline will be summarized by visit including TEC, EoS, and last assessment on treatment, last assessment off treatment.

For investigation of worsening (increased atrophy) under treatment and reversibility, these summary statistics will also be provided for the mSAF by visit including TEC, EoS, and last assessment on treatment, last assessment off treatment.

The relationship between percentage change from baseline in hippocampal and whole brain volumes and change in RBANS total score and APCC score will be examined through correlation analysis. This will be done for participants with at least 3 months exposure (mSAF). The Spearman and Pearson correlation coefficients and associated p-values will be reported.

# 2.5.3 Primary endpoint

There are two primary endpoint variables:

Time-to-event (TTE), with event defined as time to first confirmed diagnosis of MCI due to AD or dementia due to AD (whichever occurs first), and

Change in the API preclinical cognitive composite (APCC), from baseline to Week 260<sub>(M 60)</sub>

# Time to event (MCI due to AD or dementia due to AD)

Time-to-event (TTE), with event defined as the first confirmed diagnosis of MCI due to AD or dementia due to AD (whichever occurs first). An event is identified as a Progression Adjudication Committee (PAC)-confirmed diagnosis triggered either by an investigator diagnosis or an increase in the CDR global score. The confirmation by the PAC consists of two confirmed adjudications based on data from two consecutive visits.

In case of an identified event, TTE will be calculated as the time from randomization to the first confirmed diagnosis. For each event (confirmed diagnosis), the date of the initial investigator diagnosis will be used to establish the date of the event (neither the date of adjudication, nor the date of the confirmation). In case no confirmed event has been observed for an individual, the observation will be censored, and the censoring date will be defined as the last date where the diagnosis classification has been assessed. Time to censoring date will be calculated from day of randomization.

The team agreed that the date of 25 August 2019 was the cut-off date/point for the final analysis. The final TTE analysis will include data until this cut-off point. Any data collected after this cut-off point will not be used for the primary analysis of TTE. That means specifically that only confirmed events collected up to the data cut-off point will be counted. Confirmation information collected after the cut-off point to confirm an earlier (meaning before the cut-off point) adjudicated diagnosis of MCI or AD due to dementia will not be taken into consideration. As a consequence, the observation will be censored at the last date prior to cut-off point that the TTE endpoint was evaluated, and the unconfirmed diagnosis will not be counted as an event in the primary analysis.

Due to the early termination of the studies, only a small number of events following the above definition have been observed. Hence, for the abbreviated CSR, the number (%) of participants meeting the following additional situations (change in diagnosis classification) will also be reported:

- 1. Participants with a change in diagnosis classification from cognitively unimpaired by the principal investigator at any time
  - MCI due to AD,
  - MCI not due to AD,
  - Dementia due to AD,
  - Dementia not due to AD.

- 2. Participants with an increase in CDR global score from baseline at any time (any increase, increase less than 1, increase of 1 or more);
- 3. Participants where data was sent for adjudication to PAC (regardless of confirmation at the following visit) split by the result of the adjudication:
  - Cognitively unimpaired,
  - MCI due to AD,
  - MCI not due to AD,
  - Dementia due to AD,
  - Dementia not due to AD,
  - Other (Unable to adjudicate, data not collected, not known).

Note that cut-off date/point (25 August 2019) used for protocol defined event (MCI due to AD or dementia due to AD) will not be applicable for the above defined additional situations. Data up to the database lock date will be used for the analysis of these additional situations.

# **APCC** score

The APCC test score is defined as a weighted sum of the following test items:

Raven's Progressive Matrices – subset items A2, A4, A8 & B1-B6 (0-9)

#### MMSE:

- Orientation to Time (0-5)
- Orientation to Place (0-5)

RBANS (Subtest raw scores):

- List Recall (0-10)
- Story Recall (0-12)
- Coding (0-89)
- Line Orientation (0-20)

The range of the APCC test score is from 0 to 100 where higher scores in the APCC correspond to a better cognitive performance. The APCC will be derived based on the test items using the below formula and weights:

APCC test score = 1.360×RBANS List Recall + 1.100×RBANS Story Recall +1.390×Raven's Progressive Matrices (subset items A2, A4, A8, B1-B6) + 0.321×RBANS Coding + 0.510×RBANS Line Orientation + 2.140×MMSE Orientation to Place + 2.240×MMSE Orientation to Time.

# 2.5.4 Statistical hypothesis, model, and method of analysis

Except from the primary objective on the TTE endpoint, the other primary objective (for APCC) aimed to evaluate effects of CNP520 versus Placebo by comparing changes from baseline to Month 60. Due to the early termination of CNP520, no data have been collected at Month 60. Only very few participants have provided data on active treatment with CNP520 beyond one year of follow-up. Hence, the originally planned inferential and model based statistical analyses cannot be performed and are no longer applicable.

# Time to event (MCI due to AD or dementia due to AD) ), Time to first change in diagnosis classification and Time to first decrease in RBANS Total of $\geq$ 14 points

#### **Tables**

Time to Event analysis using Kaplan Meier approach will be presented for time to MCI due to AD or Dementia due to AD (events as per protocol) and for time to first change in diagnosis classification (this is an event regardless of confirmation and adjudication) from cognitively unimpaired by the investigator. Analysis of time to first change in diagnosis classification will also be performed for participants on treatment. In addition, analysis of time to first decrease in RBANS Total Score of >= 14 points will be performed for participants on treatment (for on treatment definition, refer Section 2.1.1). The Kaplan-Meier estimates of the cumulative event rate for each treatment group will be summarized and plotted. To calculate the proportion of participants with events, number of participants at risk will be used as the denominator. "Participant at risk" at a specific time point is defined as the number of participants in the study without an event at up to that time point.

These analyses will only be performed if there are at least five such events.

In addition, the number and percentage of the additional situations (Section 2.5.3) defined events overall (not by visit) will be summarized by treatment group.

#### **APCC** score

#### **Tables**

The APCC test score and the seven components (listed above in Section 2.5.3) will be summarized on the SAF.

#### 2.5.5 Handling of missing values/censoring/discontinuations

# Time to event (MCI due to AD or dementia due to AD), Time to first change in diagnosis classification and Time to first decrease in RBANS total >= 14 points

In general, an observation will be censored if no event has been observed at the TTE analysis cut-off date. The censoring date will be defined as the last date (before cut-off date) where the TTE endpoint has been assessed.

The censoring date for each participant that did not have an event (i.e., a confirmed diagnosis) is defined as follows:

- 1. For participants ongoing in the study without a confirmed diagnosis at the time of the cutoff: the last day of a diagnosis assessment (the previous visit where a diagnosis assessment occurred prior to the cut-off date).
- 2. For participants who permanently discontinued from the study prior to the cut-off: The last day of a diagnosis assessment prior to study discontinuation.
- 3. For participants who had their last diagnosis assessment prior to randomization(i.e. during screening epoch) or do not have any diagnosis assessment post randomization, their randomization date will be used as censoring date.

4. For analysis of time to first decrease in RBANS >= 14 points, the last RBANS assessment date will be used as censoring date instead of last diagnosis assessment date mentioned in above three points.

Note: For Time to MCI due to AD or dementia due to AD, the cut-off date will be 25 August 2019. For Time to First change in diagnosis classification, the cut-off date will be database lock date, additional analysis of time to first change in diagnosis classification will be performed for participants on treatment. Also time to first decrease in RBANS >= 14 points will be performed for participants on treatment.

Further details on derivation of events and censoring will be added to the programming document specifications (PDS).

# Other primary efficacy endpoint variable (APCC)

Due to the early termination of the trial, analyses of primary efficacy variable APCC will in general be based on observed cases only, i.e. there will be no imputation of missing data. Exception in primary efficacy variable APCC applies to missing data in subtests of Raven's matrices included in the primary efficacy variable APCC. Missing values for the subtests of Raven's matrices of the APCC may be imputed using the imputation rule defined in Appendix 5.1.3.3.1.

# 2.5.6 Supportive analyses

Not Applicable.

# 2.6 Analysis of the key secondary objective

#### 2.6.1 Key secondary endpoint

The key secondary endpoint variable is CDR-SOB.

#### Clinical Dementia Rating (CDR) global and Sum of Boxes (CDR-SOB)

The CDR is obtained through semi-structured interviews of participants and informants, and cognitive functioning is rated in six domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a 5-point scale of functioning as follows: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment (personal care is scored on a 4-point scale without a 0.5 rating available). The CDR global score ranges from zero to three, with greater scores indicating greater disease severity. The CDR-SOB is defined as the sum of the ratings from the six domains, ranging from 0 to 18 with a minimum increment of 0.5. A higher CDR-SOB score indicates greater disease severity.

#### 2.6.2 Statistical hypothesis, model, and method of analysis

The key secondary objective aimed to evaluate effects of CNP520 versus Placebo by comparing changes from baseline to Month 60. Due to the early termination of CNP520, no data have been collected at Month 60. Only very few participants have provided data on active treatment with CNP520 beyond one year of follow-up. Hence, the originally planned inferential and model based statistical analyses cannot be performed and are no longer applicable.

#### **Tables**

CDR-SOB and CDR global will be summarized on the SAF.

# 2.6.3 Handling of missing values/censoring/discontinuations

Due to early termination of the trial, analyses of CDR-SOB will be based on observed cases only, i.e. there will be no imputation of missing data.

# 2.7 Analysis of secondary efficacy objective(s)

# 2.7.1 Secondary endpoints

#### **RBANS Total score and Index scores**

The RBANS is comprised of the following five neurocognitive domains, with associated subtests used for Index scores:

- Immediate Memory List Learning and Story Memory (IMI)
- Visuospatial/Constructional Figure Copy and Line Orientation
- Language Picture Naming and Semantic Fluency
- Attention Digit Span and Coding
- Delayed Memory List Recognition and Sum of (List Recall, , Story Recall, and Figure Recall; DMI)

The RBANS generates age-adjusted index scores for five neurocognitive domains, which are used to calculate a Total Scale Index score using norm tables for each Index scores in Appendix 5.8. The algorithm (by vendor) to derive index scores is based on the current actual age of the participant at that visit. For longitudinal analyses this approach creates artificial variability. As a consequence, the derived data for index scores will not be used in the analyses, but will be derived from source data using the age at baseline for adjustment for all assessments. The algorithm to derive the Index scores using age at baseline will be described in the programming specifications (PDS) of this study.

A higher RBANS score indicates better cognitive function.

# Mini Mental State Examination (MMSE)

The MMSE is a brief, practical clinician reported outcome that examines cognitive status (Folstein et al., 1975). It evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, and the ability to create a sentence and copy two intersecting pentagons. The test consists of five domains (orientation, registration, attention, recall, and language) with a total score ranging from zero to 30. A higher score indicates better cognitive function. The five sub scores as well as the total score will be recorded.

#### **Raven's Progressive Matrices**

Raven's Progressive Matrices (Raven et al 2000) is a non-verbal, multiple choice measure of general ability and reasoning using a visual modality. It was designed to be culturally nonbiased, as neither language nor academic skills are required to answer items successfully.

Although all components of the Raven's Progressive Matrices Set A and Set B will be assessed, in order to calculate the APCC test score, only a subset of items from Sets A and B will be used (items A2, A4, A8, B1-B6), with a range from zero to nine.

# **Everyday Cognition scale (ECog-Subject and ECog-Informant)**

The ECog scale measures cognitively-relevant everyday abilities and is comprised of 39 items covering six cognitively-relevant domains: Everyday Memory, Everyday Language, Everyday Visuospatial Abilities, Everyday Planning, Everyday Organization, and Everyday Divided Attention (Farias et al 2008). Within each domain, the ability to perform a specific task is rated on a five-point scale ranging from: 1) no difficulty, 2) mild difficulty, 3) moderate difficulty, 4) severe difficulty, or 5) unable to do. The scale has 2 versions one for patient (PRO) and one for informant (study partner).

The total score for the 39 items ranges from 39 to 195, with greater scores indicating worse daily function.



#### Biomarkers in Cerebrospinal Fluid (CSF)

The following AD related markers in CSF are analyzed:

- total-tau and phospho-tau (p-tau)
- $A\beta_{1-40}$ ,  $A\beta_{1-42}$  and  $A\beta_{1-42}/A\beta_{1-40}$

#### Biomarkers in blood:

# **Serum Light Chain Neurofilaments (NFL)**

Available measurements for NFL from serum will be summarized.

Values below the lower limit of quantification (LLOQ) will be set to LLOQ/2 for statistical analysis, values above upper limit of quantification (ULOQ) will be imputed with ULOQ. LLOQ and ULOQ value may differ across samples according to the dilution factor applied in the specific sample. For statistical analysis, the sample specific LLOQ and ULOQ value should be used.

# Plasma Amyloid Beta-40 (Aβ<sub>1-40</sub>)

The change from baseline of the plasma A $\beta$ 1-40 concentration levels will be summarized. Values below the lower limit of quantification (LLOQ) will be set to LLOQ/2 for statistical analysis, values above upper limit of quantification (ULOQ) will be imputed with ULOQ. LLOQ and ULOQ value may differ across samples according to the dilution factor applied in the specific sample. For statistical analysis, the sample specific LLOQ and ULOQ value should be used.

# Positron Emission Tomography (PET) Standard Uptake Value Ratio (SUVR)

Across the three F<sup>18</sup> amyloid binding radiotracers used Florbetapir (FBP), Florbetaben (FBB) and Flutemetamol (Flute): Centiloids using the agreed formulae

For participants who consent to the voluntary AD-related imaging biomarker evaluations, regional activity concentration and the cortical Standardized Uptake Value (SUV) are measured based on the following brain regions of interest (ROIs):

- Parietal cortex
- Posterior cingulate or Precuneus
- Medial orbitofrontal cortex
- Anterior cingulate
- Temporal cortex

and the whole cerebellum as reference region.

Data for regional activity concentration will not be reported.

The *global* cortical amyloid load will be derived as the unweighted average cortical Standardized Uptake Value Ratio (SUVR) between the cortical ROIs and the reference region.

# Standardization of Amyloid PET SUVR values

For Amyloid PET, the baseline load obtained from different tracers (florbetapir (FBP), flutemetamol (Flute) and florbetaben (FBB)) will be converted to a standardized Centiloid scale. The conversion equation for each tracer has been obtained following a non standard analysis method (AVID method) based on level-1 (GAAIN, Klunk et al. Centiloid values) and level-2 (InVicro Centiloid values) as documented in the Image Analysis charter from InVicro:

$$CL = 183.00 * SUVr_{FBP} - 176.97$$
  
 $CL = 123.90 * SUVr_{Flute} - 114.86$   
 $CL = 156.06 * SUVr_{FBB} - 148.132$ 

The reference is Klunk et al., 2015. The % change in SUVR will be calculated as

$$\%SUVR = \frac{(SUVR_{FU} - SUVR_{BL})}{SUVR_{BL}}$$

with SUVR<sub>BL</sub> as the baseline value and SUVR<sub>FU</sub> the SUVR value at follow-up visit.

# Analysis of positive/negative amyloid levels

Amyloid level (positive/negative) is measured at baseline by two methods:

- CSF collection via Lumbar puncture
- Brain Amyloid PET radiotracers (amyloid PET: SUVr)

The studies allow either method for determination of amyloid level. CSF samples are collected and analyzed using selected validated assay. The cut-off value to determine the amyloid level as positive/negative will depend on the assay selected. The criteria for positive amyloid level in CSF is based on pTau/Ab42 ratio. The criteria for positive amyloid PET will follow specifications for the specific radiotracer used. Following Table 2-3 describes the cutoffs for both methods.

Table 2-3 Amyloid Level Stratification Criteria

| Methods | | Positive | Negative |
|---|---|---|---|
| CSF | | <ul> <li>Elecsys ratio p-Tau/ Aβ1-42&gt; 0.024 </li> <li>AND</li> <li>Elecsys Aβ1-42≤ 1700.0 pg/ml (upper limit of the measuring range)</li> </ul> | <ul> <li>Elecsys ratio p-Tau/ Aβ1-42≤ 0.024 </li> <li>Elecsys Aβ1-42&gt; 1700.0 pg/ml (upper limit of the measuring range)</li> </ul> |
| PET | Florbetapir (FBP) | SUVr_FBP ≥ 1.1 | SUVr_FBP < 1.1 |
| | Flutemetamol (Flute) | SUVr_ Flute ≥ 1.123 | SUVr_ Flute < 1.123 |
| | Florbetaben (FBB) | SUVr_FBB ≥ 1.105 | SUVr_FBB <1.105 |

Analysis of Amyloid levels will be derived as Positive/Negative as described in Table 2-3 above. However, in the database, eligibility result for Amyloid status will be Elevated/Not-Elevated as derived by vendor result (including a visual examination of the scan) or by the combination of the two results if at least one has a positive result then it will be classified as Elevated.

#### 2.7.2 Statistical hypothesis, model, and method of analysis

#### **RBANS Total score and Index scores**

#### **Tables**

RBANS total score and RBANS Index scores will be summarized on the SAF.

#### **MMSE**

#### **Tables**

MMSE total score and the sub-scores on each of the five domains (orientation, registration, attention, recall, and language) will be summarized on the SAF.

# **Raven's Progressive Matrices**

#### **Tables**

Raven's total score (sum of all items from Sets A and B) and the sub-score included in the APCC (sum of items A2, A4, A8, B1-B6) will be summarized on the SAF.

# **Everyday Cognition scale (ECog-Subject and ECog-Informant)**

#### **Tables**

ECog total score will be summarized on the SAF for participants as well as for informants.



#### **Biomarkers in CSF**

#### **Tables**

All available AD related markers will be summarized for actual values as well as for change from baseline.

Baseline ratios for p-Tau/A $\beta$ 1-42 were used to determine Elevated /Not elevated brain Amyloid status and results will be reported as described in Section 2.7.1.

#### **Figures**

Box-plots for CSF parameters (Total tau, p-tau, A $\beta$ 1-40 and A $\beta$ 1-42) and ratio A $\beta$ 1-42/A $\beta$ 1-40 over time by treatment group will be provided

#### Biomarkers in blood:

# **Serum Light Chain Neurofilaments (NFL)**

#### **Tables**

Available measurements for NFL from serum will be summarized for actual values as well as for change from baseline.

#### **Figures**

Box-plots for serum NFL over time by treatment group will be provided

# Plasma Amyloid Beta-40 (Aβ<sub>1-40</sub>)

#### **Tables**

Available measurements for  $A\beta_{1-40}$  from plasma will be summarized for actual values as well as for change from baseline.

#### **PET SUVR**

# Listing

PET SUVR listing will be reported.

# Analysis of positive/negative amyloid levels

#### **Tables**

Amyloid levels (Positive/Negative) by method CSF and PET will be summarized as frequencies and percentages.

# 2.7.3 Handling of missing values/censoring/discontinuations

Due to the early termination of the trial, analyses of secondary efficacy variables will in general be based on observed cases only, i.e. there will be no imputation of missing data. Exception applies to missing data in RBANS Index scores, i.e., missing values for RBANS Index scores may be imputed using the imputation rule defined in Appendix 5.1.3.3.1.

# 2.8 Safety analyses

Reporting of safety data will be based on the SAF. Safety assessments will include adverse events, serious adverse events, deaths, laboratory data (hematology, blood chemistry, urinalysis), vital signs, ECG, safety MRI, physical and neurological examination, prospective suicidality assessment, dermatology photo report.

Summary statistics for categorical data will typically include frequencies and percentages.

For safety parameters, the summaries will be based on worst available observation in an analysis window. The analysis window and definition of worst value is present in Appendix 5.7.

#### 2.8.1 Adverse events (AEs)

Treatment-emergent AEs (TEAEs) are events that either started after the first dose of study drug or events present prior to the start of study drug but increased in severity since the first dose. Adverse events reported within 31 days (5 half-lives) from study drug discontinuation date (i.e., last dose date) will be considered as TEAE. AEs reported more than 31 days after study drug discontinuation will not be considered treatment emergent (non-TEAE).

TEAEs and non-TEAEs will be summarized separately on the SAF.

#### **Tables**

TEAEs, SAEs, deaths and non-TEAEs will be summarized as follows

- TEAEs regardless of relationship to study drug by SOC, PT and maximum severity
- non-TEAEs, regardless of relationship to study drug by SOC and PT
- TEAEs causing study drug discontinuation by SOC, PT and maximum severity
- TEAEs related to study drug by SOC, PT and maximum severity
- TE-SAEs regardless of relationship to study drug by SOC and PT and maximum severity

Note: For missing information on AE relationship to study drug, the most conservative approach will be considered: If information on relationship of the AE to study drug is missing, the AE will be considered as related to study drug for reporting TEAEs.

If information on severity of the AE is missing or unknown, the AE will be considered in Mild/Moderate Severity category.

The above summaries are generally without exposure adjustment, except from TEAEs by SOC and PT: this summary will be presented with exposure adjustment. The exposure-adjusted incidence rate of adverse events is defined as the number of participants with the adverse event divided by total participant years at risk in the treatment group. The time at risk for each participant will differ for each adverse event. For participants with events, only the time until the first event contributes to the total participant years at risk. For participants who do not experience the event, the time at risk will be calculated using the duration of exposure as defined in Section 2.4.1. The exposure-adjusted incident rate will be summarized per 100 participant years. For participants with multiple occurrences of the same event, the event will be counted only once per participant.

Adverse events will be reported according to the latest MedDRA dictionary version available at the time of database lock.

If a participant reported more than one adverse event within the same PT, the adverse event with the greatest severity will be counted. If a participant reported more than one adverse event within the same SOC, the participant will be counted only once with the greatest severity at the SOC level, wherever applicable. Sorting order for the AE summaries will be as follows:

- For summaries by SOC, SOC will be presented in alphabetical order.
- For summaries by SOC and PT, SOC will presented in alphabetical order; PT will be sorted within system organ class in alphabetical order.

#### Listings

All AEs will be listed ordered by country/center/participant and event date. Supplementary data for dermatological adverse events will also be listed (i.e., distribution of pruritus, presence, laterality and directionality).

# 2.8.1.1 Adverse events of special interest / grouping of AEs

An adverse event of special interest (AESI) is a set of adverse events that are of scientific and medical concern specific to a compound. These groupings are defined using MedDRA terms, SMQs (standardized MedDRA queries), HLGTs (high level group terms), HLT (high level terms) and PTs (preferred terms).

Customized SMQs (Novartis MedDRA queries, NMQ) may also be used. An NMQ is a customized group of search terms which defines a medical concept for which there is no official

SMQ available or the available SMQ does not completely fit the need. It may include a combination of single terms and/or an existing SMQ, narrow or broad.

AESIs as specified in the CNP520-specific Development Safety Profiling Plan (DSPP) are grouped in the corresponding Case Retrieval Sheet (eCRS) and analysed as a specific group along with other risk search terms.

The search criteria for each of the risks and events will be based on MedDRA and will be comprised by the eCRS. The most recent eCRS at the time of database lock will be used to determine the MedDRA search criteria for identification of the adverse events of special interests

#### **Tables**

Number and percentages of participants with treatment emergent adverse events of special interest by risk and MedDRA levels will be summarized on SAF.

#### 2.8.2 Deaths

#### **Tables**

Deaths regardless of relationship to study drug by SOC and PT will be summarized on the SAF.

# Listings

Deaths will also be listed separately.

# 2.8.3 Laboratory data

#### **Tables**

Number and percentages of participants with newly occurring or worsening laboratory abnormalities meeting the clinically notable criteria at any time post-baseline visit will be summarized for all parameters as specified in Appendix 5.6 of this document.

For a participant to meet the criterion of a newly occurring clinically notable value, the participant needs to have a baseline value that is not clinically notable for that parameter. For a participant to meet the criterion of a worsening clinically notable value, the participant needs to have a baseline value that is clinically notable and also have a worse post-baseline value. For participants with missing baseline value, any post-baseline notable value will be considered as newly occurring.

For each participant, all available post-baseline laboratory tests will be used to compare with the notable criteria. If at least one of the results, for a particular parameter, exceeds the criteria, the value will be considered as clinically notable abnormal for that parameter. A participant can be counted in both, low and high categories.

The upper limit of normal (ULN) for each parameter is available in the lab dataset. All available post-baseline laboratory tests will be used to compare with the criteria specified in Appendix 5.6. If at least one of the results, for a particular parameter, exceeds the criteria, the value will be considered as notable abnormal for that parameter. To categorize the abnormality, use the worst case within a lab parameter for a participant if multiple abnormality occurrences exist for the same lab parameter.

The laboratory parameters will be reported in SI units.

The number and percentage of participants with newly occurring or worsening liver enzyme abnormalities meeting the clinically notable criteria at any time post-baseline visit as specified in Appendix 5.3 will be summarized.

#### **Figures**

Box-plots for lab parameters of hematology, biochemistry and urinalysis over time by treatment group will be provided:

#### 2.8.4 Other safety data

# 2.8.4.1 ECG and cardiac imaging data

12-lead ECGs will be performed at screening and throughout the study in supine position. The ECG values will be interpreted and analyzed centrally. The QT intervals will be corrected according to the formula by Fridericia:

Fridericia's formula:  $QTcF = QT/RR^{1/3}$ 

#### **Tables**

The number and percentage of participants with newly occurring or worsening clinically notable ECG abnormalities at any time post-baseline visit will be summarized for all parameters as specified in Appendix 5.6.

# **Figures**

Box plots over time will be presented by ECG parameter and treatment group.

# 2.8.4.2 Vital signs

#### **Tables**

Parameters to be summarized are the following:

- Change from baseline in body weight will be summarized by visit including last assessment on treatment and last assessment off treatment.
- Vital signs: clinically notable changes (Body weight change will also be split by weight loss and weight gain).

The number and percentage of participants with clinically notable vital signs abnormalities at any time post-baseline visit will be summarized. The criteria of clinically notable vital signs are provided in Appendix 5.6.

Clinically notable weight changes of participants will be further investigated with the following summaries:

Frequency table will be presented for clinically notable weight changes (decrease/increase from baseline  $\geq$ 7% from baseline weight) during the treatment phase, by baseline weight categories ( $\leq$ 55 kg, 55 -  $\leq$ 70 kg, 70 -  $\leq$ 84 kg,  $\geq$ 84 kg) and by gender (Male, Female)

Participant demographics and other baseline characteristics with clinically notable weight decrease (loss) will be summarized.

# **Figures**

For the following parameters, box-plots by visit will be created: Heart Rate, Systolic BP, Diastolic BP, body weight.

# 2.8.4.3 Prospective Suicidality Assessment

The Columbia-Suicide Severity Rating Scale (C-SSRS) is a questionnaire that prospectively assesses Suicidal Ideation and Suicidal Behavior. The electronic version, the eC-SSRS will be administered as described in the visit schedule of the study protocols and may also include unscheduled visits. At the first time of administration of the eC-SSRS, a retrospective assessment of suicidal behavior and ideation will be collected across lifetime. This data will be used to check inclusion/exclusion criteria. At all other scheduled assessments of suicidal behavior and ideation, any occurrence since the last visit will be collected.

The data will be reported by analysis period. The following three periods have been identified to cover lifetime history, the time between collection of lifetime history and start of study drug intake, and the time on study drug.

# **Tables**

The number and percentage of participants pertaining to each of the categories of suicidal ideation and behaviors will be presented by analysis period and treatment.

The analysis periods will be defined as follows

- 1. Lifetime history: Lifetime assessment occurs only once (Screening visit (Visit 201).
- 2. Post disclosure pre-treatment period: next assessment scheduled at the baseline visit (Visit 301) and unscheduled visit falling into Screening 12-week period
- 3. Post baseline: all visits after baseline visit (including unscheduled).

The summaries will show numbers and percentages of participants who have an answer "yes" to a suicidal behavior or ideation category at any time within the corresponding analysis period.

# Listings

For participants with any assessment that meets the criteria to trigger the recording of an SAE as specified in the study protocols, a full listing will be presented. The criteria for SAE reporting are as follows:

If, at any time, the score is "Yes" on item 4 or item 5 of the Suicidal Ideation section of the C-SSRS or "Yes". All such cases regardless of whether there was an SAE reported or not will be listed.

# 2.8.4.4 Safety MRI

Safety MRI findings will be summarized overall (at any visit) for ARIA-E, ARIA-H and White matter disease findings.

Worsening of white matter disease is defined on the age-related white matter changes rating Scale (ARWMC) which is rated on a 4 point (0-3) scale per region (bilaterally) on the following

5 different brain regions: Frontal Lobe, Parieto-Occipital, Temporal Lobe, Infratentorial area, Basal ganglia. ARWMC composite score is the sum of individual ARWMC scores from the 5 regions and ranges from 0 to 15. The ARWMC composite score will be used to summarize the white matter disease findings.

The definitions of the rating scores is shown in the below Table 2-4.

Table 2-4 The ARWMC Rating Scale for MRI

| Score | Definition |
|---|---|
| White matter lesions | |
| 0 | No lesions (including symmetrical, well-defined caps or bands) |
| 1 | Focal lesions |
| 2 | Beginning confluence of lesions |
| 3 | Diffuse involvement of the entire region, with or without involvement of U fibers |
| Basal ganglia lesions | |
| 0 | No lesions |
| 1 | 1 focal lesion (≥5 mm) |
| 2 | >1 focal lesion |
| 3 | Confluent lesions |

#### **Tables**

For ARIA-E, the following parameters will be presented

• Participants with any new ARIA-E (mild, moderate and severe) since Baseline,

For ARIA-H, the following parameters will be presented

- Participants with > 4 new microhemorrhages or any new macrohemorrhage ≥ 10 mm in diameter since the Baseline MRI assessment OR
- Participants with >10 microhemorrhages (new hemosiderin deposits < 10 mm) Or ≥ 2 macrohemorrhages or ≥ 2 areas of superficial siderosis (large area of hemosiderin deposition ≥ 10 mm)

For white matter disease, the following parameters will be presented

• Participants with a white matter disease score increase since Baseline

#### Listings

Detailed safety MRI listings will be produced for participants with new occurrences or worsening (including Other MRI abnormalities) of identified findings.



# 2.11 Patient reported outcomes

The analysis for the patient reported outcome ECog, along with the Informant (study partner) version, is described within the secondary efficacy variables Section 2.7, and eCSSRS is described in the safety analysis Section 2.8.

#### 2.12 Biomarkers

The biomarkers are described in secondary variables Section 2.7.



# 2.14 Interim analysis

Due to early termination of the studies, the planned IA for CNP520 will not be performed.







# 4 Change to protocol specified analyses

SAF definition (defined in Section 2.2) is different from the protocol defined SAF definition.

An additional analysis set, mSAF, has been defined.

The following analysis were defined in the protocol but will not be performed due to early termination of the study:

- Primary analysis for both the primary endpoints
- Sensitivity to the primary analysis
- Supportive analysis to primary endpoints
- MMRM analysis to key secondary endpoint
- MMRM analysis to secondary efficacy endpoints

The following analysis were not defined in the protocol but will be added:

- All the efficacy analysis(except worsening in cognition and reversibility) will be performed on the SAF
- Worsening in cognition and reversibility as efficacy analysis using the mSAF

# 5 Appendix

# 5.1 Imputation rules

# 5.1.1 Study drug

If study treatment end date is missing, then treatment epoch completion date will be considered the last dose date, the rule will be provided in Programming Dataset Specification (PDS) document in details.

# 5.1.2 AE date imputation

Rules for imputing AE end date or start date will be provided in Programming Dataset Specification (PDS) document in details.

# 5.1.3 Concomitant medication date imputation

Rules for imputing the CM end date or start date will be provided in Programming Dataset Specification (PDS) document in details.

# 5.1.3.1 Prior therapies date imputation

Not Applicable.

# 5.1.3.2 Post therapies date imputation

Rules for imputing the post non-drug therapies end date or start date will be provided in Programming Dataset Specification (PDS) document in details.

# 5.1.3.3 Other imputations

# 5.1.3.3.1 Missing values from the same latent variable

For subtests that contribute to the same latent construct variable (Table 5-1), the following rule for missing subtests will be applied: When less than or equal to 50% of the related subtests within a constructed latent variable is missing, these missing subtests will be imputed from the remaining subtests contributing to its latent variable, standardized so that each subtest contributes the same weight to the construct as it would have if measured.

Table 5-1 Latent construct variables and their corresponding subtests

| Latent construct variable | Subtests |
|---|---|
| Immediate Memory Index score | List Learning and Story Memory |
| Visuospatial/Constructional Index Score | Figure Copy and Line Orientation |
| Language Index Score | Semantic Fluency and Picture Naming |
| Attention Index Score | Coding and Digital Span |
| Delayed Memory Index Score | List Recall, Story Recall, Figure Recall and List Recognition |
| Raven's matrices contributing to APCC | A2, A4, A8, B1-B6 |

This is done by calculating the total subscale-weight adjusted observed subtests (i), divided by the maximum weight-adjusted values possible for the observed subtests (i). This will provide the proportion to apply to the missing subtest (j) maximum possible value in order to obtain its imputed value as follows:

```
 missing \ subtest_{j} \\ = \frac{\sum_{i=1}^{n} (weight_{i} \times observed \ subtest_{i})}{\sum_{i=1}^{n} (weight_{i} \times observed \ subtest \ max_{i})} \times \ missing \ subtest_{j} \ max.
```

Missing subtests that could not borrow information from observed related subtests and construct variable values which could not be calculated from their underlying observed/imputed values will be regarded as MAR and will not be imputed.

# 5.2 AEs coding/grading

The MedDRA version which will be available at the time of database lock, will be used for the coding purpose of the adverse events.

# 5.3 Laboratory parameters derivations

Table 5-2 Liver Event and Laboratory Trigger Definitions

| | Definition/ threshold |
|---|---|
| LIVER<br>LABORATORY<br>TRIGGERS | 3×ULN < ALT / AST ≤ 5×ULN<br>1.5×ULN < TBL ≤ 2×ULN |

| LIVER EVENTS | ALT or AST > 5 × ULN |
|---|---|
| | ALP > 2×ULN (in the absence of known bone pathology) |
| | TBL > 2×ULN (in the absence of known Gilbert syndrome) |
| | ALT or AST > 3×ULN and INR > 1.5 |
| | Potential Hy's Law cases (defined as ALT or AST > 3×ULN and TBL > 2×ULN [mainly conjugated fraction] without notable increase in ALP to > 2×ULN) |
| | Any clinical event of jaundice (or equivalent term) |
| | ALT or AST > 3×ULN accompanied# by (general) malaise, fatigue, abdominal pain, nausea, or vomiting, or rash with eosinophilia Any adverse event potentially indicative of a liver toxicity * |

<sup>\*</sup>These events cover the following: hepatic failure, fibrosis and cirrhosis, and other liver damagerelated conditions; the non-infectious hepatitis; the benign, malignant and unspecified liver neoplasms

ALP = alkaline phosphatase; ALT = Alanine aminotransferase; AST = Aspartate aminotransferase TBL: total bilirubin; ULN: upper limit of normal

<sup>#</sup>Consider these adverse events in a window from 30 days before the liver event criteria (ALT or AST >  $3 \times ULN$ ) to 30 days after the liver event criteria (ALT or AST >  $3 \times ULN$ ).

| Table 3-3 Specific ferial alert criteria and action | Table 5-3 | Specific renal alert criteria and actions |
|---|---|---|
|---|---|---|

| | Definition/ threshold |
|---|---|
| Serum event | Serum creatinine increase 25 – 49% compared to baseline |
| | Acute Kidney Injury: Serum creatinine increase ≥ 50% compared to baseline |
| Urine event | New dipstick proteinuria ≥ 1+ |
| | Albumin- or Protein-creatinine ratio increase ≥ 2-fold |
| | ACR $\geq$ 30 mg/g or $\geq$ 3 mg/mmol; |
| | PCR ≥ 150 mg/g or > 15 mg/mmol |
| | New dipstick glycosuria ≥ 1+ not due to diabetes |
| | New dipstick hematuria ≥ 1+ not due to trauma* |

ACR = Albumin-creatinine ratio; PCR = Protein-creatinine ratio

#### 5.4 Statistical models

SAS codes for all statistical methodology described in this section will be included as programming note in TFL Shells.

# 5.4.1 Primary analysis

# Kaplan Meier approach for TTE

The Kaplan-Meier estimates of the survival functions for each treatment will be plotted. The plot will include the number of participants at risk for each treatment group at pre-specified timepoints. Median time to event and quartiles including 95% confidence intervals, if estimable, will be provided for each treatment group using the SAS procedure LIFETEST. The confidence intervals will be based on log-log transformation. For each treatment group and time interval: participants at risk, participants with event, participants with event divided by participants at risk, cumulative participants with event and cumulative event probability including 95% confidence interval will be provided.

#### **5.4.2** Additional SAS outputs

For the below mentioned analyses, additional (raw) SAS outputs resulted from SAS/STAT procedures or statistical derivations will be presented and used for CSR Appendix 16.1.9:

- Effect Size and 80% Confidence Intervals for APCC score, RBANS Total, RBANS Index scores
- Time to event (TTE) analyses:
  - Time to first confirmed diagnosis of MCI due to AD or Dementia due to AD-SAF
  - Time to first change in diagnosis classification-SAF
  - Time to first change in diagnosis classification when participants are on treatment-SAF
  - Time to first change in diagnosis classification when participants are on treatmentmSAF

<sup>\*</sup>Consider adverse event (injury) in a window from 30 days before the hematuria criteria.
- Time to first decrease in RBANS Total >= 14 points when participants are on treatment-SAF
- Baseline comparability

Further details for these additional SAS outputs will be described in the programming notes of the respective shells in the TFL shells Section 16.1.9.

### 5.5 Rule of exclusion criteria of analysis sets

The important protocol deviations are defined in below Table 5-4 with deviation ID, deviation code and it's corresponding text description.

Rule of exclusion criteria from analysis sets due to important protocol deviations (if any) will be included prior to database lock in a separate document in CREDI.

The Non-PD criteria for exclusion from analysis sets is explained in below Table 5-5.

Table 5-4 Deviation codes description

| Deviation code | Text description | Deviation ID |
|---|---|---|
| 1 | SELECTION CRITERIA NOT MET | INCLXX<br>EXCLXX |
| 2 | PARTICIPANT NOT WITHDRAWN AS PER<br>PROTOCOL | WITHXX |
| 4 | TREATMENT DEVIATION | TRTXX |
| 5 | PROHIBITED CONCOMITANT MEDICATION | COMDXX |
| 998 | OTHER | OTHXX |

### Table 5-5 Participant Classification

| | = | |
|---|---|---|
| Analysis Set | PD ID that | Non-PD criteria that cause |
| | cause patients to be excluded | patients to be excluded |
| Screened Set | NA | Not having informed consent; |
| | | Not having screening epoch disposition |
| | | page |
| RAS | NA | Not randomized |
| SAF | NA | No double-blind study drug taken |

# 5.6 Notable and abnormality criteria

Table 5-6 Clinically notable criteria for vital signs

| Vital Sign Variable | Notable Criteria |
|---------------------|----------------------------------------------------|
| Pulse (beats/min) | > 120bpm or Increase of ≥15 bpm from baseline |
| | or |
| | < 50bpm or Decrease of ≥15 bpm from baseline |
| Systolic BP (mmHg) | >180 mm Hg or Increase of ≥20 mm Hg from baseline |
| | Or |
| | < 90 mm Hg or Decrease of ≥ 20 mm Hg from baseline |
| Diastolic BP (mmHg) | > 105 mmHg or Increase of ≥ 15 mm Hg from baseline |
| | Or |
| | < 50 mmHg or Decrease of ≥ 15 mm Hg from baseline |
| Body weight (kg) | Decrease ≥ 7% from baseline weight |
| | Increase ≥ 7% from baseline weight |

Table 5-7 Clinically notable criteria for selected hematology tests

| | SI units | | US or other units | |
|---|---|---|---|---|
| Laboratory parameter | Lower bound | Upper bound | Lower bound | Upper bound |
| Hemoglobin | 70 (g/L) | 200 (g/L) | 7 (g/dL) | 20 (g/dL) |
| White Cell count | 2 (x10 <sup>9</sup> /L) | 30 (x10 <sup>9</sup> /L) | 2 (x10 <sup>3</sup> /uL) | 30 (x10 <sup>3</sup> /uL) |

| | SI units | | US or other units | |
|---|---|---|---|---|
| Laboratory parameter | Lower bound | Upper bound | Lower bound | Upper bound |
| Platelets | 50 (x10 <sup>9</sup> /L) | 1000<br>(x10 <sup>9</sup> /L) | 50 (x10 <sup>3</sup> /uL) | 1000<br>x10 <sup>3</sup> /uL) |

# Table 5-8 Clinically notable criteria for selected blood chemistry tests

| | • | | | • |
|---|---|---|---|---|
| | SI units | | US or other units | |
| Laboratory parameter | Lower bound | Upper bound | Lower bound | Upper bound |
| Sodium | 125 (mmol/L) | 155 (mmol/L) | 125 (mmol/L) | 155 (mmol/L) |
| Potassium | 3 (mmol/L) | 6 (mmol/L) | 3 (mmol/L) | 6 (mmol/L) |
| Calcium | 1.5 (mmol/L) | 3 (mmol/L) | 6 (mg/dL) | 12 (mg/dL) |
| Magnesium | 0.4 (mmol/L) | 1.2 (mmol/L) | 1 (mg/dL) | 3 (mg/dL) |
| Bilirubin (Total) | - | 41 (umol/L) | - | 2.4 (mg/dL) |
| AST | - | > 3×ULN | - | > 3×ULN |
| ALT | - | > 3×ULN | - | > 3×ULN |
| Alkaline<br>Phosphatase<br>(Male) | - | > 2×ULN | - | > 2×ULN |
| Alkaline<br>Phosphatase<br>(Female) | - | > 2×ULN | - | > 2×ULN |
| Creatinine | - | increase 25 –<br>49% compared<br>to baseline | - | increase 25 –<br>49% compared<br>to baseline |
| | | increase<br>≥ 50%<br>compared to<br>baseline | | increase ≥ 50% compared to baseline |

### Table 5-9 ECG Abnormality Ranges

| | Abnormality Flags |
|-----------------------------------------|----------------------|
| ECG Parameter | Absolute |
| PR interval | > 250 msec |
| QRS Interval | > 140 msec |
| OT-F lot-mad | >= 500 msec (All) |
| QTcF Interval (Fridericia's correction) | >= 450 msec (Male) |
| (i riuericia s correction) | >= 470 msec (Female) |

| ECG Parameter | Abnormality Flags Absolute |
|-------------------------|----------------------------|
| QT change from baseline | >60 msec |

# 5.7 Analysis windows rules

Table 5-10 Raven's, MMSE and CDR, ECog

| | | Analysis | Analysis window* | |
|---|---|---|---|---|
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 301 | Baseline (Day 1) | -1 | 1 | Baseline |
| 302 | | | | |
| 303 | | | | |
| 304 | | | | |
| 305 | | | | |
| 306 | Week 26 (Day 182) | 2 | 272 | Week 26 |
| 307 | | | | |
| 308 | Week 52 (Day 364) | 273 | 454 | Week 52 |
| 309 | | | | |
| 310 | Week 78 (Day 546) | 455 | 636 | Week 78 |
| 311 | | | | |
| 312 | Week 104 (Day 728) | 637 | 818 | Week 104 |
| 313 | | | | |
| 314 | Week 130 (Day 910) | 819 | 1000 | Week 130 |
| 315 | | | | |
| 316 | Week 156 (Day 1092) | 1001 | 1182 | Week 156 |
| 317 | | | | |
| 318 | Week 182 (Day 1274) | 1183 | 1364 | Week 182 |
| 319 | | | | |
| 320 | Week 208 (Day 1456) | 1365 | 1546 | Week 208 |
| 321 | | | | |
| 322 | Week 234 (Day 1638) | 1547 | 1728 | Week 234 |
| 323 | | | | |
| 324 | Week 260 (Day 1820) | 1729 | 1910 | Week 260 |
| 325 | | | | |
| 326 | Week 286 (Day 2002) | 1911 | 2092 | Week 286 |
| 327 | | | | |
| 328 | Week 312 (Day 2184) | 2093 | 2274 | Week 312 |
| 329 | | | | |
| 330 | Week 338 (Day 2366) | 2275 | 2456 | Week 338 |
| 331 | | | | |
| 332 | Week 364 (Day 2548) | 2457 | 2638 | Week 364 |

| | | Analysis w | Analysis window* | |
|---|---|---|---|---|
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 333 | | | | |
| 334 | Week 390 (Day 2730) | 2639 | 2820 | Week 390 |
| 335 | | | | |
| 336 | Week 416 (Day 2912) | 2821 | Until EOS | Week 416 |

# Table 5-11 RBANS,

| | | Analysis | Analysis window* | |
|---|---|---|---|---|
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 301 | Baseline (Day 1) | -1 | 1 | Baseline |
| 302 | | | | |
| 303 | | | | |
| 304 | Week 13 (Day 91) | 2 | 136 | Week 13 |
| 305 | | | | |
| 306 | Week 26 (Day 182) | 137 | 272 | Week 26 |
| 307 | | | | |
| 308 | Week 52 (Day 364) | 273 | 454 | Week 52 |
| 309 | | | | |
| 310 | Week 78 (Day 546) | 455 | 636 | Week 78 |
| 311 | | | | |
| 312 | Week 104 (Day 728) | 637 | 818 | Week 104 |
| 313 | | | | |
| 314 | Week 130 (Day 910) | 819 | 1000 | Week 130 |
| 315 | | | | |
| 316 | Week 156 (Day 1092) | 1001 | 1182 | Week 156 |
| 317 | | | | |
| 318 | Week 182 (Day 1274) | 1183 | 1364 | Week 182 |
| 319 | | | | |
| 320 | Week 208 (Day 1456) | 1365 | 1546 | Week 208 |
| 321 | | | | |
| 322 | Week 234 (Day 1638) | 1547 | 1728 | Week 234 |
| 323 | | | | |
| 324 | Week 260 (Day 1820) | 1729 | 1910 | Week 260 |
| 325 | | | | |
| 326 | Week 286 (Day 2002) | 1911 | 2092 | Week 286 |
| 327 | | | | |
| 328 | Week 312 (Day 2184) | 2093 | 2274 | Week 312 |
| 329 | | | | |
| 330 | Week 338 (Day 2366) | 2275 | 2456 | Week 338 |
| 331 | | | | |
| 332 | Week 364 (Day 2548) | 2457 | 2638 | Week 364 |

| | | Analysis | Analysis window* | |
|---|---|---|---|---|
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 333 | | | | |
| 334 | Week 390 (Day 2730) | 2639 | 2820 | Week 390 |
| 335 | | | | |
| 336 | Week 416 (Day 2912) | 2821 | Until EOS | Week 416 |

 Table 5-12
 Physical / Neurological exams, ECG, laboratory tests

| | , | | , | • |
|--------------|---------------------|----------|-----------|-------------|
| | | Analysis | window* | |
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 301 | Baseline (Day 1) | -1 | 1 | Baseline |
| 302 | | | | |
| 303 | | | | |
| 304 | Week 13 (Day 91) | 2 | 136 | Week 13 |
| 305 | , , , | | | |
| 306 | Week 26 (Day 182) | 137 | 272 | Week 26 |
| 307 | | | | |
| 308 | Week 52 (Day 364) | 273 | 454 | Week 52 |
| 309 | , , | | | |
| 310 | Week 78 (Day 546) | 455 | 636 | Week 78 |
| 311 | | | | |
| 312 | Week 104 (Day 728) | 637 | 818 | Week 104 |
| 313 | | | | |
| 314 | Week 130 (Day 910) | 819 | 1000 | Week 130 |
| 315 | | | | |
| 316 | Week 156 (Day 1092) | 1001 | 1182 | Week 156 |
| 317 | | | | |
| 318 | Week 182 (Day 1274) | 1183 | 1364 | Week 182 |
| 319 | | | | |
| 320 | Week 208 (Day 1456) | 1365 | 1546 | Week 208 |
| 321 | | | | |
| 322 | Week 234 (Day 1638) | 1547 | 1728 | Week 234 |
| 323 | | | | |
| 324 | Week 260 (Day 1820) | 1729 | 1910 | Week 260 |
| 325 | | | | |
| 326 | Week 286 (Day 2002) | 1911 | 2092 | Week 286 |
| 327 | | | | |
| 328 | Week 312 (Day 2184) | 2093 | 2274 | Week 312 |
| 329 | | | | |
| 330 | Week 338 (Day 2366) | 2275 | 2456 | Week 338 |
| 331 | | | | |
| 332 | Week 364 (Day 2548) | 2457 | 2638 | Week 364 |
| 333 | | | | |
| 334 | Week 390 (Day 2730) | 2639 | 2820 | Week 390 |
| 335 | | | | |
| 336 | Week 416 (Day 2912) | 2821 | Until EOS | Week 416 |

Table 5-13 Safety MRI, volumetric MRI, functional MRI

| 302 303 304 305 306 Week 26 (Day 182) 2 272 Week 26 307 308 Week 52 (Day 364) 273 545 Week 52 309 310 311 312 Week 104 (Day 728) 546 909 Week 104 313 314 315 316 Week 156 (Day 1092) 910 1273 Week 156 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | | | Analysis | window* | |
|---|---|---|---|---|---|
| 302 303 304 305 306 Week 26 (Day 182) 2 272 Week 26 307 308 Week 52 (Day 364) 273 545 Week 52 309 310 311 312 Week 104 (Day 728) 546 909 Week 104 313 314 315 316 Week 156 (Day 1092) 910 1273 Week 156 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 302 303 304 305 306 Week 26 (Day 182) 2 272 Week 26 307 308 Week 52 (Day 364) 273 545 Week 52 309 310 311 312 Week 104 (Day 728) 546 909 Week 104 313 314 315 316 Week 156 (Day 1092) 910 1273 Week 156 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | | | | | |
| 303 304 305 306 Week 26 (Day 182) 2 272 Week 26 307 308 Week 52 (Day 364) 273 545 Week 52 309 310 311 312 Week 104 (Day 728) 546 909 Week 104 313 314 315 316 Week 156 (Day 1092) 910 1273 Week 156 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 301 | Baseline (Day 1) | -1 | 1 | Baseline |
| 304 305 306 Week 26 (Day 182) 2 272 Week 26 307 308 Week 52 (Day 364) 273 545 Week 52 309 310 311 312 Week 104 (Day 728) 546 909 Week 104 313 314 315 316 Week 156 (Day 1092) 910 1273 Week 156 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 326 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 302 | | | | |
| 305 | 303 | | | | |
| 306 Week 26 (Day 182) 2 272 Week 26 307 308 Week 52 (Day 364) 273 545 Week 52 309 310 311 312 Week 104 (Day 728) 546 909 Week 104 313 314 315 316 Week 156 (Day 1092) 910 1273 Week 156 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 304 | | | | |
| 307 308 Week 52 (Day 364) 273 545 Week 52 309 310 311 312 Week 104 (Day 728) 546 909 Week 104 313 314 315 316 Week 156 (Day 1092) 910 1273 Week 156 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 305 | | | | |
| 308 | 306 | Week 26 (Day 182) | 2 | 272 | Week 26 |
| 309 310 311 312 Week 104 (Day 728) 546 909 Week 104 313 314 315 316 Week 156 (Day 1092) 910 1273 Week 156 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 307 | | | | |
| 310 311 312 Week 104 (Day 728) 546 909 Week 104 313 314 315 316 Week 156 (Day 1092) 910 1273 Week 156 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 308 | Week 52 (Day 364) | 273 | 545 | Week 52 |
| 311 | 309 | | | | |
| 312 Week 104 (Day 728) 546 909 Week 104 313 314 315 316 Week 156 (Day 1092) 910 1273 Week 156 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 310 | | | | |
| 313 314 315 316 Week 156 (Day 1092) 910 1273 Week 156 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 311 | | | | |
| 314 | 312 | Week 104 (Day 728) | 546 | 909 | Week 104 |
| 315 316 Week 156 (Day 1092) 910 1273 Week 156 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 313 | | | | |
| 316 Week 156 (Day 1092) 910 1273 Week 156 317 | 314 | | | | |
| 317 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 315 | | | | |
| 318 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 316 | Week 156 (Day 1092) | 910 | 1273 | Week 156 |
| 319 320 Week 208 (Day 1456) 1274 1637 Week 208 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 317 | | | | |
| 320 Week 208 (Day 1456) 1274 1637 Week 208 321 | 318 | | | | |
| 321 322 323 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 319 | | | | |
| 322 | 320 | Week 208 (Day 1456) | 1274 | 1637 | Week 208 |
| 323 | 321 | | | | |
| 324 Week 260 (Day 1820) 1638 2001 Week 260 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 334 335 | 322 | | | | |
| 325 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 323 | | | | |
| 326 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 324 | Week 260 (Day 1820) | 1638 | 2001 | Week 260 |
| 327 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 325 | | | | |
| 328 Week 312 (Day 2184) 2002 2365 Week 312 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 334 335 | 326 | | | | |
| 329 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 | 327 | | | | |
| 330 331 332 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 335 | 328 | Week 312 (Day 2184) | 2002 | 2365 | Week 312 |
| 331 Week 364 (Day 2548) 2366 2729 Week 364 333 334 335 335 | 329 | | | | |
| 332 Week 364 (Day 2548) 2366 2729 Week 364<br>333 334 335 | 330 | | | | |
| 333<br>334<br>335 | 331 | | | | |
| 334<br>335 | 332 | Week 364 (Day 2548) | 2366 | 2729 | Week 364 |
| 335 | 333 | | | | |
| | 334 | | | | |
| 336 Wook 416 (Day 2012) 2720 Until EOS Wook 446 | 335 | | | | |
| 330 Week 410 (Day 2312) 2730 Ullill EOS Week 416 | 336 | Week 416 (Day 2912) | 2730 | Until EOS | Week 416 |



Table 5.15 Vital signs

| | | Analysis | window* | |
|--------------|---------------------|----------|-----------|-------------|
| Visit Number | Scheduled Timepoint | Lower | Upper | Visit Label |
| 301 | Baseline (Day 1) | -1 | 1 | Baseline |
| 302 | | | | |
| 303 | | | | |
| 304 | Week 13 (Day 91) | 2 | 136 | Week 13 |
| 305 | | | | |
| 306 | Week 26 (Day 182) | 137 | 227 | Week 26 |
| 307 | Week 39 (Day 273) | 228 | 318 | Week 39 |
| 308 | Week 52 (Day 364) | 319 | 409 | Week 52 |
| 309 | Week 65 (Day 455) | 410 | 500 | Week 65 |
| 310 | Week 78 (Day 546) | 501 | 591 | Week 78 |
| 311 | Week 91 (Day 637) | 592 | 682 | Week 91 |
| 312 | Week 104 (Day 728) | 683 | 773 | Week 104 |
| 313 | Week 117 (Day 819) | 774 | 864 | Week 117 |
| 314 | Week 130 (Day 910) | 865 | 955 | Week 130 |
| 315 | Week 143 (Day 1001) | 956 | 1046 | Week 143 |
| 316 | Week 156 (Day 1092) | 1047 | 1137 | Week 156 |
| 317 | Week 169 (Day 1183) | 1138 | 1228 | Week 169 |
| 318 | Week 182 (Day 1274) | 1229 | 1319 | Week 182 |
| 319 | Week 195 (Day 1365) | 1320 | 1410 | Week 195 |
| 320 | Week 208 (Day 1456) | 1411 | 1501 | Week 208 |
| 321 | Week 221 (Day 1547) | 1502 | 1592 | Week 221 |
| 322 | Week 234 (Day 1638) | 1593 | 1683 | Week 234 |
| 323 | Week 247 (Day 1729) | 1684 | 1774 | Week 247 |
| 324 | Week 260 (Day 1820) | 1775 | 1865 | Week 260 |
| 325 | Week 273 (Day 1911) | 1866 | 1956 | Week 273 |
| 326 | Week 286 (Day 2002) | 1957 | 2092 | Week 286 |
| 327 | | | | |
| 328 | Week 312 (Day 2184) | 2093 | 2274 | Week 312 |
| 329 | | | | |
| 330 | Week 338 (Day 2366) | 2275 | 2456 | Week 338 |
| 331 | | | | |
| 332 | Week 364 (Day 2548) | 2457 | 2638 | Week 364 |
| 333 | | | | |
| 334 | Week 390 (Day 2730) | 2639 | 2820 | Week 390 |
| 335 | | | | |
| 336 | Week 416 (Day 2912) | 2821 | Until EOS | Week 416 |

### **Analyses not by Analysis windows**

The following domains will not be analysed by analysis window, but according to the scheduled visit and/or visit day as applicable. Analysis windows will not be provided for these.

- Amyloid PET
- Tau PET
- CSF biomarkers
- Blood biomarkers (Serum/Plasma)
- T-cell response (Cohort I only)
- Drug administration
- C-SSRS

#### 5.8 RBANS Index tables

The RBANS index scores are obtained from the following five age adjusted tables corresponding to the respective total subtest scores.

Table 5-17 Immediate Memory Index Score Equivalents of Subtest Raw Score

| | | | Stor | y Mem | ory Tot | al Sco | re | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 |
| | | 0 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 1 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 2 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 3 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 4 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 5 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 6 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 7 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 8 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 9 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 10 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 11 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | | 12 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| | | 13 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| | | 14 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| ē | | 15 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| Score | | 16 | 49 | 49 | 49 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 69 | 76 | 78 | 83 | 83 | 83 | 83 | 83 | 87 | 94 | 100 |
| Total ( | | 17 | 49 | 49 | 49 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 69 | 76 | 78 | 83 | 83 | 83 | 83 | 83 | 87 | 94 | 100 |
| | | 18 | 53 | 53 | 53 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 73 | 78 | 81 | 85 | 85 | 85 | 85 | 85 | 90 | 97 | 103 |
| Learning | 50-59 | 19 | 53 | 53 | 53 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 73 | 78 | 81 | 85 | 85 | 85 | 85 | 85 | 90 | 97 | 103 |
| earı | | 20 | 53 | 53 | 53 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 73 | 78 | 81 | 85 | 85 | 85 | 85 | 85 | 90 | 97 | 103 |
| ist L | Ages | 21 | 57 | 57 | 57 | 57 | 57 | 61 | 61 | 61 | 65 | 65 | 69 | 69 | 73 | 76 | 76 | 81 | 83 | 87 | 87 | 87 | 87 | 87 | 94 | 100 | 106 |
| Ľ | 1 | 22 | 61 | 61 | 61 | 61 | 61 | 65 | 65 | 65 | 69 | 69 | 73 | 73 | 76 | 78 | 78 | 83 | 85 | 90 | 90 | 90 | 90 | 90 | 97 | 103 | 109 |

| | | Story | Memo | ory Tota | al Scor | e | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 |
| | 23 | 61 | 61 | 61 | 61 | 61 | 65 | 65 | 65 | 69 | 69 | 73 | 73 | 76 | 78 | 78 | 83 | 85 | 90 | 90 | 90 | 90 | 90 | 97 | 103 | 109 |
| • | 24 | 65 | 65 | 65 | 65 | 65 | 69 | 69 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 81 | 85 | 87 | 94 | 94 | 94 | 94 | 94 | 100 | 106 | 112 |
| • | 25 | 69 | 69 | 69 | 69 | 69 | 73 | 73 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 83 | 87 | 90 | 97 | 97 | 97 | 97 | 97 | 103 | 109 | 114 |
| | 26 | 73 | 73 | 73 | 73 | 73 | 76 | 76 | 76 | 78 | 78 | 81 | 81 | 83 | 85 | 85 | 90 | 94 | 100 | 100 | 100 | 100 | 100 | 106 | 112 | 117 |
| | 27 | 76 | 76 | 76 | 76 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 87 | 87 | 94 | 97 | 103 | 103 | 103 | 103 | 103 | 109 | 114 | 120 |
| | 28 | 76 | 76 | 76 | 76 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 87 | 87 | 94 | 97 | 103 | 103 | 103 | 103 | 103 | 109 | 114 | 120 |
| ĺ | 29 | 78 | 78 | 78 | 78 | 78 | 81 | 81 | 81 | 83 | 83 | 85 | 85 | 87 | 90 | 90 | 97 | 100 | 106 | 106 | 106 | 106 | 106 | 112 | 117 | 123 |
| | 30 | 81 | 81 | 81 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 94 | 100 | 103 | 109 | 109 | 109 | 109 | 109 | 114 | 120 | 126 |
| | 31 | 81 | 81 | 81 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 94 | 100 | 103 | 109 | 109 | 109 | 109 | 109 | 114 | 120 | 126 |
| | 32 | 81 | 81 | 81 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 94 | 100 | 103 | 109 | 109 | 109 | 109 | 109 | 114 | 120 | 126 |
| ĺ | 33 | 83 | 83 | 83 | 83 | 83 | 85 | 85 | 85 | 87 | 87 | 90 | 90 | 94 | 97 | 97 | 103 | 106 | 112 | 112 | 112 | 112 | 112 | 117 | 123 | 129 |
| | 34 | 85 | 85 | 85 | 85 | 85 | 87 | 87 | 87 | 90 | 90 | 94 | 94 | 97 | 100 | 100 | 106 | 109 | 114 | 114 | 114 | 114 | 114 | 120 | 126 | 132 |
| | 35 | 87 | 87 | 87 | 87 | 87 | 90 | 90 | 90 | 94 | 94 | 97 | 97 | 100 | 103 | 103 | 109 | 112 | 117 | 117 | 117 | 117 | 117 | 123 | 129 | 136 |
| | 36 | 87 | 87 | 87 | 87 | 87 | 90 | 90 | 90 | 94 | 94 | 97 | 97 | 100 | 103 | 103 | 109 | 112 | 117 | 117 | 117 | 117 | 117 | 123 | 129 | 136 |
| | 37 | 90 | 90 | 90 | 90 | 90 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 103 | 106 | 106 | 112 | 114 | 120 | 120 | 120 | 120 | 120 | 126 | 132 | 140 |
| | 38 | 94 | 94 | 94 | 94 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 109 | 114 | 117 | 123 | 123 | 123 | 123 | 123 | 129 | 136 | 144 |
| | 39 | 97 | 97 | 97 | 97 | 97 | 100 | 100 | 100 | 103 | 103 | 106 | 106 | 109 | 112 | 112 | 117 | 120 | 126 | 126 | 126 | 126 | 126 | 132 | 140 | 148 |
| | 40 | 100 | 100 | 100 | 100 | 100 | 103 | 103 | 103 | 106 | 106 | 109 | 109 | 112 | 114 | 114 | 120 | 123 | 129 | 129 | 129 | 129 | 129 | 136 | 144 | 152 |
| | 0 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | 1 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | 2 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | 3 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | 4 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | 5 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| | 6 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| - 69 | 7 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| 09 | 8 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| ges | 9 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |
| Ag | 10 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 44 | 49 | 49 | 53 | 53 | 57 | 61 | 61 | 69 | 73 | 78 | 78 | 78 | 78 | 78 | 83 | 87 | 94 |

| | Stor | y Mem | ory Tot | al Sco | re | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 |
| 11 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| 12 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| 13 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| 14 | 44 | 44 | 44 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 65 | 73 | 76 | 81 | 81 | 81 | 81 | 81 | 85 | 90 | 97 |
| 15 | 49 | 49 | 49 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 69 | 76 | 78 | 83 | 83 | 83 | 83 | 83 | 87 | 94 | 10 |
| 16 | 49 | 49 | 49 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 69 | 76 | 78 | 83 | 83 | 83 | 83 | 83 | 87 | 94 | 10 |
| 17 | 49 | 49 | 49 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 69 | 76 | 78 | 83 | 83 | 83 | 83 | 83 | 87 | 94 | 100 |
| 18 | 53 | 53 | 53 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 73 | 78 | 81 | 85 | 85 | 85 | 85 | 85 | 90 | 97 | 103 |
| 19 | 53 | 53 | 53 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 73 | 78 | 81 | 85 | 85 | 85 | 85 | 85 | 90 | 97 | 10 |
| 20 | 53 | 53 | 53 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 73 | 78 | 81 | 85 | 85 | 85 | 85 | 85 | 90 | 97 | 103 |
| 21 | 57 | 57 | 57 | 57 | 57 | 61 | 61 | 61 | 65 | 65 | 69 | 69 | 73 | 76 | 76 | 81 | 83 | 87 | 87 | 87 | 87 | 87 | 94 | 100 | 100 |
| 22 | 61 | 61 | 61 | 61 | 61 | 65 | 65 | 65 | 69 | 69 | 73 | 73 | 76 | 78 | 78 | 83 | 85 | 90 | 90 | 90 | 90 | 90 | 97 | 103 | 10 |
| 23 | 61 | 61 | 61 | 61 | 61 | 65 | 65 | 65 | 69 | 69 | 73 | 73 | 76 | 78 | 78 | 83 | 85 | 90 | 90 | 90 | 90 | 90 | 97 | 103 | 10 |
| 24 | 65 | 65 | 65 | 65 | 65 | 69 | 69 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 81 | 85 | 87 | 94 | 94 | 94 | 94 | 94 | 100 | 106 | 11: |
| 25 | 69 | 69 | 69 | 69 | 69 | 73 | 73 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 83 | 87 | 90 | 97 | 97 | 97 | 97 | 97 | 103 | 109 | 114 |
| 26 | 73 | 73 | 73 | 73 | 73 | 76 | 76 | 76 | 78 | 78 | 81 | 81 | 83 | 85 | 85 | 90 | 94 | 100 | 100 | 100 | 100 | 100 | 106 | 112 | 11 |
| 27 | 76 | 76 | 76 | 76 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 87 | 87 | 94 | 97 | 103 | 103 | 103 | 103 | 103 | 109 | 114 | 12 |
| 28 | 78 | 78 | 78 | 78 | 78 | 81 | 81 | 81 | 83 | 83 | 85 | 85 | 87 | 90 | 90 | 97 | 100 | 106 | 106 | 106 | 106 | 106 | 112 | 117 | 12 |
| 29 | 78 | 78 | 78 | 78 | 78 | 81 | 81 | 81 | 83 | 83 | 85 | 85 | 87 | 90 | 90 | 97 | 100 | 106 | 106 | 106 | 106 | 106 | 112 | 117 | 12 |
| 30 | 81 | 81 | 81 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 94 | 100 | 103 | 109 | 109 | 109 | 109 | 109 | 114 | 120 | 12 |
| 31 | 81 | 81 | 81 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 94 | 100 | 103 | 109 | 109 | 109 | 109 | 109 | 114 | 120 | 120 |
| 32 | 81 | 81 | 81 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 94 | 100 | 103 | 109 | 109 | 109 | 109 | 109 | 114 | 120 | 12 |
| 33 | 83 | 83 | 83 | 83 | 83 | 85 | 85 | 85 | 87 | 87 | 90 | 90 | 94 | 97 | 97 | 103 | 106 | 112 | 112 | 112 | 112 | 112 | 117 | 123 | 12 |
| 34 | 85 | 85 | 85 | 85 | 85 | 87 | 87 | 87 | 90 | 90 | 94 | 94 | 97 | 100 | 100 | 106 | 109 | 114 | 114 | 114 | 114 | 114 | 120 | 126 | 13 |
| 35 | 87 | 87 | 87 | 87 | 87 | 90 | 90 | 90 | 94 | 94 | 97 | 97 | 100 | 103 | 103 | 109 | 112 | 117 | 117 | 117 | 117 | 117 | 123 | 129 | 13 |
| 36 | 90 | 90 | 90 | 90 | 90 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 103 | 106 | 106 | 112 | 114 | 120 | 120 | 120 | 120 | 120 | 126 | 132 | 14 |
| 37 | 94 | 94 | 94 | 94 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 109 | 114 | 117 | 123 | 123 | 123 | 123 | 123 | 129 | 136 | 14 |
| 38 | 94 | 94 | 94 | 94 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 109 | 114 | 117 | 123 | 123 | 123 | 123 | 123 | 129 | 136 | 14 |
| 39 | 97 | 97 | 97 | 97 | 97 | 100 | 100 | 100 | 103 | 103 | 106 | 106 | 109 | 112 | 112 | 117 | 120 | 126 | 126 | 126 | 126 | 126 | 132 | 140 | 14 |

| | | Story | / Memo | ory Tota | al Scor | re | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 |
| | 40 | 100 | 100 | 100 | 100 | 100 | 103 | 103 | 103 | 106 | 106 | 109 | 109 | 112 | 114 | 114 | 120 | 123 | 129 | 129 | 129 | 129 | 129 | 136 | 144 | 152 |
| | 0 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 1 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 2 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 3 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 4 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 5 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 6 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 7 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 8 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 9 | 40 | 40 | 40 | 40 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 65 | 69 | 73 | 73 | 78 | 78 | 78 | 81 | 83 | 87 | 90 | 94 |
| | 10 | 44 | 44 | 44 | 44 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 73 | 76 | 76 | 81 | 81 | 81 | 83 | 85 | 90 | 94 | 97 |
| | 11 | 44 | 44 | 44 | 44 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 73 | 76 | 76 | 81 | 81 | 81 | 83 | 85 | 90 | 94 | 97 |
| | 12 | 44 | 44 | 44 | 44 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 73 | 76 | 76 | 81 | 81 | 81 | 83 | 85 | 90 | 94 | 97 |
| | 13 | 44 | 44 | 44 | 44 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 69 | 73 | 76 | 76 | 81 | 81 | 81 | 83 | 85 | 90 | 94 | 97 |
| | 14 | 49 | 49 | 49 | 49 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 73 | 76 | 78 | 78 | 83 | 83 | 83 | 85 | 87 | 94 | 97 | 100 |
| | 15<br>16 | 49<br>53 | 49<br>53 | 49<br>53 | 49<br>53 | 53<br>57 | 57<br>61 | 57<br>61 | 57<br>61 | 61<br>65 | 61<br>65 | 65<br>69 | 65<br>69 | 69<br>73 | 73<br>76 | 76<br>78 | 78<br>81 | 78<br>81 | 83<br>85 | 83<br>85 | 83<br>85 | 85<br>87 | 87<br>90 | 94<br>97 | 97 | 100 |
| | 17 | 53 | 53 | 53 | 53 | 57 | 61 | 61 | 61 | 65 | 65 | 69 | 69 | 73 | 76 | 78 | 81 | 81 | 85 | 85 | 85 | 87 | 90 | 97 | 100 | 103 |
| | 18 | 57 | 57 | 57 | 57 | 61 | 65 | 65 | 65 | 69 | 69 | 73 | 73 | 76 | 78 | 81 | 83 | 83 | 87 | 87 | 87 | 90 | 94 | 100 | 103 | 103 |
| | 19 | 61 | 61 | 61 | 61 | 65 | 69 | 69 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 85 | 85 | 90 | 90 | 90 | 94 | 97 | 103 | 106 | 100 |
| | 20 | 61 | 61 | 61 | 61 | 65 | 69 | 69 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 85 | 85 | 90 | 90 | 94 | 97 | 100 | 106 | 109 | 112 |
| | 21 | 65 | 65 | 65 | 65 | 69 | 73 | 73 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 85 | 87 | 87 | 94 | 94 | 94 | 97 | 100 | 106 | 109 | 112 |
| | 22 | 65 | 65 | 65 | 65 | 69 | 73 | 73 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 85 | 87 | 87 | 94 | 94 | 94 | 97 | 100 | 106 | 109 | 112 |
| | 23 | 69 | 69 | 69 | 69 | 73 | 76 | 76 | 76 | 78 | 78 | 81 | 81 | 83 | 85 | 87 | 90 | 90 | 97 | 97 | 97 | 100 | 103 | 109 | 112 | 114 |
| _ | 24 | 73 | 73 | 73 | 73 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 87 | 90 | 94 | 94 | 100 | 100 | 100 | 103 | 106 | 112 | 114 | 117 |
| 6/-0/ | 25 | 73 | 73 | 73 | 73 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 87 | 90 | 94 | 94 | 100 | 100 | 100 | 103 | 106 | 112 | 114 | 117 |
| <b>.</b> | 26 | 76 | 76 | 76 | 76 | 78 | 81 | 81 | 81 | 83 | 83 | 85 | 85 | 87 | 90 | 94 | 97 | 97 | 103 | 103 | 103 | 106 | 109 | 114 | 117 | 120 |
| Ages | 27 | 78 | 78 | 78 | 78 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 97 | 100 | 100 | 106 | 106 | 106 | 109 | 112 | 117 | 120 | 123 |

| | | | Story | / Mem | ory Tot | al Scoi | re | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 |
| | | 28 | 78 | 78 | 78 | 78 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 97 | 100 | 100 | 106 | 106 | 106 | 109 | 112 | 117 | 120 | 123 |
| | | 29 | 81 | 81 | 81 | 81 | 83 | 85 | 85 | 85 | 87 | 87 | 90 | 90 | 94 | 97 | 100 | 103 | 103 | 109 | 109 | 109 | 112 | 114 | 120 | 123 | 126 |
| | | 30 | 81 | 81 | 81 | 81 | 83 | 85 | 85 | 85 | 87 | 87 | 90 | 90 | 94 | 97 | 100 | 103 | 103 | 109 | 109 | 109 | 112 | 114 | 120 | 123 | 126 |
| | | 31 | 83 | 83 | 83 | 83 | 85 | 87 | 87 | 87 | 90 | 90 | 94 | 94 | 97 | 100 | 103 | 106 | 106 | 112 | 112 | 112 | 114 | 117 | 123 | 126 | 129 |
| | | 32 | 85 | 85 | 85 | 85 | 87 | 90 | 90 | 90 | 94 | 94 | 97 | 97 | 100 | 103 | 106 | 109 | 109 | 114 | 114 | 114 | 117 | 120 | 126 | 129 | 132 |
| | | 33 | 87 | 87 | 87 | 87 | 90 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 103 | 106 | 109 | 112 | 112 | 117 | 117 | 117 | 120 | 123 | 129 | 132 | 136 |
| | | 34 | 87 | 87 | 87 | 87 | 90 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 103 | 106 | 109 | 112 | 112 | 117 | 117 | 117 | 120 | 123 | 129 | 132 | 136 |
| | | 35 | 90 | 90 | 90 | 90 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 112 | 114 | 114 | 120 | 120 | 120 | 123 | 126 | 132 | 136 | 140 |
| | | 36 | 90 | 90 | 90 | 90 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 112 | 114 | 114 | 120 | 120 | 120 | 123 | 126 | 132 | 136 | 140 |
| | | 37 | 94 | 94 | 94 | 94 | 97 | 100 | 100 | 100 | 103 | 103 | 106 | 106 | 109 | 112 | 114 | 117 | 117 | 123 | 123 | 123 | 126 | 129 | 136 | 140 | 144 |
| | | 38 | 97 | 97 | 97 | 97 | 100 | 103 | 103 | 103 | 106 | 106 | 109 | 109 | 112 | 114 | 117 | 120 | 120 | 126 | 126 | 126 | 129 | 132 | 140 | 144 | 148 |
| | | 39 | 97 | 97 | 97 | 97 | 100 | 103 | 103 | 103 | 106 | 106 | 109 | 109 | 112 | 114 | 117 | 120 | 120 | 126 | 126 | 126 | 129 | 132 | 140 | 144 | 148 |
| | | 40 | 100 | 100 | 100 | 100 | 103 | 106 | 106 | 106 | 109 | 109 | 112 | 112 | 114 | 117 | 120 | 123 | 123 | 129 | 129 | 129 | 132 | 136 | 144 | 148 | 152 |
| | | 0 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | | 1 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | ļ | 2 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | ļ | 3 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | | 4 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | | 5 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | - | 6 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | - | 7 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | | 8 | 40 | 40 | 44 | 44 | 49 | 49 | 49 | 53 | 53 | 57 | 57 | 61 | 69 | 73 | 73 | 76 | 76 | 78 | 81 | 83 | 83 | 85 | 87 | 90 | 94 |
| | - | 9 | 44 | 44 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 85 | 85 | 87 | 90 | 94 | 97 |
| | - | 10 | 44 | 44 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 85 | 85 | 87 | 90 | 94 | 97 |
| | | 11 | 44 | 44 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 85 | 85 | 87 | 90 | 94 | 97 |
| | ŀ | 12 | 44 | 44 | 49 | 49 | 53 | 53 | 53 | 57 | 57 | 61 | 61 | 65 | 73 | 76 | 76 | 78 | 78 | 81 | 83 | 85 | 85 | 87 | 90 | 94 | 97 |
| | 68 | 13 | 49 | 49 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 76 | 78 | 78 | 81 | 81 | 83 | 85 | 87 | 87 | 90 | 94 | 97 | 100 |
| 8 | 60-00 | 14 | 49 | 49 | 53 | 53 | 57 | 57 | 57 | 61 | 61 | 65 | 65 | 69 | 76 | 78 | 78 | 81 | 81 | 83 | 85 | 87 | 87 | 90 | 94 | 97 | 100 |
| - | des | 15 | 53 | 53 | 57 | 57 | 61 | 61 | 61 | 65 | 65 | 69 | 69 | 73 | 78 | 81 | 81 | 83 | 83 | 85 | 87 | 90 | 90 | 94 | 97 | 100 | 103 |
| | ď | 16 | 57 | 57 | 61 | 61 | 65 | 65 | 65 | 69 | 69 | 73 | 73 | 76 | 81 | 83 | 83 | 85 | 85 | 87 | 90 | 94 | 94 | 97 | 100 | 103 | 106 |

| | Stor | y Mem | ory Tot | al Scor | re | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 |
| 17 | 61 | 61 | 65 | 65 | 69 | 69 | 69 | 73 | 73 | 76 | 76 | 78 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 97 | 97 | 100 | 103 | 106 | 10 |
| 18 | 61 | 61 | 65 | 65 | 69 | 69 | 69 | 73 | 73 | 76 | 76 | 78 | 83 | 85 | 85 | 87 | 87 | 90 | 94 | 97 | 97 | 100 | 103 | 106 | 10 |
| 19 | 65 | 65 | 69 | 69 | 73 | 73 | 73 | 76 | 76 | 78 | 78 | 81 | 85 | 87 | 87 | 90 | 90 | 94 | 97 | 100 | 100 | 103 | 106 | 109 | 11 |
| 20 | 69 | 69 | 73 | 73 | 76 | 76 | 76 | 78 | 78 | 81 | 81 | 83 | 87 | 90 | 90 | 94 | 94 | 97 | 100 | 103 | 103 | 106 | 109 | 112 | 1 |
| 21 | 73 | 73 | 76 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 90 | 94 | 94 | 97 | 97 | 100 | 103 | 106 | 106 | 109 | 112 | 114 | 1 |
| 22 | 73 | 73 | 76 | 76 | 78 | 78 | 78 | 81 | 81 | 83 | 83 | 85 | 90 | 94 | 94 | 97 | 97 | 100 | 103 | 106 | 106 | 109 | 112 | 114 | 1 |
| 23 | 76 | 76 | 78 | 78 | 81 | 81 | 81 | 83 | 83 | 85 | 85 | 87 | 94 | 97 | 97 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 114 | 117 | 1 |
| 24 | 78 | 78 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 112 | 112 | 114 | 117 | 120 | 1 |
| 25 | 78 | 78 | 81 | 81 | 83 | 83 | 83 | 85 | 85 | 87 | 87 | 90 | 97 | 100 | 100 | 103 | 103 | 106 | 109 | 112 | 112 | 114 | 117 | 120 | 1 |
| 26 | 81 | 81 | 83 | 83 | 85 | 85 | 85 | 87 | 87 | 90 | 90 | 94 | 100 | 103 | 103 | 106 | 106 | 109 | 112 | 114 | 114 | 117 | 120 | 123 | 1 |
| 27 | 83 | 83 | 85 | 85 | 87 | 87 | 87 | 90 | 90 | 94 | 94 | 97 | 103 | 106 | 106 | 109 | 109 | 112 | 114 | 117 | 117 | 120 | 123 | 126 | , |
| 28 | 83 | 83 | 85 | 85 | 87 | 87 | 87 | 90 | 90 | 94 | 94 | 97 | 103 | 106 | 106 | 109 | 109 | 112 | 114 | 117 | 117 | 120 | 123 | 126 | , |
| 29 | 85 | 85 | 87 | 87 | 90 | 90 | 90 | 94 | 94 | 97 | 97 | 100 | 106 | 109 | 109 | 112 | 112 | 114 | 117 | 120 | 120 | 123 | 126 | 129 | |
| 30 | 85 | 85 | 87 | 87 | 90 | 90 | 90 | 94 | 94 | 97 | 97 | 100 | 106 | 109 | 109 | 112 | 112 | 114 | 117 | 120 | 120 | 123 | 126 | 129 | |
| 31 | 87 | 87 | 90 | 90 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 103 | 109 | 112 | 112 | 114 | 114 | 117 | 120 | 123 | 123 | 126 | 129 | 132 | |
| 32 | 87 | 87 | 90 | 90 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 103 | 109 | 112 | 112 | 114 | 114 | 117 | 120 | 123 | 123 | 126 | 129 | 132 | |
| 33 | 90 | 90 | 94 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 112 | 114 | 114 | 117 | 117 | 120 | 123 | 126 | 126 | 129 | 132 | 136 | |
| 34 | 90 | 90 | 94 | 94 | 97 | 97 | 97 | 100 | 100 | 103 | 103 | 106 | 112 | 114 | 114 | 117 | 117 | 120 | 123 | 126 | 126 | 129 | 132 | 136 | |
| 35 | 94 | 94 | 97 | 97 | 100 | 100 | 100 | 103 | 103 | 106 | 106 | 109 | 114 | 117 | 117 | 120 | 120 | 123 | 126 | 129 | 129 | 132 | 136 | 140 | |
| 36 | 94 | 94 | 97 | 97 | 100 | 100 | 100 | 103 | 103 | 106 | 106 | 109 | 114 | 117 | 117 | 120 | 120 | 123 | 126 | 129 | 129 | 132 | 136 | 140 | |
| 37 | 97 | 97 | 100 | 100 | 103 | 103 | 103 | 106 | 106 | 109 | 109 | 112 | 117 | 120 | 120 | 123 | 123 | 126 | 129 | 132 | 132 | 136 | 140 | 144 | - |
| 38 | 97 | 97 | 100 | 100 | 103 | 103 | 103 | 106 | 106 | 109 | 109 | 112 | 117 | 120 | 120 | 123 | 123 | 126 | 129 | 132 | 132 | 136 | 140 | 144 | ŀ |
| 39 | 100 | 100 | 103 | 103 | 106 | 106 | 106 | 109 | 109 | 112 | 112 | 114 | 120 | 123 | 123 | 126 | 126 | 129 | 132 | 136 | 136 | 140 | 144 | 148 | ŀ |
| 40 | 100 | 100 | 103 | 103 | 106 | 106 | 106 | 109 | 109 | 112 | 112 | 114 | 120 | 123 | 123 | 126 | 126 | 129 | 132 | 136 | 136 | 140 | 144 | 148 | |

Table 5-18 Visuospatial/Constructional Index Score Equivalents of Subtest Raw Scores

| | Line | Orient | tation 1 | Γotal S | core | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 |
| Ag Ag | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |

| | | | Line | Orient | ation 1 | Total So | core | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | | 19 | 20 |
| | | 1 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | | 81 | 84 |
| | | 2 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | | 81 | 84 |
| | | 3 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | | 81 | 84 |
| | | 4 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | | 81 | 84 |
| | | 5 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | | 81 | 84 |
| | | 6 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | | 81 | 84 |
| | | 7 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | | 81 | 84 |
| | | 8 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | | 81 | 84 |
| | | 9 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | | 81 | 84 |
| | | 10 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | | 81 | 84 |
| | | 11 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | | 81 | 84 |
| | | 12 | 53 | 53 | 53 | 53 | 53 | 53 | 56 | 56 | 58 | 60 | 62 | 62 | 64 | 66 | 66 | 69 | 72 | 75 | 81 | | 84 | 87 |
| | | 13 | 56 | 56 | 56 | 56 | 56 | 56 | 58 | 58 | 60 | 62 | 64 | 64 | 66 | 69 | 69 | 72 | 75 | 78 | 84 | | 87 | 89 |
| | | 14 | 58 | 58 | 58 | 58 | 58 | 58 | 60 | 60 | 62 | 64 | 66 | 66 | 69 | 72 | 72 | 75 | 78 | 81 | 87 | | 89 | 92 |
| | | 15 | 60 | 60 | 60 | 60 | 60 | 60 | 62 | 62 | 64 | 66 | 69 | 69 | 72 | 75 | 75 | 78 | 81 | 84 | 89 | | 92 | 96 |
| | | 16 | 62 | 62 | 62 | 62 | 62 | 62 | 64 | 64 | 66 | 69 | 72 | 72 | 75 | 78 | 78 | 81 | 84 | 87 | 92 | | 96 | 100 |
| | | 17 | 66 | 66 | 66 | 66 | 66 | 66 | 69 | 69 | 72 | 75 | 78 | 78 | 81 | 84 | 84 | 87 | 89 | 92 | 10 | 0 | 102 | 105 |
| | | 18 | 72 | 72 | 72 | 72 | 72 | 72 | 75 | 75 | 78 | 81 | 84 | 84 | 87 | 89 | 89 | 92 | 96 | 100 | 10 | 5 | 109 | 112 |
| | | 19 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 78 | 81 | 84 | 87 | 87 | 89 | 92 | 92 | 96 | 100 | 102 | 109 | 9 | 112 | 116 |
| | | 20 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 84 | 87 | 89 | 92 | 92 | 96 | 100 | 100 | 102 | 105 | 109 | 110 | 6 | 121 | 126 |
| | | | Line | Orienta | ation T | otal Sc | ore | | | | | | | | | | | | | | | | | |
| 1 | | I _ | 0 | 1 | 2 | 3 | 4 | | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 |
| | | 0 | 50 | 50 | 50 | 50 | | 0 | 50 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| Copy | | 1 | 50 | 50<br>50 | 50 | 50 | | 0 | 50 | 53 | 56 | 56<br>56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78<br>70 | 81 | 84 |
| Figure Cog<br>Total Scor | 69-09 | 3 | 50<br>50 | 50 | 50<br>50 | 50<br>50 | | 50<br>50 | 50<br>50 | 53<br>53 | 56<br>56 | 56<br>56 | 58<br>58 | 60<br>60 | 60<br>60 | 62<br>62 | 64<br>64 | 64<br>64 | 66<br>66 | 69 | 72<br>72 | 78<br>78 | 81<br>81 | 84<br>84 |
| are | 9 60 | 4 | 50 | 50<br>50 | 50<br>50 | 50<br>50 | | 50<br>50 | 50<br>50 | 53<br>53 | 56<br>56 | 56<br>56 | 58<br>58 | 60<br>60 | 60<br>60 | 62<br>62 | 64<br>64 | 64<br>64 | 66<br>66 | 69<br>69 | 72<br>72 | 78 | 81<br>81 | 84 |
| <b>₹</b> | des | 7 | 50 | 50 | 50 | 50 | , | | 00 | 00 | 50 | 50 | 50 | 00 | 00 | 02 | 07 | 0+ | 00 | 00 | 1 4 | 7 0 | 01 | 04 |

Novartis

SAP Addendum 2

| | | | Line | Orienta | ation T | otal Sco | е | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 4 | 1 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | • | 19 | 20 |
| | 6 | 5 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 7 | , | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 8 | 3 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 9 | ) | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 1 | 0 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 1 | 1 | 53 | 53 | 53 | 53 | 53 | 53 | 56 | 58 | 58 | 60 | 62 | 62 | 64 | 66 | 66 | 69 | 72 | 75 | 81 | 84 | 87 |
| | 1 | 2 | 53 | 53 | 53 | 53 | 53 | 53 | 56 | 58 | 58 | 60 | 62 | 62 | 64 | 66 | 66 | 69 | 72 | 75 | 81 | 84 | 87 |
| | 1 | 3 | 56 | 56 | 56 | 56 | 56 | 56 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 69 | 72 | 75 | 78 | 84 | 87 | 89 |
| | 1 | 4 | 58 | 58 | 58 | 58 | 58 | 58 | 60 | 62 | 62 | 64 | 66 | 66 | 69 | 72 | 72 | 75 | 78 | 81 | 87 | 89 | 92 |
| | 1 | 5 | 60 | 60 | 60 | 60 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 69 | 72 | 75 | 75 | 78 | 81 | 84 | 89 | 92 | 96 |
| | 1 | 6 | 62 | 62 | 62 | 62 | 62 | 62 | 64 | 66 | 66 | 69 | 72 | 72 | 75 | 78 | 78 | 81 | 84 | 87 | 92 | 96 | 100 |
| | 1 | 7 | 66 | 66 | 66 | 66 | 66 | 66 | 69 | 72 | 72 | 75 | 78 | 78 | 81 | 84 | 84 | 87 | 89 | 92 | 100 | 102 | 105 |
| | 1 | 8 | 72 | 72 | 72 | 72 | 72 | 72 | 75 | 78 | 78 | 81 | 84 | 84 | 87 | 89 | 89 | 92 | 96 | 100 | 105 | 109 | 112 |
| | 1 | 9 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 81 | 84 | 87 | 87 | 89 | 92 | 92 | 96 | 100 | 102 | 109 | 112 | 116 |
| | 2 | 20 | 84 | 84 | 84 | 84 | 84 | 84 | 87 | 89 | 89 | 92 | 96 | 96 | 100 | 102 | 102 | 105 | 109 | 112 | 121 | 126 | 131 |
| | 0 | ) | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 1 | | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 2 | 2 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 3 | 3 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 4 | ŀ | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 5 | 5 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 6 | 5 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 7 | <i>'</i> | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 8 | 3 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | 9 | ) | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| | ł | 0 | 50 | 50 | 50 | 50 | 50 | 50 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 69 | 72 | 78 | 81 | 84 |
| و ا | ღ 1 | 1 | 53 | 53 | 53 | 53 | 53 | 53 | 56 | 58 | 60 | 60 | 62 | 62 | 64 | 66 | 66 | 69 | 72 | 75 | 81 | 84 | 87 |
| 2 | <u>ا</u> و | 2 | 56 | 56 | 56 | 56 | 56 | 56 | 58 | 60 | 62 | 62 | 64 | 64 | 66 | 69 | 69 | 72 | 75 | 78 | 84 | 87 | 89 |
| 6 | O) | 3 | 58 | 58 | 58 | 58 | 58 | 58 | 60 | 62 | 64 | 64 | 66 | 66 | 69 | 72 | 72 | 75 | 78 | 81 | 87 | 89 | 92 |
| 5 | <b>Y</b> 1 | 4 | 58 | 58 | 58 | 58 | 58 | 58 | 60 | 62 | 64 | 64 | 66 | 66 | 69 | 72 | 72 | 75 | 78 | 81 | 87 | 89 | 92 |

| | | Line | Orient | ation To | otal Sco | re | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | • | 19 | 20 |
| | 15 | 60 | 60 | 60 | 60 | 60 | 60 | 62 | 64 | 66 | 66 | 69 | 69 | 72 | 75 | 75 | 78 | 81 | 84 | 89 | 92 | 96 |
| | 16 | 64 | 64 | 64 | 64 | 64 | 64 | 66 | 69 | 72 | 72 | 75 | 75 | 78 | 81 | 81 | 84 | 87 | 89 | 96 | 100 | 10 |
| | 17 | 69 | 69 | 69 | 69 | 69 | 69 | 72 | 75 | 78 | 78 | 81 | 81 | 84 | 87 | 87 | 89 | 92 | 96 | 102 | 105 | 10 |
| | 18 | 72 | 72 | 72 | 72 | 72 | 72 | 75 | 78 | 81 | 81 | 84 | 84 | 87 | 89 | 89 | 92 | 96 | 100 | 105 | 109 | 11 |
| | 19 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 87 | 87 | 89 | 89 | 92 | 96 | 96 | 100 | 102 | 105 | 112 | 116 | 12 |
| | 20 | 84 | 84 | 84 | 84 | 84 | 84 | 87 | 89 | 92 | 92 | 96 | 96 | 100 | 102 | 102 | 105 | 109 | 112 | 121 | 126 | 13 |
| | 0 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 1 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 2 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 3 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 4 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 5 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 6 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 7 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 8 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 9 | 50 | 50 | 50 | 50 | 50 | 53 | 53 | 56 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 69 | 72 | 78 | 81 | 84 | 87 |
| | 10 | 53 | 53 | 53 | 53 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 62 | 64 | 66 | 66 | 72 | 75 | 81 | 84 | 87 | 89 |
| | 11 | 53 | 53 | 53 | 53 | 53 | 56 | 56 | 58 | 60 | 60 | 62 | 62 | 64 | 66 | 66 | 72 | 75 | 81 | 84 | 87 | 89 |
| | 12 | 56 | 56 | 56 | 56 | 56 | 58 | 58 | 60 | 62 | 62 | 64 | 64 | 66 | 69 | 69 | 75 | 78 | 84 | 87 | 89 | 92 |
| | 13 | 58 | 58 | 58 | 58 | 58 | 60 | 60 | 62 | 64 | 64 | 66 | 66 | 69 | 72 | 72 | 78 | 81 | 87 | 89 | 92 | 96 |
| | 14 | 60 | 60 | 60 | 60 | 60 | 62 | 62 | 64 | 66 | 66 | 69 | 69 | 72 | 75 | 75 | 81 | 84 | 89 | 92 | 96 | 10 |
| | 15 | 62 | 62 | 62 | 62 | 62 | 64 | 64 | 66 | 69 | 69 | 72 | 72 | 75 | 78 | 78 | 84 | 87 | 92 | 96 | 100 | 10 |
| 68 | 16 | 66 | 66 | 66 | 66 | 66 | 69 | 69 | 72 | 75 | 75 | 78 | 78 | 81 | 84 | 84 | 89 | 92 | 100 | 102 | 105 | 10 |
| 80-1 | 17 | 72 | 72 | 72 | 72 | 72 | 75 | 75 | 78 | 81 | 81 | 84 | 84 | 87 | 89 | 89 | 96 | 100 | 105 | 109 | 112 | 1 |
| Ages 80-89 | 18 | 75 | 75 | 75 | 75 | 75 | 78 | 78 | 81 | 84 | 84 | 87 | 87 | 89 | 92 | 92 | 100 | 102 | 109 | 112 | 116 | 12 |
| Αg | 19 | 78 | 78 | 78 | 78 | 78 | 81 | 81 | 84 | 87 | 87 | 89 | 89 | 92 | 96 | 96 | 102 | 105 | 112 | 116 | 121 | 12 |
| | 20 | 84 | 84 | 84 | 84 | 84 | 87 | 87 | 89 | 92 | 92 | 96 | 96 | 100 | 102 | 102 | 109 | 112 | 121 | 126 | 131 | 13 |

 Table 5-19
 Language Index Score Equivalents of Subtest Raw Scores

| | | | Picture N | laming Total Sco | ore | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9–10 |
| | | 0 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| | | 1 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| | | 2 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| | | 3 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| | | 4 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| | | 5 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| | | 6 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 71 |
| | | 7 | 44 | 44 | 44 | 44 | 44 | 47 | 51 | 54 | 60 | 75 |
| | | 8 | 44 | 44 | 44 | 44 | 44 | 47 | 51 | 54 | 60 | 75 |
| | | 9 | 47 | 47 | 47 | 47 | 47 | 51 | 54 | 57 | 64 | 79 |
| | | 10 | 47 | 47 | 47 | 47 | 47 | 51 | 54 | 57 | 64 | 79 |
| | | 11 | 47 | 47 | 47 | 47 | 47 | 51 | 54 | 57 | 64 | 79 |
| | | 12 | 51 | 51 | 51 | 51 | 51 | 54 | 57 | 60 | 68 | 82 |
| | | 13 | 51 | 51 | 51 | 51 | 51 | 54 | 57 | 60 | 68 | 82 |
| | | 14 | 54 | 54 | 54 | 54 | 54 | 57 | 60 | 64 | 71 | 84 |
| | | 15 | 57 | 57 | 57 | 57 | 57 | 60 | 64 | 68 | 75 | 87 |
| | | 16 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 71 | 79 | 90 |
| | | 17 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 71 | 79 | 90 |
| | | 18 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 75 | 83 | 94 |
| | | 19 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 75 | 83 | 94 |
| ഉ | | 20 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 79 | 87 | 97 |
| 000 | | 21 | 71 | 71 | 71 | 71 | 71 | 75 | 79 | 83 | 90 | 99 |
| ta | | 22 | 71 | 71 | 71 | 71 | 71 | 75 | 79 | 83 | 90 | 99 |
| Ď | | 23 | 75 | 75 | 75 | 75 | 75 | 79 | 83 | 87 | 92 | 102 |
| incy | | 24 | 75 | 75 | 75 | 75 | 75 | 79 | 83 | 87 | 92 | 102 |
| Flue | 0 | 25 | 79 | 79 | 79 | 79 | 79 | 83 | 87 | 90 | 94 | 105 |
| Iţic I | 50-59 | 26 | 83 | 83 | 83 | 83 | 83 | 87 | 90 | 92 | 96 | 109 |
| Semantic Fluency Total Score | 9S 5 | 27 | 83 | 83 | 83 | 83 | 83 | 87 | 90 | 92 | 96 | 109 |
| Ser | Ages | 28 | 87 | 87 | 87 | 87 | 87 | 90 | 92 | 94 | 100 | 113 |

| | | Picture Na | aming Total Sco | re | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9–10 |
| | 29 | 87 | 87 | 87 | 87 | 87 | 90 | 92 | 94 | 100 | 113 |
| | 30 | 90 | 90 | 90 | 90 | 90 | 92 | 94 | 96 | 102 | 117 |
| | 31 | 92 | 92 | 92 | 92 | 92 | 94 | 96 | 100 | 104 | 120 |
| | 32 | 92 | 92 | 92 | 92 | 92 | 94 | 96 | 100 | 104 | 120 |
| | 33 | 94 | 94 | 94 | 94 | 94 | 96 | 100 | 102 | 108 | 124 |
| | 34 | 96 | 96 | 96 | 96 | 96 | 100 | 102 | 104 | 112 | 127 |
| | 35 | 100 | 100 | 100 | 100 | 100 | 102 | 104 | 108 | 116 | 131 |
| | 36+ | 100 | 100 | 100 | 100 | 100 | 102 | 104 | 108 | 116 | 131 |
| | 0 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 74 |
| | 1 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 74 |
| | 2 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 74 |
| | 3 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 74 |
| | 4 | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 74 |
| | <u>5</u> | 40 | 40 | 40 | 40 | 40 | 44 | 47 | 51 | 57 | 74 |
| | 6 | 44 | 44 | 44 | 44 | 44 | 47 | 51 | 54 | 60 | 78 |
| | 7 | 44 | 44 | 44 | 44 | 44 | 47 | 51 | 54 | 60 | 78 |
| | 8 | 44 | 44 | 44 | 44 | 44 | 47 | 51 | 54 | 60 | 78 |
| | 9 | 47 | 47 | 47 | 47 | 47 | 51 | 54 | 57 | 64 | 82 |
| | 10 | 47 | 47 | 47 | 47 | 47 | 51 | 54 | 57 | 64 | 82 |
| | 11 | 47 | 47 | 47 | 47 | 47 | 51 | 54 | 57 | 64 | 82 |
| | 12 | 51 | 51 | 51 | 51 | 51 | 54 | 57 | 60 | 68 | 85 |
| | 13 | 51 | 51 | 51 | 51 | 51 | 54 | 57 | 60 | 68 | 85 |
| | 14 | 54 | 54 | 54 | 54 | 54 | 57 | 60 | 64 | 71 | 87 |
| | 15 | 57 | 57 | 57 | 57 | 57 | 60 | 64 | 68 | 75 | 90 |
| | 16 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 71 | 79 | 92 |
| Ö | වූ 17 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 71 | 79 | 92 |
| 0 | 18 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 75 | 83 | 96 |
| 9 | 60-00 17<br>18<br>19 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 75 | 83 | 96 |
| 4 | ₹ 20 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 79 | 87 | 98 |

| | | Picture Nami | ng Total Score | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| _ | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9–10 |
| | 21 | 71 | 71 | 71 | 71 | 71 | 75 | 79 | 83 | 90 | 101 |
| | 22 | 71 | 71 | 71 | 71 | 71 | 75 | 79 | 83 | 90 | 101 |
| | 23 | 75 | 75 | 75 | 75 | 75 | 79 | 83 | 87 | 92 | 104 |
| | 24 | 75 | 75 | 75 | 75 | 75 | 79 | 83 | 87 | 92 | 104 |
| | 25 | 79 | 79 | 79 | 79 | 79 | 83 | 87 | 90 | 94 | 108 |
| | 26 | 83 | 83 | 83 | 83 | 83 | 87 | 90 | 92 | 96 | 111 |
| | 27 | 87 | 87 | 87 | 87 | 87 | 90 | 92 | 94 | 100 | 116 |
| | 28 | 87 | 87 | 87 | 87 | 87 | 90 | 92 | 94 | 100 | 116 |
| | 29 | 90 | 90 | 90 | 90 | 90 | 92 | 94 | 96 | 102 | 120 |
| | 30 | 90 | 90 | 90 | 90 | 90 | 92 | 94 | 96 | 102 | 120 |
| | 31 | 94 | 94 | 94 | 94 | 94 | 96 | 100 | 102 | 108 | 127 |
| | 32 | 94 | 94 | 94 | 94 | 94 | 96 | 100 | 102 | 108 | 127 |
| | 33 | 94 | 94 | 94 | 94 | 94 | 96 | 100 | 102 | 108 | 127 |
| | 34 | 96 | 96 | 96 | 96 | 96 | 100 | 102 | 104 | 112 | 130 |
| | 35 | 100 | 100 | 100 | 100 | 100 | 102 | 104 | 108 | 116 | 134 |
| | 36+ | 100 | 100 | 100 | 100 | 100 | 102 | 104 | 108 | 116 | 134 |
| | 0 | 40 | 40 | 40 | 40 | 40 | 47 | 47 | 51 | 57 | 74 |
| | 1 | 40 | 40 | 40 | 40 | 40 | 47 | 47 | 51 | 57 | 74 |
| | 2 | 40 | 40 | 40 | 40 | 40 | 47 | 47 | 51 | 57 | 74 |
| | 3 | 40 | 40 | 40 | 40 | 40 | 47 | 47 | 51 | 57 | 74 |
| | 4 | 40 | 40 | 40 | 40 | 40 | 47 | 47 | 51 | 57 | 74 |
| | <u>5</u> | 40 | 40 | 40 | 40 | 40 | 47 | 47 | 51 | 57 | 74 |
| | 6 | 44 | 44 | 44 | 44 | 44 | 51 | 51 | 54 | 60 | 78 |
| | 7 | 44 | 44 | 44 | 44 | 44 | 51 | 51 | 54 | 60 | 78 |
| | 8 | 47 | 47 | 47 | 47 | 47 | 54 | 54 | 57 | 64 | 82 |
| | 9 | 47 | 47 | 47 | 47 | 47 | 54 | 54 | 57 | 64 | 82 |
| 6 | 10 | 51 | 51 | 51 | 51 | 51 | 57 | 57 | 60 | 68 | 85 |
| Ages 70-79 | 11 | 51 | 51 | 51 | 51 | 51 | 57 | 57 | 60 | 68 | 85 |
| es 7 | 12 | 54 | 54 | 54 | 54 | 54 | 60 | 60 | 64 | 71 | 88 |
| Ag | 13 | 54 | 54 | 54 | 54 | 54 | 60 | 60 | 64 | 71 | 88 |

| | | Picture Na | ming Total Sco | re | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9–10 |
| | 14 | 57 | 57 | 57 | 57 | 57 | 64 | 64 | 68 | 75 | 90 |
| | 15 | 60 | 60 | 60 | 60 | 60 | 68 | 68 | 71 | 79 | 92 |
| | 16 | 60 | 60 | 60 | 60 | 60 | 68 | 68 | 71 | 79 | 92 |
| | 17 | 64 | 64 | 64 | 64 | 64 | 71 | 71 | 75 | 83 | 96 |
| | 18 | 64 | 64 | 64 | 64 | 64 | 71 | 71 | 75 | 83 | 96 |
| | 19 | 68 | 68 | 68 | 68 | 68 | 75 | 75 | 79 | 87 | 99 |
| | 20 | 71 | 71 | 71 | 71 | 71 | 79 | 79 | 83 | 90 | 101 |
| | 21 | 75 | 75 | 75 | 75 | 75 | 83 | 83 | 87 | 92 | 105 |
| | 22 | 75 | 75 | 75 | 75 | 75 | 83 | 83 | 87 | 92 | 105 |
| | 23 | 79 | 79 | 79 | 79 | 79 | 87 | 87 | 90 | 94 | 108 |
| | 24 | 79 | 79 | 79 | 79 | 79 | 87 | 87 | 90 | 94 | 108 |
| | 25 | 83 | 83 | 83 | 83 | 83 | 90 | 90 | 92 | 96 | 112 |
| | 26 | 83 | 83 | 83 | 83 | 83 | 90 | 90 | 92 | 96 | 112 |
| | 27 | 87 | 87 | 87 | 87 | 87 | 92 | 92 | 94 | 100 | 117 |
| | 28 | 90 | 90 | 90 | 90 | 90 | 94 | 94 | 96 | 102 | 120 |
| | 29 | 92 | 92 | 92 | 92 | 92 | 96 | 96 | 100 | 104 | 124 |
| | 30 | 92 | 92 | 92 | 92 | 92 | 96 | 96 | 100 | 104 | 124 |
| | 31 | 94 | 94 | 94 | 94 | 94 | 100 | 100 | 102 | 108 | 128 |
| | 32 | 94 | 94 | 94 | 94 | 94 | 100 | 100 | 102 | 108 | 128 |
| | 33 | 96 | 96 | 96 | 96 | 96 | 102 | 102 | 104 | 112 | 131 |
| | 34 | 100 | 100 | 100 | 100 | 100 | 104 | 104 | 108 | 116 | 134 |
| | 35 | 100 | 100 | 100 | 100 | 100 | 104 | 104 | 108 | 116 | 134 |
| | 36+ | 100 | 100 | 100 | 100 | 100 | 104 | 104 | 108 | 116 | 134 |
| | 0 | 40 | 40 | 40 | 40 | 40 | 47 | 51 | 54 | 57 | 76 |
| | 1 | 40 | 40 | 40 | 40 | 40 | 47 | 51 | 54 | 57 | 76 |
| | 2 | 40 | 40 | 40 | 40 | 40 | 47 | 51 | 54 | 57 | 76 |
| 6 | 3 | 40 | 40 | 40 | 40 | 40 | 47 | 51 | 54 | 57 | 76 |
| Ages 80-89 | 4 | 40 | 40 | 40 | 40 | 40 | 47 | 51 | 54 | 57 | 76 |
| 98 88 | <u>5</u> | 44 | 44 | 44 | 44 | 44 | 51 | 54 | 57 | 60 | 80 |
| Age | 6 | 44 | 44 | 44 | 44 | 44 | 51 | 54 | 57 | 60 | 80 |

| | Picture N | aming Total Sco | re | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9–10 |
| 7 | 44 | 44 | 44 | 44 | 44 | 51 | 54 | 57 | 60 | 80 |
| 8 | 47 | 47 | 47 | 47 | 47 | 54 | 57 | 60 | 64 | 83 |
| 9 | 51 | 51 | 51 | 51 | 51 | 57 | 60 | 64 | 68 | 86 |
| 10 | 51 | 51 | 51 | 51 | 51 | 57 | 60 | 64 | 68 | 86 |
| 11 | 54 | 54 | 54 | 54 | 54 | 60 | 64 | 68 | 71 | 89 |
| 12 | 57 | 57 | 57 | 57 | 57 | 64 | 68 | 71 | 75 | 92 |
| 13 | 57 | 57 | 57 | 57 | 57 | 64 | 68 | 71 | 75 | 92 |
| 14 | 60 | 60 | 60 | 60 | 60 | 68 | 71 | 75 | 79 | 95 |
| 15 | 64 | 64 | 64 | 64 | 64 | 71 | 75 | 79 | 83 | 97 |
| 16 | 68 | 68 | 68 | 68 | 68 | 75 | 79 | 83 | 87 | 99 |
| 17 | 71 | 71 | 71 | 71 | 71 | 79 | 83 | 87 | 90 | 103 |
| 18 | 71 | 71 | 71 | 71 | 71 | 79 | 83 | 87 | 90 | 103 |
| 19 | 75 | 75 | 75 | 75 | 75 | 83 | 87 | 90 | 92 | 107 |
| 20 | 79 | 79 | 79 | 79 | 79 | 87 | 90 | 92 | 94 | 110 |
| 21 | 83 | 83 | 83 | 83 | 83 | 90 | 92 | 94 | 96 | 113 |
| 22 | 87 | 87 | 87 | 87 | 87 | 92 | 94 | 96 | 100 | 117 |
| 23 | 90 | 90 | 90 | 90 | 90 | 94 | 96 | 100 | 102 | 122 |
| 24 | 90 | 90 | 90 | 90 | 90 | 94 | 96 | 100 | 102 | 122 |
| 25 | 92 | 92 | 92 | 92 | 92 | 96 | 100 | 102 | 104 | 125 |
| 26 | 92 | 92 | 92 | 92 | 92 | 96 | 100 | 102 | 104 | 125 |
| 27 | 94 | 94 | 94 | 94 | 94 | 100 | 102 | 104 | 108 | 129 |
| 28 | 94 | 94 | 94 | 94 | 94 | 100 | 102 | 104 | 108 | 129 |
| 29 | 94 | 94 | 94 | 94 | 94 | 100 | 102 | 104 | 108 | 129 |
| 30 | 96 | 96 | 96 | 96 | 96 | 102 | 104 | 108 | 112 | 133 |
| 31 | 96 | 96 | 96 | 96 | 96 | 102 | 104 | 108 | 112 | 133 |
| 32 | 96 | 96 | 96 | 96 | 96 | 102 | 104 | 108 | 112 | 133 |
| 33 | 100 | 100 | 100 | 100 | 100 | 104 | 108 | 112 | 116 | 137 |
| 34 | 100 | 100 | 100 | 100 | 100 | 104 | 108 | 112 | 116 | 137 |
| 35 | 100 | 100 | 100 | 100 | 100 | 104 | 108 | 112 | 116 | 137 |
| 36+ | 100 | 100 | 100 | 100 | 100 | 104 | 108 | 112 | 116 | 137 |

| | | | Digit S | Span To | otal Sco | re | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| | | 0 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 1 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 2 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 3 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 4 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 5 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 6 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 7 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 8 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 9 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 10 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 11 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 64 | 72 | 75 | 79 | 82 | 85 | 88 | 91 |
| | | 12 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| | | 13 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| | | 14 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| | | 15 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| | | 16 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| | | 17 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| e C | | 18 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 68 | 75 | 79 | 82 | 85 | 88 | 91 | 94 |
| SC | | 19 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |
| Coding Total Score | 6 | 20 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |
| Ĭ l | 50-59 | 21 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |
| dinç | es & | 22 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |
| Ŝ | Ages | 23 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |

| | Digit | Span To | otal Sco | re | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| 24 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |
| 25 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 72 | 79 | 82 | 85 | 88 | 91 | 94 | 97 |
| 26 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 75 | 82 | 85 | 88 | 91 | 94 | 97 | 100 |
| 27 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 75 | 82 | 85 | 88 | 91 | 94 | 97 | 100 |
| 28 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 75 | 82 | 85 | 88 | 91 | 94 | 97 | 100 |
| 29 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 75 | 82 | 85 | 88 | 91 | 94 | 97 | 100 |
| 30 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 75 | 82 | 85 | 88 | 91 | 94 | 97 | 100 |
| 31 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 72 | 79 | 85 | 88 | 91 | 94 | 97 | 100 | 103 |
| 32 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 72 | 79 | 85 | 88 | 91 | 94 | 97 | 100 | 103 |
| 33 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 72 | 79 | 85 | 88 | 91 | 94 | 97 | 100 | 103 |
| 34 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 75 | 82 | 88 | 91 | 94 | 97 | 100 | 103 | 106 |
| 35 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 75 | 82 | 88 | 91 | 94 | 97 | 100 | 103 | 106 |
| 36 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 75 | 82 | 88 | 91 | 94 | 97 | 100 | 103 | 106 |
| 37 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 79 | 85 | 91 | 94 | 97 | 100 | 103 | 106 | 109 |
| 38 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 79 | 85 | 91 | 94 | 97 | 100 | 103 | 106 | 109 |
| 39 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 79 | 85 | 91 | 94 | 97 | 100 | 103 | 106 | 109 |
| 40 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 79 | 85 | 91 | 94 | 97 | 100 | 103 | 106 | 109 |
| 41 | 64 | 64 | 64 | 64 | 68 | 72 | 75 | 79 | 82 | 88 | 94 | 97 | 100 | 103 | 106 | 109 | 112 |
| 42 | 64 | 64 | 64 | 64 | 68 | 72 | 75 | 79 | 82 | 88 | 94 | 97 | 100 | 103 | 106 | 109 | 112 |
| 43 | 68 | 68 | 68 | 68 | 72 | 75 | 79 | 82 | 85 | 91 | 97 | 100 | 103 | 106 | 109 | 112 | 115 |
| 44 | 68 | 68 | 68 | 68 | 72 | 75 | 79 | 82 | 85 | 91 | 97 | 100 | 103 | 106 | 109 | 112 | 115 |
| 45 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 88 | 94 | 100 | 103 | 106 | 109 | 112 | 115 | 118 |
| 46 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 88 | 94 | 100 | 103 | 106 | 109 | 112 | 115 | 118 |
| 47 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 88 | 94 | 100 | 103 | 106 | 109 | 112 | 115 | 118 |
| 48 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 88 | 94 | 100 | 103 | 106 | 109 | 112 | 115 | 118 |

| | | ı | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Digit S | Span To | tal Sco | | 1 | | ı | 1 | | | 1 | 1 | | | | | |
| i | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| | 4 | 19 | 75 | 75 | 75 | 75 | 79 | 82 | 85 | 88 | 91 | 97 | 103 | 106 | 109 | 112 | 115 | 118 | 122 |
| | 5 | 50 | 75 | 75 | 75 | 75 | 79 | 82 | 85 | 88 | 91 | 97 | 103 | 106 | 109 | 112 | 115 | 118 | 122 |
| | 5 | 51 | 79 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 94 | 100 | 106 | 109 | 112 | 115 | 118 | 122 | 125 |
| | 5 | 52 | 79 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 94 | 100 | 106 | 109 | 112 | 115 | 118 | 122 | 125 |
| | 5 | 53 | 79 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 94 | 100 | 106 | 109 | 112 | 115 | 118 | 122 | 125 |
| | 5 | 54 | 82 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 97 | 103 | 109 | 112 | 115 | 118 | 122 | 125 | 128 |
| | 5 | 55 | 82 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 97 | 103 | 109 | 112 | 115 | 118 | 122 | 125 | 128 |
| | 5 | 56 | 82 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 97 | 103 | 109 | 112 | 115 | 118 | 122 | 125 | 128 |
| | 5 | 57 | 85 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 100 | 106 | 112 | 115 | 118 | 122 | 125 | 128 | 132 |
| | 5 | 58 | 85 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 100 | 106 | 112 | 115 | 118 | 122 | 125 | 128 | 132 |
| | 5 | 59 | 85 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 100 | 106 | 112 | 115 | 118 | 122 | 125 | 128 | 132 |
| | 6 | 60 | 85 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 100 | 106 | 112 | 115 | 118 | 122 | 125 | 128 | 132 |
| | 6 | 31 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 103 | 109 | 115 | 118 | 122 | 125 | 128 | 132 | 135 |
| | 6 | 32 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 103 | 109 | 115 | 118 | 122 | 125 | 128 | 132 | 135 |
| | 6 | 3 | 91 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 106 | 112 | 118 | 122 | 125 | 128 | 132 | 135 | 138 |
| | 6 | 64 | 91 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 106 | 112 | 118 | 122 | 125 | 128 | 132 | 135 | 138 |
| | 6 | 35 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 115 | 122 | 125 | 128 | 132 | 135 | 138 | 142 |
| | 6 | 66 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 115 | 122 | 125 | 128 | 132 | 135 | 138 | 142 |
| | 6 | 67 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 115 | 122 | 125 | 128 | 132 | 135 | 138 | 142 |
| | 6 | 88 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 118 | 125 | 128 | 132 | 135 | 138 | 142 | 146 |
| | 6 | 69 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 118 | 125 | 128 | 132 | 135 | 138 | 142 | 146 |
| | 7 | 70 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 118 | 125 | 128 | 132 | 135 | 138 | 142 | 146 |
| | 7 | 71 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 118 | 125 | 128 | 132 | 135 | 138 | 142 | 146 |
| | 7 | 72 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | 7 | 73 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |

| | | | Digit ( | Onan Ta | tal Cas | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Digit 8 | Span To | tal Sco | е<br>3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| j | | 74 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 75 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 76 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 77 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 78 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 79 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 80 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 81 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 82 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 83 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 84 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 85 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 86 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 87 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 88 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 89 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 122 | 128 | 132 | 135 | 138 | 142 | 146 | 150 |
| | | 0 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | | 1 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | | 2 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | | 3 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | | 4 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | 69 | 5 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | 69-09 | 6 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | es | 7 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | Ą | 8 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |

| | 1 | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Digi | t Span T | | | 1 | 1 | T | | T | | 1 | Т | 1 | | 1 | Т | т — |
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| 9 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 10 | 40 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| 11 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 12 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 13 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 14 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 15 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 16 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 17 | 43 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| 18 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 19 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 20 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 21 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 22 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 23 | 46 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 24 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 25 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 26 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 27 | 49 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 28 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 75 | 79 | 85 | 88 | 91 | 97 | 100 | 103 | 103 |
| 29 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 75 | 79 | 85 | 88 | 91 | 97 | 100 | 103 | 103 |
| 30 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 75 | 79 | 85 | 88 | 91 | 97 | 100 | 103 | 103 |
| 31 | 53 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 75 | 79 | 85 | 88 | 91 | 97 | 100 | 103 | 103 |
| 32 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 33 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |

| | Digit 9 | Span To | otal Sco | re | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| 34 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 35 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 36 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 37 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 38 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 39 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 40 | 60 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 41 | 64 | 64 | 64 | 64 | 68 | 72 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |
| 42 | 64 | 64 | 64 | 64 | 68 | 72 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |
| 43 | 68 | 68 | 68 | 68 | 72 | 75 | 79 | 82 | 88 | 91 | 97 | 100 | 103 | 109 | 112 | 115 | 115 |
| 44 | 68 | 68 | 68 | 68 | 72 | 75 | 79 | 82 | 88 | 91 | 97 | 100 | 103 | 109 | 112 | 115 | 115 |
| 45 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| 46 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| 47 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| 48 | 72 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| 49 | 75 | 75 | 75 | 75 | 79 | 82 | 85 | 88 | 94 | 97 | 103 | 106 | 109 | 115 | 118 | 122 | 122 |
| 50 | 79 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 97 | 100 | 106 | 109 | 112 | 118 | 122 | 125 | 125 |
| 51 | 79 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 97 | 100 | 106 | 109 | 112 | 118 | 122 | 125 | 125 |
| 52 | 82 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 100 | 103 | 109 | 112 | 115 | 122 | 125 | 128 | 128 |
| 53 | 82 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 100 | 103 | 109 | 112 | 115 | 122 | 125 | 128 | 128 |
| 54 | 85 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 103 | 106 | 112 | 115 | 118 | 125 | 128 | 132 | 132 |
| 55 | 85 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 103 | 106 | 112 | 115 | 118 | 125 | 128 | 132 | 132 |
| 56 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 106 | 109 | 115 | 118 | 122 | 128 | 132 | 135 | 135 |
| 57 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 106 | 109 | 115 | 118 | 122 | 128 | 132 | 135 | 135 |
| 58 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 106 | 109 | 115 | 118 | 122 | 128 | 132 | 135 | 135 |

| | Digit 9 | Span To | 1 | 1 | 1 | 1 | T | 1 | 1 | T | 1 | 1 | 1 | 1 | 1 | 1 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| 59 | 91 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 109 | 112 | 118 | 122 | 125 | 132 | 135 | 138 | 138 |
| 60 | 91 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 109 | 112 | 118 | 122 | 125 | 132 | 135 | 138 | 138 |
| 61 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| 62 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| 63 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| 64 | 94 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| 65 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| 66 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| 67 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| 68 | 97 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| 69 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 70 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 71 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 72 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 73 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 74 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 75 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 76 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 77 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 78 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 79 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 80 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 81 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 82 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 83 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |

| | | Dinit On an Tatal Cooks | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Digit Span Total Score | | | | | | | | | | | | 1 | 1 | 1 | | |
| i | 1 | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| | 84 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 85 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 86 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 87 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 88 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 89 | 100 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 70-79 | 0 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| , 70 | 1 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| Ages | 2 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| ⋖ | 3 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | 4 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | 5 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | 6 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | 7 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | 8 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | 9 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | 10 | 40 | 40 | 40 | 43 | 46 | 49 | 49 | 53 | 60 | 64 | 72 | 75 | 79 | 85 | 88 | 91 | 91 |
| | 11 | 43 | 43 | 43 | 46 | 49 | 53 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| | 12 | 43 | 43 | 43 | 46 | 49 | 53 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| | 13 | 43 | 43 | 43 | 46 | 49 | 53 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| | 14 | 43 | 43 | 43 | 46 | 49 | 53 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| | 15 | 43 | 43 | 43 | 46 | 49 | 53 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| | 16 | 43 | 43 | 43 | 46 | 49 | 53 | 53 | 56 | 64 | 68 | 75 | 79 | 82 | 88 | 91 | 94 | 94 |
| | 17 | 46 | 46 | 46 | 49 | 53 | 56 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| | 18 | 46 | 46 | 46 | 49 | 53 | 56 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |

| | Digit | Span To | ntal Sco | re | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| 19 | 46 | 46 | 46 | 49 | 53 | 56 | 56 | 60 | 68 | 72 | 79 | 82 | 85 | 91 | 94 | 97 | 97 |
| 20 | 49 | 49 | 49 | 53 | 56 | 60 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 21 | 49 | 49 | 49 | 53 | 56 | 60 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 22 | 49 | 49 | 49 | 53 | 56 | 60 | 60 | 64 | 72 | 75 | 82 | 85 | 88 | 94 | 97 | 100 | 100 |
| 23 | 53 | 53 | 53 | 56 | 60 | 64 | 64 | 68 | 75 | 79 | 85 | 88 | 91 | 97 | 100 | 103 | 103 |
| 24 | 53 | 53 | 53 | 56 | 60 | 64 | 64 | 68 | 75 | 79 | 85 | 88 | 91 | 97 | 100 | 103 | 103 |
| 25 | 56 | 56 | 56 | 60 | 64 | 68 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 26 | 56 | 56 | 56 | 60 | 64 | 68 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 27 | 56 | 56 | 56 | 60 | 64 | 68 | 68 | 72 | 79 | 82 | 88 | 91 | 94 | 100 | 103 | 106 | 106 |
| 28 | 60 | 60 | 60 | 64 | 68 | 72 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 29 | 60 | 60 | 60 | 64 | 68 | 72 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 30 | 60 | 60 | 60 | 64 | 68 | 72 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 31 | 60 | 60 | 60 | 64 | 68 | 72 | 72 | 75 | 82 | 85 | 91 | 94 | 97 | 103 | 106 | 109 | 109 |
| 32 | 64 | 64 | 64 | 68 | 72 | 75 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |
| 33 | 64 | 64 | 64 | 68 | 72 | 75 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |
| 34 | 64 | 64 | 64 | 68 | 72 | 75 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |
| 35 | 64 | 64 | 64 | 68 | 72 | 75 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |
| 36 | 64 | 64 | 64 | 68 | 72 | 75 | 75 | 79 | 85 | 88 | 94 | 97 | 100 | 106 | 109 | 112 | 112 |
| 37 | 68 | 68 | 68 | 72 | 75 | 79 | 79 | 82 | 88 | 91 | 97 | 100 | 103 | 109 | 112 | 115 | 115 |
| 38 | 68 | 68 | 68 | 72 | 75 | 79 | 79 | 82 | 88 | 91 | 97 | 100 | 103 | 109 | 112 | 115 | 115 |
| 39 | 68 | 68 | 68 | 72 | 75 | 79 | 79 | 82 | 88 | 91 | 97 | 100 | 103 | 109 | 112 | 115 | 115 |
| 40 | 72 | 72 | 72 | 75 | 79 | 82 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| 41 | 72 | 72 | 72 | 75 | 79 | 82 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| 42 | 72 | 72 | 72 | 75 | 79 | 82 | 82 | 85 | 91 | 94 | 100 | 103 | 106 | 112 | 115 | 118 | 118 |
| 43 | 75 | 75 | 75 | 79 | 82 | 85 | 85 | 88 | 94 | 97 | 103 | 106 | 109 | 115 | 118 | 122 | 122 |

| | Digit 9 | Snan To | tal Sco | re | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| 44 | 75 | 75 | 75 | 79 | 82 | 85 | 85 | 88 | 94 | 97 | 103 | 106 | 109 | 115 | 118 | 122 | 122 |
| 45 | 75 | 75 | 75 | 79 | 82 | 85 | 85 | 88 | 94 | 97 | 103 | 106 | 109 | 115 | 118 | 122 | 122 |
| 46 | 79 | 79 | 79 | 82 | 85 | 88 | 88 | 91 | 97 | 100 | 106 | 100 | 112 | 118 | 122 | 125 | 125 |
| 47 | 79 | 79 | 79 | 82 | 85 | 88 | 88 | 91 | 97 | 100 | 106 | 109 | 112 | 118 | 122 | 125 | 125 |
| 48 | 82 | 82 | 82 | 85 | 88 | 91 | 91 | 94 | 100 | 103 | 100 | 112 | 115 | 122 | 125 | 128 | 128 |
| 49 | 82 | 82 | 82 | 85 | 88 | 91 | 91 | 94 | 100 | 103 | 109 | 112 | 115 | 122 | 125 | 128 | 128 |
| 50 | 82 | 82 | 82 | 85 | 88 | 91 | 91 | 94 | 100 | 103 | 109 | 112 | 115 | 122 | 125 | 128 | 128 |
| 51 | 85 | 85 | 85 | 88 | 91 | 94 | 94 | 97 | 103 | 106 | 112 | 115 | 118 | 125 | 128 | 132 | 132 |
| 52 | 85 | 85 | 85 | 88 | 91 | 94 | 94 | 97 | 103 | 106 | 112 | 115 | 118 | 125 | 128 | 132 | 132 |
| 53 | 85 | 85 | 85 | 88 | 91 | 94 | 94 | 97 | 103 | 106 | 112 | 115 | 118 | 125 | 128 | 132 | 132 |
| 54 | 88 | 88 | 88 | 91 | 94 | 97 | 97 | 100 | 106 | 109 | 115 | 118 | 122 | 128 | 132 | 135 | 135 |
| 55 | 88 | 88 | 88 | 91 | 94 | 97 | 97 | 100 | 106 | 109 | 115 | 118 | 122 | 128 | 132 | 135 | 135 |
| 56 | 88 | 88 | 88 | 91 | 94 | 97 | 97 | 100 | 106 | 109 | 115 | 118 | 122 | 128 | 132 | 135 | 135 |
| 57 | 91 | 91 | 91 | 94 | 97 | 100 | 100 | 103 | 109 | 112 | 118 | 122 | 125 | 132 | 135 | 138 | 138 |
| 58 | 91 | 91 | 91 | 94 | 97 | 100 | 100 | 103 | 109 | 112 | 118 | 122 | 125 | 132 | 135 | 138 | 138 |
| 59 | 91 | 91 | 91 | 94 | 97 | 100 | 100 | 103 | 109 | 112 | 118 | 122 | 125 | 132 | 135 | 138 | 138 |
| 60 | 91 | 91 | 91 | 94 | 97 | 100 | 100 | 103 | 109 | 112 | 118 | 122 | 125 | 132 | 135 | 138 | 138 |
| 61 | 94 | 94 | 94 | 97 | 100 | 103 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| 62 | 94 | 94 | 94 | 97 | 100 | 103 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| 63 | 94 | 94 | 94 | 97 | 100 | 103 | 103 | 106 | 112 | 115 | 122 | 125 | 128 | 135 | 138 | 142 | 142 |
| 64 | 97 | 97 | 97 | 100 | 103 | 106 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| 65 | 97 | 97 | 97 | 100 | 103 | 106 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| 66 | 97 | 97 | 97 | 100 | 103 | 106 | 106 | 109 | 115 | 118 | 125 | 128 | 132 | 138 | 142 | 146 | 146 |
| 67 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 68 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | | T | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | ľ | tal Sco | | ı | 1 | 1 | 1 | | | 1 | 1 | | | | 1 | |
| Ī | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| | 69 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 70 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 71 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 72 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 73 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 74 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 75 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 76 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 77 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 78 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 79 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 80 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 81 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 82 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 83 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 84 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 85 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 86 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 87 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 88 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| | 89 | 100 | 100 | 100 | 103 | 106 | 109 | 109 | 112 | 118 | 122 | 128 | 132 | 135 | 142 | 146 | 150 | 150 |
| 6 | 0 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| 8-0 | 1 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| Ages 80-89 | 2 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| Age | 3 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |

| | Digit | Snan To | otal Sco | re | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| 4 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| 5 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| 6 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| 7 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| 8 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| 9 | 40 | 40 | 40 | 43 | 46 | 49 | 53 | 56 | 68 | 72 | 79 | 82 | 85 | 88 | 88 | 91 | 94 |
| 10 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 72 | 75 | 82 | 85 | 88 | 91 | 91 | 94 | 97 |
| 11 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 72 | 75 | 82 | 85 | 88 | 91 | 91 | 94 | 97 |
| 12 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 72 | 75 | 82 | 85 | 88 | 91 | 91 | 94 | 97 |
| 13 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 72 | 75 | 82 | 85 | 88 | 91 | 91 | 94 | 97 |
| 14 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 72 | 75 | 82 | 85 | 88 | 91 | 91 | 94 | 97 |
| 15 | 43 | 43 | 43 | 46 | 49 | 53 | 56 | 60 | 72 | 75 | 82 | 85 | 88 | 91 | 91 | 94 | 97 |
| 16 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 75 | 79 | 85 | 88 | 91 | 94 | 94 | 97 | 100 |
| 17 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 75 | 79 | 85 | 88 | 91 | 94 | 94 | 97 | 100 |
| 18 | 46 | 46 | 46 | 49 | 53 | 56 | 60 | 64 | 75 | 79 | 85 | 88 | 91 | 94 | 94 | 97 | 100 |
| 19 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 79 | 82 | 88 | 91 | 94 | 97 | 97 | 100 | 103 |
| 20 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 79 | 82 | 88 | 91 | 94 | 97 | 97 | 100 | 103 |
| 21 | 49 | 49 | 49 | 53 | 56 | 60 | 64 | 68 | 79 | 82 | 88 | 91 | 94 | 97 | 97 | 100 | 103 |
| 22 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 72 | 82 | 85 | 91 | 94 | 97 | 100 | 100 | 103 | 106 |
| 23 | 53 | 53 | 53 | 56 | 60 | 64 | 68 | 72 | 82 | 85 | 91 | 94 | 97 | 100 | 100 | 103 | 106 |
| 24 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 75 | 85 | 88 | 94 | 97 | 100 | 103 | 103 | 106 | 109 |
| 25 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 75 | 85 | 88 | 94 | 97 | 100 | 103 | 103 | 106 | 109 |
| 26 | 56 | 56 | 56 | 60 | 64 | 68 | 72 | 75 | 85 | 88 | 94 | 97 | 100 | 103 | 103 | 106 | 109 |
| 27 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 79 | 88 | 91 | 97 | 100 | 103 | 106 | 106 | 109 | 112 |
| 28 | 60 | 60 | 60 | 64 | 68 | 72 | 75 | 79 | 88 | 91 | 97 | 100 | 103 | 106 | 106 | 109 | 112 |

| | Divit | O T | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Span To | 1 | 1 | 1 . | T _ | | Τ_ | | | 10 | | 10 | 10 | | 1.5 | 10 |
| I | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| 29 | 64 | 64 | 64 | 68 | 72 | 75 | 79 | 82 | 91 | 94 | 100 | 103 | 106 | 109 | 109 | 112 | 115 |
| 30 | 64 | 64 | 64 | 68 | 72 | 75 | 79 | 82 | 91 | 94 | 100 | 103 | 106 | 109 | 109 | 112 | 115 |
| 31 | 68 | 68 | 68 | 72 | 75 | 79 | 82 | 85 | 94 | 97 | 103 | 106 | 109 | 112 | 112 | 115 | 118 |
| 32 | 68 | 68 | 68 | 72 | 75 | 79 | 82 | 85 | 94 | 97 | 103 | 106 | 109 | 112 | 112 | 115 | 118 |
| 33 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 88 | 97 | 100 | 106 | 109 | 112 | 115 | 115 | 118 | 122 |
| 34 | 72 | 72 | 72 | 75 | 79 | 82 | 85 | 88 | 97 | 100 | 106 | 109 | 112 | 115 | 115 | 118 | 122 |
| 35 | 75 | 75 | 75 | 79 | 82 | 85 | 88 | 91 | 100 | 103 | 109 | 112 | 115 | 118 | 118 | 122 | 125 |
| 36 | 75 | 75 | 75 | 79 | 82 | 85 | 88 | 91 | 100 | 103 | 109 | 112 | 115 | 118 | 118 | 122 | 125 |
| 37 | 75 | 75 | 75 | 79 | 82 | 85 | 88 | 91 | 100 | 103 | 109 | 112 | 115 | 118 | 118 | 122 | 125 |
| 38 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 94 | 103 | 106 | 112 | 115 | 118 | 122 | 122 | 125 | 128 |
| 39 | 79 | 79 | 79 | 82 | 85 | 88 | 91 | 94 | 103 | 106 | 112 | 115 | 118 | 122 | 122 | 125 | 128 |
| 40 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 97 | 106 | 109 | 115 | 118 | 122 | 125 | 125 | 128 | 132 |
| 41 | 82 | 82 | 82 | 85 | 88 | 91 | 94 | 97 | 106 | 109 | 115 | 118 | 122 | 125 | 125 | 128 | 132 |
| 42 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 100 | 109 | 112 | 118 | 122 | 125 | 128 | 128 | 132 | 135 |
| 43 | 85 | 85 | 85 | 88 | 91 | 94 | 97 | 100 | 109 | 112 | 118 | 122 | 125 | 128 | 128 | 132 | 135 |
| 44 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 103 | 112 | 115 | 122 | 125 | 128 | 132 | 132 | 135 | 138 |
| 45 | 88 | 88 | 88 | 91 | 94 | 97 | 100 | 103 | 112 | 115 | 122 | 125 | 128 | 132 | 132 | 135 | 138 |
| 46 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 106 | 115 | 118 | 125 | 128 | 132 | 135 | 135 | 138 | 142 |
| 47 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 106 | 115 | 118 | 125 | 128 | 132 | 135 | 135 | 138 | 142 |
| 48 | 91 | 91 | 91 | 94 | 97 | 100 | 103 | 106 | 115 | 118 | 125 | 128 | 132 | 135 | 135 | 138 | 142 |
| 49 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 118 | 122 | 128 | 132 | 135 | 138 | 138 | 142 | 146 |
| 50 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 118 | 122 | 128 | 132 | 135 | 138 | 138 | 142 | 146 |
| 51 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 118 | 122 | 128 | 132 | 135 | 138 | 138 | 142 | 146 |
| 52 | 94 | 94 | 94 | 97 | 100 | 103 | 106 | 109 | 118 | 122 | 128 | 132 | 135 | 138 | 138 | 142 | 146 |
| 53 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 122 | 125 | 132 | 135 | 138 | 142 | 142 | 146 | 150 |
| 1 00 | 1 | 1 | 1 | 1 | | 1 | 1 | | | 1 | | 1 | 1 | 1 | 1 | 1 | |

| | | Digit S | pan To | tal Sco | | 1 | T | 1 | T | T | 1 | 1 | T | 1 | Т | Т | 1 | т — |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| 54 | 4 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 122 | 125 | 132 | 135 | 138 | 142 | 142 | 146 | 150 |
| 5 | 5 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 122 | 125 | 132 | 135 | 138 | 142 | 142 | 146 | 150 |
| 56 | 6 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 122 | 125 | 132 | 135 | 138 | 142 | 142 | 146 | 150 |
| 57 | 7 | 97 | 97 | 97 | 100 | 103 | 106 | 109 | 112 | 122 | 125 | 132 | 135 | 138 | 142 | 142 | 146 | 150 |
| 58 | 8 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 59 | 9 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 60 | 0 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 6 | 1 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 62 | 2 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 63 | 3 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 64 | 4 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 65 | 5 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 66 | 6 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 67 | 7 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 68 | 8 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 69 | 9 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 70 | 0 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 7 | 1 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 72 | 2 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 73 | 3 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 74 | 4 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 75 | 5 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 76 | 6 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 77 | 7 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 78 | 8 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |

| | Digit S | Span To | tal Sco | re | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 |
| 79 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 80 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 81 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 82 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 83 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 84 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 85 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 86 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 87 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 88 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |
| 89 | 100 | 100 | 100 | 103 | 106 | 109 | 112 | 115 | 125 | 128 | 135 | 138 | 142 | 146 | 146 | 150 | 154 |

Table 5-21 Delayed Memory Index Score Equivalents of Subtest Raw Scores

| | | | List | Recog | gnitior | n Tota | Scor | е | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19–<br>20 |
| ure | | 0 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| Figu | | 1 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| _ | | 2 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| ist/Story | | 3 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| st/8 | 29 | 4 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| of Li | -09 | 5 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| o mu | S | 6 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |
| Sur | Age | 7 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 44 | 48 | 48 | 52 | 60 | 77 |

| | List | Reco | gnitio | n Tota | l Scor | е | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19-<br>20 |
| 8 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 48 | 52 | 52 | 56 | 64 | 80 |
| 9 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 48 | 52 | 52 | 56 | 64 | 80 |
| 7 | <b>0</b> 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 52 | 56 | 56 | 60 | 68 | 82 |
| • | <b>1</b> 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 52 | 56 | 56 | 60 | 68 | 82 |
| • | <b>2</b> 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 52 | 56 | 56 | 60 | 68 | 82 |
| • | <b>3</b> 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 56 | 60 | 60 | 64 | 71 | 85 |
| • | <b>4</b> 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 56 | 60 | 60 | 64 | 71 | 85 |
| • | <b>5</b> 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 60 | 60 | 64 | 64 | 68 | 75 | 88 |
| • | <b>6</b> 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 64 | 68 | 68 | 71 | 78 | 91 |
| • | <b>7</b> 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 64 | 68 | 68 | 71 | 78 | 91 |
| • | <b>8</b> 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 64 | 68 | 68 | 71 | 78 | 91 |
| | <b>9</b> 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 64 | 68 | 68 | 71 | 78 | 91 |
| 2 | <b>6</b> 0 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 64 | 68 | 68 | 71 | 78 | 91 |
| 2 | 2 <b>1</b> 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 68 | 71 | 71 | 75 | 81 | 94 |
| 2 | <b>2</b> 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 68 | 71 | 71 | 75 | 81 | 94 |
| 2 | <b>3</b> 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 68 | 71 | 71 | 75 | 81 | 94 |
| 2 | <b>4</b> 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 68 | 71 | 71 | 75 | 81 | 94 |
| 2 | <b>.5</b> 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 71 | 75 | 75 | 78 | 84 | 97 |
| 2 | <b>6</b> 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 71 | 75 | 75 | 78 | 84 | 97 |
| 2 | ? <b>7</b> 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 75 | 78 | 78 | 81 | 86 | 99 |
| 2 | <b>8</b> 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 75 | 78 | 78 | 81 | 86 | 99 |
| 2 | <b>9</b> 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 78 | 81 | 81 | 84 | 88 | 101 |
| [ : | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 78 | 81 | 81 | 84 | 88 | 101 |
| | <b>1</b> 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 81 | 84 | 84 | 86 | 91 | 105 |

| | | List | Recog | gnition | n Tota | l Scor | е | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19-<br>20 |
| | 32 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 81 | 84 | 84 | 86 | 91 | 105 |
| | 33 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 84 | 86 | 86 | 88 | 94 | 108 |
| | 34 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 84 | 86 | 86 | 88 | 94 | 108 |
| | 35 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 86 | 88 | 88 | 91 | 97 | 111 |
| | 36 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 88 | 88 | 91 | 91 | 94 | 100 | 115 |
| | 37 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 91 | 94 | 94 | 97 | 102 | 119 |
| | 38 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 91 | 94 | 94 | 97 | 102 | 119 |
| | 39 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 94 | 97 | 97 | 100 | 104 | 124 |
| | 40 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 94 | 97 | 97 | 100 | 104 | 124 |
| | 41 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 97 | 97 | 100 | 100 | 102 | 108 | 127 |
| | 42 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 100 | 100 | 102 | 102 | 104 | 112 | 131 |
| | 0 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| | 1 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| | 2 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| | 3 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| | 4 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| | 5 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| | 6 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 48 | 56 | 60 | 78 |
| | 7 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 52 | 60 | 64 | 81 |
| | 8 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 52 | 60 | 64 | 81 |
| 69 | 9 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 52 | 60 | 64 | 81 |
| 69-09 | 10 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 56 | 56 | 64 | 68 | 84 |
| Ages ( | 11 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 56 | 56 | 64 | 68 | 84 |
| Ag | 12 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 56 | 56 | 64 | 68 | 84 |

| | List | Recog | gnition | 1 Tota | l Scor | e | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19–<br>20 |
| 13 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 60 | 60 | 60 | 68 | 71 | 86 |
| 14 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 60 | 60 | 60 | 68 | 71 | 86 |
| 15 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 60 | 64 | 64 | 64 | 71 | 75 | 89 |
| 16 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 68 | 68 | 75 | 78 | 92 |
| 17 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 68 | 68 | 75 | 78 | 92 |
| 18 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 68 | 68 | 75 | 78 | 92 |
| 19 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 71 | 78 | 81 | 95 |
| 20 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 71 | 78 | 81 | 95 |
| 21 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 71 | 78 | 81 | 95 |
| 22 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 71 | 78 | 81 | 95 |
| 23 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 75 | 75 | 81 | 84 | 98 |
| 24 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 75 | 75 | 81 | 84 | 98 |
| 25 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 75 | 75 | 81 | 84 | 98 |
| 26 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 78 | 78 | 84 | 86 | 100 |
| 27 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 78 | 78 | 84 | 86 | 100 |
| 28 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 81 | 81 | 86 | 88 | 102 |
| 29 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 81 | 81 | 86 | 88 | 102 |
| 30 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 81 | 81 | 86 | 88 | 102 |
| 31 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 84 | 84 | 88 | 91 | 106 |
| 32 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 84 | 84 | 88 | 91 | 106 |
| 33 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 86 | 86 | 86 | 91 | 94 | 110 |
| 34 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 88 | 88 | 94 | 97 | 112 |
| 35 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 88 | 88 | 94 | 97 | 112 |
| 36 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 88 | 91 | 91 | 91 | 97 | 100 | 116 |

| | | List | Recog | nitior | n Tota | l Scor | <b>e</b> | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19-<br>20 |
| | 37 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 94 | 94 | 100 | 102 | 121 |
| | 38 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 94 | 94 | 100 | 102 | 121 |
| | 39 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 97 | 97 | 97 | 102 | 104 | 126 |
| | 40 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 97 | 97 | 97 | 102 | 104 | 126 |
| | 41 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 97 | 100 | 100 | 100 | 104 | 108 | 129 |
| | 42 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 100 | 102 | 102 | 102 | 108 | 112 | 133 |
| | 0 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 52 | 56 | 60 | 79 |
| | 1 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 52 | 56 | 60 | 79 |
| | 2 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 52 | 56 | 60 | 79 |
| | 3 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 52 | 56 | 60 | 79 |
| | 4 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 48 | 52 | 56 | 60 | 79 |
| | 5 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 56 | 60 | 64 | 82 |
| | 6 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 56 | 60 | 64 | 82 |
| | 7 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 56 | 60 | 64 | 82 |
| | 8 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 52 | 56 | 60 | 64 | 82 |
| | 9 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 56 | 60 | 64 | 68 | 85 |
| | 10 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 56 | 60 | 64 | 68 | 85 |
| | 11 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 56 | 60 | 64 | 68 | 85 |
| | 12 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 60 | 60 | 64 | 68 | 71 | 87 |
| | 13 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 60 | 60 | 64 | 68 | 71 | 87 |
| 79 | 14 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 60 | 64 | 64 | 68 | 71 | 75 | 90 |
| 70-79 | 15 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 68 | 71 | 75 | 78 | 93 |
| Ages | 16 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 68 | 71 | 75 | 78 | 93 |
| _ ¥ | 17 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 68 | 71 | 75 | 78 | 93 |

| | | List | Recog | nitior | 1 Tota | l Scor | e | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19–<br>20 |
| | 18 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 75 | 78 | 81 | 95 |
| | 19 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 75 | 78 | 81 | 95 |
| | 20 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 71 | 75 | 78 | 81 | 95 |
| | 21 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 75 | 78 | 81 | 84 | 98 |
| | 22 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 75 | 78 | 81 | 84 | 98 |
| | 23 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 78 | 81 | 84 | 86 | 101 |
| | 24 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 78 | 81 | 84 | 86 | 101 |
| | 25 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 78 | 81 | 84 | 86 | 101 |
| | 26 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 81 | 84 | 86 | 88 | 103 |
| | 27 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 81 | 84 | 86 | 88 | 103 |
| | 28 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 84 | 86 | 88 | 91 | 107 |
| | 29 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 84 | 86 | 88 | 91 | 107 |
| | 30 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 86 | 86 | 88 | 91 | 94 | 110 |
| | 31 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 86 | 86 | 88 | 91 | 94 | 110 |
| | 32 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 88 | 91 | 94 | 97 | 113 |
| | 33 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 88 | 91 | 94 | 97 | 113 |
| | 34 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 88 | 91 | 91 | 94 | 97 | 100 | 117 |
| | 35 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 88 | 91 | 91 | 94 | 97 | 100 | 117 |
| | 36 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 94 | 97 | 100 | 102 | 122 |
| | 37 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 94 | 97 | 100 | 102 | 122 |
| | 38 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 94 | 97 | 100 | 102 | 122 |
| | 39 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 97 | 97 | 100 | 102 | 104 | 127 |
| <u> </u> | 40 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 97 | 100 | 100 | 102 | 104 | 108 | 130 |
| | 41 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 100 | 102 | 102 | 104 | 108 | 112 | 134 |

| | | List | Recog | nitior | Tota | Score | <b>e</b> | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19-<br>20 |
| | 42 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 102 | 104 | 104 | 108 | 112 | 115 | 137 |
| | 0 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 52 | 52 | 56 | 64 | 80 |
| | 1 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 40 | 44 | 48 | 52 | 52 | 56 | 64 | 80 |
| | 2 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 56 | 56 | 60 | 68 | 82 |
| | 3 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 56 | 56 | 60 | 68 | 82 |
| | 4 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 44 | 48 | 52 | 56 | 56 | 60 | 68 | 82 |
| | 5 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 60 | 60 | 64 | 71 | 85 |
| | 6 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 60 | 60 | 64 | 71 | 85 |
| | 7 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 48 | 52 | 56 | 60 | 60 | 64 | 71 | 85 |
| | 8 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 60 | 64 | 64 | 68 | 75 | 88 |
| | 9 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 56 | 60 | 64 | 64 | 68 | 75 | 88 |
| | 10 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 68 | 71 | 78 | 90 |
| | 11 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 68 | 71 | 78 | 90 |
| | 12 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 56 | 60 | 64 | 68 | 68 | 71 | 78 | 90 |
| | 13 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 71 | 71 | 75 | 81 | 93 |
| | 14 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 60 | 64 | 68 | 71 | 71 | 75 | 81 | 93 |
| | 15 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 75 | 75 | 78 | 84 | 96 |
| | 16 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 64 | 68 | 71 | 75 | 75 | 78 | 84 | 96 |
| | 17 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 78 | 78 | 81 | 86 | 98 |
| | 18 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 68 | 71 | 75 | 78 | 78 | 81 | 86 | 98 |
| 89 | 19 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 81 | 81 | 84 | 88 | 101 |
| 80-89 | 20 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 81 | 81 | 84 | 88 | 101 |
| Ages ( | 21 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 71 | 75 | 78 | 81 | 81 | 84 | 88 | 101 |
| Ag | 22 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 84 | 84 | 86 | 91 | 104 |

| | List | List Recognition Total Score | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19–<br>20 |
| 23 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 84 | 84 | 86 | 91 | 104 |
| 24 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 75 | 78 | 81 | 84 | 84 | 86 | 91 | 104 |
| 25 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 86 | 86 | 88 | 94 | 107 |
| 26 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 86 | 86 | 88 | 94 | 107 |
| 27 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 78 | 81 | 84 | 86 | 86 | 88 | 94 | 107 |
| 28 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 86 | 88 | 88 | 91 | 97 | 110 |
| 29 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 81 | 84 | 86 | 88 | 88 | 91 | 97 | 110 |
| 30 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 91 | 91 | 94 | 100 | 114 |
| 31 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 91 | 91 | 94 | 100 | 114 |
| 32 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 84 | 86 | 88 | 91 | 91 | 94 | 100 | 114 |
| 33 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 88 | 91 | 94 | 94 | 97 | 102 | 119 |
| 34 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 86 | 88 | 91 | 94 | 94 | 97 | 102 | 119 |
| 35 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 97 | 100 | 104 | 123 |
| 36 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 88 | 91 | 94 | 97 | 97 | 100 | 104 | 123 |
| 37 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 97 | 100 | 100 | 102 | 108 | 126 |
| 38 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 91 | 94 | 97 | 100 | 100 | 102 | 108 | 126 |
| 39 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 97 | 100 | 102 | 102 | 104 | 112 | 131 |
| 40 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 94 | 97 | 100 | 102 | 102 | 104 | 112 | 131 |
| 41 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 97 | 100 | 102 | 104 | 104 | 108 | 115 | 134 |
| 42 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 100 | 102 | 104 | 108 | 108 | 112 | 119 | 137 |

The RBANS Total scores (Total Scale of Index scores) corresponds to the Sum of Index scores in the table below.

Table 5-22 Total Scale Index Score Equivalents of Sum of Index Scores

| Sum of Index<br>Scores | Total Scale<br>of Index<br>Scores | Percentiles | Sum of<br>Index<br>Scores | Total<br>Scale of<br>Index<br>Scores | Percentiles | Sum of Index<br>Scores | Total<br>Scale of<br>Index<br>Scores | Percentiles |
|---|---|---|---|---|---|---|---|---|
| 200–207 | 40 | <0.1 | 427–430 | 81 | 10 | 574–576 | 122 | 93 |
| 208–215 | 41 | <0.1 | 431–435 | 82 | 12 | 577–580 | 123 | 94 |
| 216–223 | 42 | <0.1 | 436-440 | 83 | 13 | 581–583 | 124 | 95 |
| 224–231 | 43 | <0.1 | 441–444 | 84 | 14 | 584–586 | 125 | 95 |
| 232–239 | 44 | <0.1 | 445–449 | 85 | 16 | 587–588 | 126 | 96 |
| 240–247 | 45 | <0.1 | 450–454 | 86 | 18 | 589–591 | 127 | 96 |
| 248–255 | 46 | <0.1 | 455–458 | 87 | 19 | 592–593 | 128 | 97 |
| 256–263 | 47 | <0.1 | 459-461 | 88 | 21 | 594–596 | 129 | 97 |
| 264–271 | 48 | <0.1 | 462-464 | 89 | 23 | 597–598 | 130 | 98 |
| 272–279 | 49 | <0.1 | 465–468 | 90 | 25 | 599–600 | 131 | 98 |
| 280–287 | 50 | <0.1 | 469–471 | 91 | 27 | 601–602 | 132 | 98 |
| 288–295 | 51 | 0.1 | 472–475 | 92 | 30 | 603–604 | 133 | 99 |
| 296–303 | 52 | 0.1 | 476–479 | 93 | 32 | 605–606 | 134 | 99 |
| 304–311 | 53 | 0.1 | 480–483 | 94 | 34 | 607–608 | 135 | 99 |
| 312–319 | 54 | 0.1 | 484–487 | 95 | 37 | 609–610 | 136 | 99 |
| 320–327 | 55 | 0.1 | 488–490 | 96 | 39 | 611–612 | 137 | 99 |
| 328–330 | 56 | 0.2 | 491–493 | 97 | 42 | 613 | 138 | 99 |
| 331–333 | 57 | 0.2 | 494–496 | 98 | 45 | 614–615 | 139 | 99.5 |
| 334–336 | 58 | 0.3 | 497–499 | 99 | 47 | 616–617 | 140 | 99.6 |
| 337–339 | 59 | 0.3 | 500-505 | 100 | 50 | 618–619 | 141 | 99.7 |
| 340–343 | 60 | 0.4 | 506-509 | 101 | 53 | 620–621 | 142 | 99.7 |
| 344–347 | 61 | 0.5 | 510–513 | 102 | 55 | 622–624 | 143 | 99.8 |

| Sum of Index<br>Scores | Total Scale<br>of Index<br>Scores | Percentiles | Sum of<br>Index<br>Scores | Total<br>Scale of<br>Index<br>Scores | Percentiles | Sum of Index<br>Scores | Total<br>Scale of<br>Index<br>Scores | Percentiles |
|---|---|---|---|---|---|---|---|---|
| 348–351 | 62 | 1 | 514–516 | 103 | 58 | 625–628 | 144 | 99.8 |
| 352–355 | 63 | 1 | 517-520 | 104 | 61 | 629–632 | 145 | 99.9 |
| 356–359 | 64 | 1 | 521-523 | 105 | 63 | 633–636 | 146 | 99.9 |
| 360–363 | 65 | 1 | 524-527 | 106 | 66 | 637–639 | 147 | 99.9 |
| 364–367 | 66 | 1 | 528-530 | 107 | 68 | 640–651 | 148 | 99.9 |
| 368–372 | 67 | 1 | 531–533 | 108 | 70 | 652–663 | 149 | 99.9 |
| 373–376 | 68 | 2 | 534-536 | 109 | 73 | 664–675 | 150 | >99.9 |
| 377–380 | 69 | 2 | 537-539 | 110 | 75 | 676–687 | 151 | >99.9 |
| 381–384 | 70 | 2 | 540-542 | 111 | 77 | 688–699 | 152 | >99.9 |
| 385–387 | 71 | 3 | 543-545 | 112 | 79 | 700–711 | 153 | >99.9 |
| 388–391 | 72 | 3 | 546-548 | 113 | 81 | 712–723 | 154 | >99.9 |
| 392–394 | 73 | 4 | 549-551 | 114 | 82 | 724–735 | 155 | >99.9 |
| 395–398 | 74 | 4 | 552-554 | 115 | 84 | 736–748 | 156 | >99.9 |
| 399–402 | 75 | 5 | 555-556 | 116 | 86 | 749–761 | 157 | >99.9 |
| 403–405 | 76 | 5 | 557-559 | 117 | 87 | 762–774 | 158 | >99.9 |
| 406–409 | 77 | 6 | 560-562 | 118 | 88 | 775–787 | 159 | >99.9 |
| 410–414 | 78 | 7 | 563-566 | 119 | 90 | 788–800 | 160 | >99.9 |
| 415–419 | 79 | 8 | 567–570 | 120 | 91 | | | |
| 420–426 | 80 | 9 | 571–573 | 121 | 92 | | | |

## 6 References

Folstein MF, Folstein SE, McHugh PR (1975) A practical method for grading the cognitive state of patients for the clinician. J. psychiat. Res.; 12:189-98.

Raven JC (2000) Standard Progressive Matrices-1998 Edition, updated 2000. Manual for Standard Progressive Matrices (Section 3): NCS Person, Inc.; San Antonio.

Farias ST, Mungas D, Reed BR, et al (2008) The measurement of everyday cognition (ECog): Scale development and psychometric properties. Neuropsychology; 22(4):531-44.

Klunk et al. The Centiloid Project: Standardizing quantitative amyloid plaque estimation by PET. Alzheimer and Dementia 2015 (11): 1-15.

Nakagawa, S., and Cuthill, I. C. (2007). Effect size, confidence interval and statistical Effect size, confidence interval and statistical significance: a practical guide for biologists. Biol. Rev. 82, 591–605.

Bretz F, Maurer W, Brannath W, et al (2009) A graphical approach to sequentially rejective multiple test procedures. Statist. Med.; 28: 586-604.

Jansen W, Ossenkoppele R, Knol D et al (2015) Prevalence of cerebral amyloid pathology in persons without dementia. JAMA; 313(19):1924-38.

Schoenfeld DA (1983). Sample-size formula for the proportional-hazards regression model. Biometrics; 39(2): 499-503.